208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| | · |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase I/II, randomized, placebo-controlled, observer-blind, multicenter study to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' investigational respiratory syncytial virus (RSV) vaccine (adjuvanted with AS01 <sub>E</sub> or AS01 <sub>B</sub> or unadjuvanted) when administered intramuscularly according to a 0, 2 month schedule in adults aged 18-40 or 60-80 years. |
| eTrack study number and<br>Abbreviated Title | 208851 (RSV OA=ADJ-002) |
| Scope: | All data pertaining to the above study (except IDMC analyses) |
| Date of Statistical Analysis<br>Plan | Amendment 2: 17-Mar-2020 |
| Co-ordinating author: | PPD (Statistician) |
| Reviewed by: | (Clinical and Epidemiology Project Lead) (Clinic) (Lead statistician) (Lead statistical analyst) (Scientific writer) (Stat Peer Reviewer) (Regulatory Affairs) (SERM physician) (Safety scientist) (Public disclosure representative) (CLS – Clinical Read-outs) PPD (CMI Expert representative) |
| Approved by: | PPD (Clinical and Epidemiology Project Lead) PPD (Lead statistician) PPD (Statistician) PPD (Lead Scientific writer) PPD (Lead stat Analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 01NOV2018)

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | ABBREVIA | ATIONS | 13 |
| 1. | DOCI | JMENT H | ISTORY | 15 |
| 2. | STUL | DY DESIG | N | 15 |
| 3. | OBJE | | ENDPOINTS | |
| | 3.1. | • | /es | |
| | | 3.1.1. | Primary objective | |
| | | 3.1.2. | Secondary objectives | |
| | | 3.1.3. | Tertiary objectives | |
| | 3.2. | • | nts | |
| | | 3.2.1. | Primary endpoints | |
| | | 3.2.2. | Secondary endpoints | |
| | | 3.2.3. | Tertiary endpoints | 24 |
| 4. | | | TS | |
| | 4.1. | | n | |
| | | 4.1.1. | Exposed Set | |
| | | 4.1.2. | | |
| | 4.2. | | for eliminating data from Analysis Sets | |
| | | 4.2.1. | | |
| | | 4.2.2. | Elimination from Per-protocol analysis Set (PPS) | |
| | | | 4.2.2.1. Excluded subjects | 26 |
| <b>5</b> . | STAT | ISTICAL A | ANALYSES | 30 |
| | 5.1. | | aphy | |
| | | 5.1.1. | Analysis of demographics/baseline characteristics planned | |
| | | | in the protocol | |
| | - 0 | 5.1.2. | | |
| | 5.2. | | re | |
| | | | Analysis of exposure planned in the protocol | |
| | <b>-</b> 0 | 5.2.2. | Additional considerations | |
| | 5.3. | | genicity | |
| | | 5.3.1. | Analysis of immunogenicity planned in the protocol | 31 |
| | | | 5.3.1.1. Within groups evaluation - humoral immune response | 31 |
| | | | 5.3.1.2. Within groups evaluation - Cell-mediated | |
| | | | immune response | 32 |
| | | | 5.3.1.3. Between groups evaluation (Part B only) | |
| | | 5.3.2. | Additional considerations | |
| | | 0.0.2. | 5.3.2.1. Within groups – humoral immune response | |
| | | | 5.3.2.2. Within groups – Cell-mediated immune | |
| | | | response | 35 |
| | | | 5.3.2.3. Between groups analysis | |
| | 5.4. | | s of safety and reactogenicity | 40 |
| | | 5.4.1. | Analysis of safety and reactogenicity planned in the | |
| | | | protocol | |
| | | 5.4.2. | Additional considerations | 41 |

| | | | | 208851 (RSV OA=AL<br>Statistical Analysis Plan Amend | |
|---|---|---|---|---|---|
| | | | 5.4.2.1. | Solicited Adverse Events | |
| | | | 5.4.2.2. | Unsolicited Adverse Events | |
| | | | 5.4.2.3. | Combined Solicited and Unsolicited Adverse | |
| | | | | Events | 43 |
| | | | 5.4.2.4. | Clinical Safety Laboratory Investigations | |
| | | | 5.4.2.5. | | |
| | 5.5. | Analysis | of RTI for I | Part B | 44 |
| | | 5.5.1. | | of RTI planned in the protocol | |
| | | 5.5.2. | Additional | considerations | 44 |
| 6. | ANAL | YSIS INTI | ERPRETAT | TON | 45 |
| 7 | CONIE | NUCT OF | A NIA I VOE | | 4.5 |
| 7. | | | | S | |
| | 7.1.<br>7.2. | | | es | |
| | 1.2. | Statistica | ai considera | ations for interim analyses | 40 |
| 8. | CHAN | IGES FRO | M PLANNI | ED ANALYSES | 47 |
| 9. | NON | STANDAE | ם מדא ח | ERIVATION RULES AND STATISTICAL | |
| ٥. | | | | | 48 |
| | 9.1. | | | data | |
| | 0.1. | 9.1.1. | | | |
| | 9.2. | Duration | | | |
| 10. | | | | | |
| | 10.1. | | | tandard data derivations and statistical methods | |
| | | | | events to vaccine doses | |
| | | 10.1.2. | | of missing data | |
| | | | | Dates | |
| | | | 10.1.2.2. | Laboratory data Daily recording of solicited symptoms | |
| | | | 10.1.2.3. | 10.1.2.3.1. Studies with electronic diaries | |
| | | | 10.1.2.4. | Unsolicited adverse events | |
| | | 10.1.3. | | vation | |
| | | 10.1.0. | 10.1.3.1. | Age at vaccination in years | |
| | | | 10.1.3.2. | Temperature | |
| | | | 10.1.3.3. | Numerical serology results | |
| | | | 10.1.3.4. | Geometric mean titers (GMTs) and | |
| | | | | concentrations (GMCs) | 52 |
| | | | 10.1.3.5. | Onset day | 52 |
| | | | 10.1.3.6. | Duration of events | |
| | | | 10.1.3.7. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 52 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | |
| | | | | adverse events | |
| | | 10.1.4. | | decimals | |
| | | | | Percentages | |
| | | | 10.1.4.2. | <b>0</b> 1 | |
| | | 40.4.5 | 10.1.4.3. | , | |
| | | 10.1.5. | | methodology | |
| | | | | Exact confidence intervals around proportions | |
| | | | ロロコカン | Adjusted GMT or GMC ratios | 54 |

# 208851 | Statistical Analysis Plan Amendment 2 17 Mar 2020 | TMF-1721000 | 2.0

| | | Statistical Analysis Pla | n Amendment 2 |
|-----|-------|------------------------------------|---------------|
| | 10.2. | TFL ToC | 54 |
| 11. | REFE | RENCES | 54 |
| 12. | STUD | Y MOCK TFLS | 55 |
| | 12.1. | Demography | 55 |
| | 12.2. | Exposure | 61 |
| | 12.3. | Immunogenicity | 62 |
| | | 12.3.1. Within groups | |
| | | 12.3.2. Between groups | 73 |
| | 12.4. | Safety | 76 |
| | | Analysis of RTI | |
| | | Additional templates (Amendment 1) | |

| 208851 | Statistical | Analysis Plan | Amendment 2 | 17 Mar | 2020 | TMF | 1721000 L | 20 |
|---|---|---|---|---|---|---|---|---|
| ZUあるこ L | i Statistical . | Anaivsis Pian | Amenament Z | i / Wiar | ZUZU | I I IVIT- | 1/210001 | Z.U |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# **LIST OF TABLES**

| PAG | įΕ |
|---------|----|
| ription | 19 |

| 208851 Statistical Analysis Plan Amendr | nent 2 |
|-------------------------------------------|--------|
|-------------------------------------------|--------|

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study design | 15 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# LIST OF TEMPLATE TABLES

| | | PAGE |
|---|---|---|
| Template Table 1 | Summary of demography and baseline characteristics (Exposed Set) | 55 |
| Template Table 2 | Number of subjects by country and center (Exposed Set) | 56 |
| Template Table 3 | Number of subjects by study steps (Exposed Set) | 56 |
| Template Table 4 | Summary of vital signs (Exposed Set) | 57 |
| Template Table 5 | Summary of study completion with reason for withdrawal (Exposed Set) | 58 |
| Template Table 6 | Summary of visit attendance (Exposed Set) | 58 |
| Template Table 7 | Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set) | 58 |
| Template Table 8 | Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set) | 58 |
| Template Table 9 | Summary of subject disposition from Randomized Set to Exposed set (Randomized set) | 59 |
| Template Table 10 | Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set) | 59 |
| Template Table 11 | Summary of subject disposition from Exposed Set to End of study (Exposed set) | 60 |
| Template Table 12 | Deviations from protocol for age and intervals between study visits (Exposed set) | 60 |
| Template Table 13 | Number of enrolled subjects by country | 60 |
| Template Table 14 | Number of enrolled subjects by age category | 61 |
| Template Table 15 | Minimum and maximum visit dates <analysis name="" set=""></analysis> | 61 |
| Template Table 16 | Exposure to study vaccines by vaccine (Exposed Set) | 61 |
| Template Table 17 | Number and percentage of subjects with <antibody concentration="" titer=""> equal to or above <cut-off unit=""> and <gmt cs=""> <analysis name="" set=""></analysis></gmt></cut-off></antibody> | 62 |
| Template Table 18 | Geometric mean of the individual ratio of <antibody (units)="" concentrations="" titers=""> post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | 63 |

| Tamplete Table 10 | 208851 (RSV OA=A<br>Statistical Analysis Plan Amen | |
|---|---|---|
| Template Table 19 | Distribution of <antibody concentrations="" titers=""> fold increase post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | 63 |
| Template Table 20 | Geometric mean ratios of the fold increase (Pre to Post - vaccination) between RSVPreF3 IgG antibody concentrations and <rsv-a, rsv-b=""> neutralising antibody titers <per protocol="" set=""></per></rsv-a,> | 68 |
| Template Table 21 | Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 69 |
| Template Table 22 | Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by pre-vaccination category <per protocol="" set=""></per> | 69 |
| Template Table 23 | Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 71 |
| Template Table 24 | Descriptive statistics of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <per protocol="" set=""></per> | 72 |
| Template Table 25 | Descriptive statistics of the fold increase (post over pre-<br>vaccination) of the frequency of RSVPreF3 specific-<br>memory B-cells (per million of memory B cells, by Elispot)<br>– Part B <per protocol="" set=""></per> | 72 |
| Template Table 26 | Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 73 |
| Template Table 27 | Comparisons of the 9 RSV formulations versus Placebo in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at one month post <dose (day="" 1="" 2="" 31),="" 91)="" dose=""> (ANCOVA model, Dunnett's test) – Part B <per protocol="" set=""></per></dose></rsv> | 73 |
| Template Table 28 | Comparisons of the mean responses post dose 2 (Day 91) versus post dose 1 (Day 31) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" td="" titers,="" tnfa,<=""><td></td></rsv> | |

| | Statistical Analysis Plan Amendm | |
|---|---|---|
| | IFNg> on pooled groups according to adjuvant content (ANCOVA model) – Part B <per protocol="" set=""></per> | |
| Template Table 29 | Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) - Part B <per protocol="" set=""></per></rsv> | 74 |
| Template Table 30 | Comparisons of the RSV groups (by antigen dose level) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) – Part B <per protocol="" set=""></per></rsv> | 75 |
| Template Table 31 | Parameters of the ANCOVA model for the comparison between RSV groups in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,="">- Part B <analysis name="" set=""></analysis></rsv> | 76 |
| Template Table 32 | Compliance in completing solicited adverse events information (Exposed Set) | 76 |
| Template Table 33 | Incidence and nature of <grade 3=""> symptoms (solicited and unsolicited) <with causal="" relationship="" to="" vaccination=""> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis name="" set=""></analysis></with></grade> | 77 |
| Template Table 34 | Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <a href="mailto:reported-analysis">analysis set name&gt;</a> | 78 |
| Template Table 35 | Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <analysis name="" set=""></analysis> | 78 |
| Template Table 36 | Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <cohort name=""></cohort> | 79 |
| Template Table 37 | Number of days with < local/general> solicited symptoms during < the 7-day (Days 1-7), the whole> post-vaccination period < analysis set name> | 81 |
| Template Table 38 | Percentage of subjects reporting the occurrence of <grade 3=""> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> within the 30-day (Days 1-30) post-</with></grade> | |
| | vaccination period <analysis name="" set=""></analysis> | 83 |

| | 208851 (RSV OA=AI<br>Statistical Analysis Plan Amend | |
|---|---|---|
| Template Table 39 | List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <exposed set=""></exposed> | 83 |
| Template Table 40 | Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment <analysis name="" set=""></analysis> | 83 |
| Template Table 41 | Listing of SAEs <analysis name="" set=""></analysis> | 84 |
| Template Table 42 | Listing of pregnancies reported during the study period in Part A <analysis name="" set=""></analysis> | 84 |
| Template Table 43 | Number and percentage of subjects taking concomitant medication during the <xx>-day (Days 1-<xx>) post-vaccination period by dose and overall <analysis name="" set=""></analysis></xx></xx> | 85 |
| Template Table 44 | Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges, 7 days post dose <1, 2> <analysis name="" set=""></analysis> | 86 |
| Template Table 45 | Summary of hematology and biochemistry results by grade at 7 days post dose <1, 2 > versus baseline ( <day 1,="" 61="" day="">) <analysis name="" set=""></analysis></day> | 86 |
| Template Table 46 | Summary of hemoglobin change from baseline at 7 days post-dose <1, 2> (Exposed set) | 87 |
| Template Table 47 | Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis name="" set=""></analysis> | 88 |
| Template Table 48 | Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis name="" set=""></analysis> | 88 |
| Template Table 49 | Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis name="" set=""></analysis> | 89 |
| Template Table 50 | Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis name="" set=""></analysis> | 89 |
| Template Table 51 | Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <exposed set=""></exposed> | 90 |
| Template Table 52 | Descriptive statistics of the viral load of the RSV- confirmed RTI episodes, as measured by qRT-PCR in nasal/throat | |

| | 208851 (RSV OA=AD.<br>Statistical Analysis Plan Amendn | |
|---|---|---|
| | swab samples collected at assessment visit <at home=""> <exposed set=""></exposed></at> | |
| Template Table 53 | Number and percentage of subjects reporting co-infections with respiratory viruses, as measured by multiplex PCR on RSV A/B positive RTI samples collected <at assessment="" at="" home="" visit,=""> <exposed set=""></exposed></at> | 91 |
| Template Table 54 | Clinical signs and symptoms associated with RTI episodes (Exposed set) | 91 |
| Template Table 55 | Listing of RTI episodes reported during RTI surveillance in Part B (Exposed set) | 92 |
| Template Table 56 | Distribution of hematology and biochemistry parameters at baseline with respect to normal laboratory ranges <analysis name="" set=""></analysis> | 94 |
| Template Table 57 | Summary of follow-up time (in days) up to <dlp contact="" last="" or=""> (Exposed Set)</dlp> | 94 |
| Template Table 58 | Summary of subjects by unsolicited adverse event category | 95 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# **LIST OF TEMPLATE FIGURES**

| | | PAGE |
|---|---|---|
| Template Figure 1 | <gmt cs=""> and their 95% CIs for <antibody concentrations="" titers=""> <analysis name="" set=""></analysis></antibody></gmt> | 62 |
| Template Figure 2 | Reverse cumulative distribution curve of <antibody concentrations="" titers=""> in the <group label=""> group <per protocol="" set=""></per></group></antibody> | 64 |
| Template Figure 3 | Kinetics of < antibody GMT/Cs> on subjects with results available at all timepoints up to <day 14="" 91,="" month=""> <per protocol="" set=""></per></day> | 65 |
| Template Figure 4 | Individual results of <rsv a="" antibody="" neutralizing="" titer=""> at <time point=""> versus pre-vaccination in <group label=""> and Placebo_B groups <per protocol="" set=""></per></group></time></rsv> | 66 |
| Template Figure 5 | Individual results of <rsv a="" antibody="" b="" neutralizing="" rsv="" titer="" versus=""> at <time point=""> , on pooled RSV groups <per protocol="" set=""></per></time></rsv> | 67 |
| Template Figure 6 | Individual results of the fold increase (post over prevaccination) of RSVPreF3 IgG antibody concentrations versus <rsv a,="" b="" rsv=""> neutralizing antibody titers at <time point=""> in <group label=""> <per protocol="" set=""></per></group></time></rsv> | 68 |
| Template Figure 7 | Boxplots with individual data of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 70 |
| Template Figure 8 | Frequency of RSVPreF3 specific CD4+ T-cells expressing any combination of markers among IL-2, CD40L, TNFa, IFNg in <group label=""> group at Day 31 and Day 91 (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per></group> | 71 |
| Template Figure 9 | Incidence of solicited <local, general=""> adverse events reported during the 7-day (Days 1-7) post-vaccination period following each dose <exposed set=""></exposed></local,> | 82 |
| Template Figure 10 | Boxplot of <each biochemistry="" hematology="" parameter=""> (Exposed Set)</each> | 87 |
| Template Figure 11 | GMTs and 95% CIs of RSV A Neutralizing antibody titer at baseline for subjects reporting RTI episodes (RSV RTI vs or non RSV RTI vs No RTI), by groups pooled according to the adjuvant content <exposed set=""></exposed> | 93 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### LIST OF ABBREVIATIONS

AE Adverse event

ALT Alanine Aminotransferase
ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

AST Aspartate Aminotransferase

BUN Blood Urea Nitrogen

CD40L Cluster of Differentiation 40 Ligand

CI Confidence Interval

CMI Cell-Mediated Immunity

CMV Cytomegalovirus

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

DLP Data Lock Point

eCRF electronic Case Report Form

eDiary electronic Diary

ELU/ml ELISA unit per milliliter

ELISA Enzyme-linked immunosorbent assay

EoS End of Study
ES Exposed Set

FDA Food and Drug Administration

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICS Intracellular Cytokine Staining

IDMC Independent Data Monitoring Committee

IFN-γ Interferon Gamma
IgG Immunoglobulin G

IL Interleukin

LL Lower Limit of the confidence interval

LLOQ Lower Limit Of Quantification

Mcg or µg Microgram

MedDRA Medical Dictionary for Regulatory Activities

### 208851 | Statistical Analysis Plan Amendment 2 17 Mar 2020 | TMF-1721000 | 2.0


208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

PBMC Peripheral Blood Mononuclear Cells

PCR Polymerase Chain Reaction

PD Protocol Deviation

pIMD Potential Immune-Mediated Disease

PPS Per Protocol Set
PT Preferred Term

qRT-PCR Quantitative Reverse Transcription Polymerase Chain Reaction

RSV Respiratory Syncitial Virus RTI Respiratory Tract Infection

SAE Serious adverse event
SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

TFL Tables Figures and ListingsTNF-α Tumor Necrosis Factor alpha

TOC Table of Content

UL Upper Limit of the confidence interval

WBC White Blood cells

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 14-JAN-2019 | first version | Final: 11 SEP 2018 |
| 27-JAN-2020 | Amendment 1: implement changes discussed at the KOM Dry-run and progress meetings | Final: 11 SEP 2018 |
| 17-MAR-2020 | Amendment 2: updates in CMI model notations following comments received by FDA | Final: 11 SEP 2018 |

### 2. STUDY DESIGN

Figure 1 Study design



BS S: Blood sample for safety (hematology/biochemistry)

BS H: Blood sample for humoral immune responses

BS C: Blood sample for cell-mediated immune responses (for CD4+/CD8+ and/or memory B-cell testing)

FU: Follow-up; PCR: Polymerase Chain Reaction

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- \* Visit 1 should take place no longer than 30 days after the Screening Visit. In case Visit 1 occurs more than 30 days after the Screening Visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection for safety laboratory assessment must be repeated (maximum one re-screening per subject is allowed). Only laboratory results from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF. Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. The subject can only be randomized once the investigator receives the results and confirms the eligibility criteria.
- \*\* In Part A, a first IDMC evaluation of safety data up to Day 31 based on all subjects (~12 per group or at least 8 per group in case of slow recruitment) will be performed before proceeding with administration of Dose 2 in Part A and Dose 1 in Part B. A second IDMC evaluation will be performed based on safety data up to Day 68 for all subjects. Part B of the study can only be initiated upon favorable outcome of the first IDMC safety evaluation in Part A.
- \*\*\* In Part B, a third and fourth IDMC evaluation of safety data up to Day 8 and Day 68, respectively, for the first enrolled and vaccinated subjects (~10 per group or at least 8 per group in case of slow recruitment) will be performed. Additional IDMC evaluations will happen during the conduct of the study.
- <sup>†</sup> In case of RTI symptoms during the RSV seasons (approximately from October to March), the subject will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab at the site. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- <sup>£</sup> Analysis 1 will be performed on all data collected up to Day 91 for at least primary and secondary endpoints based on both study parts (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). Analysis 2 will be performed when all safety data up to Month 8 (Visit 7) are available. The analyses will be based on data as clean as possible.
- **Experimental design:** Phase I/II, observer-blind, randomized, controlled, multicountry study with 2 parts (i.e., Part A in young adults aged 18-40 years with 4 parallel groups and Part B in older adults aged 60-80 years with 10 parallel groups).
- **Primary Completion Date (PCD):** last visit of the vaccination phase in Part B (Visit 6 [Day 91]).
- End of Study (EoS): Last testing results released of samples collected up to Visit 8 in Part B (Month 14) (for assays related to primary and secondary endpoints only).
- **Treatment allocation:** Subjects will be randomized using a centralised randomization system on internet (SBIR) on Day 1.

In Part A, the aim is to enrol approximately 48 subjects (~12 per group) aged 18-40 years. The randomization algorithm will use a minimisation procedure accounting for center and gender.

In Part B, the aim is to enrol approximately 700 subjects (~70 per group) aged 60-69 years and approximately 300 subjects (~30 per group) aged 70-80 years. The randomization algorithm will use a minimisation procedure accounting for age, center and gender in each step.

### • Study groups:

For the investigational RSV vaccines in Part A and Step 1 in Part B, the RSVPreF3 high-dose formulation containing 120  $\mu$ g RSVPreF3 will be used to prepare the vaccines for all dose groups (i.e., 30  $\mu$ g, 60  $\mu$ g and 120  $\mu$ g dose groups). For Step 2 in Part B, the RSVPreF3 low-dose and mid-dose formulations (containing 30  $\mu$ g and 60  $\mu$ g RSVPreF3, respectively) will be used for the groups receiving 30  $\mu$ g and 60  $\mu$ g of RSVPreF3, respectively, and the RSVPreF3 high-dose formulation will be used for the 120  $\mu$ g dose groups. As the reconstitution methods for the vaccines

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

administered to subjects enrolled in Step 1 and 2 of Part B will be different, separate study groups have been identified (referred to as B1 and B2). Throughout this document, the combined groups for Steps 1 and 2 are mentioned when referring to the number of groups in Part B (10 groups).

- Control: placebo.
- **Vaccination schedule:** Two vaccine doses administered intramuscularly at Day 1 and Day 61.
- **Blinding**: observer-blind.

The vaccination phases of each study part (Epoch 002) will be observer-blind. A first statistical analysis will be performed on data available up to one month post-Dose 2 (Visit 6, Day 91). Given that summary safety results may unblind some specific subjects, the persistence phase of Part B (Epoch 003) will be considered as single-blind with subjects remaining blinded up to study end (Visit 8 [Month 14]). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

- RTI surveillance in Part B: Active and passive surveillance will only be carried out during RSV seasons (approximately from October to March) throughout the entire Part B of the study:
  - Active surveillance: study participants will be contacted by the investigator/study staff every 2 weeks to identify if they experience an RTI.
  - Passive surveillance: study participants are instructed to contact the investigator/study staff as soon as they experience an RTI.

At the beginning of RSV seasons, study participants will be reminded of the start of the RTI surveillance.

### • Sampling schedule:

### In Part A:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the electronic Case Report Form (eCRF). The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for cytomegalovirus (CMV) status determination will be drawn from all subjects.
- Blood samples for safety assessment (hematology/biochemistry) will be drawn from all subjects on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- Blood samples for humoral immunogenicity and cell-mediated immunity (CMI) testing will be drawn from all subjects at Days 1, 31, 61 and 91 (Visits 1, 3, 4 and 6).

### In Part B:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF. The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for CMV status determination will be drawn from all subjects.
- **Blood samples for safety assessment** (hematology/biochemistry) will be drawn from all subjects and on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).
- **Blood samples for humoral immunogenicity and CMI** testing will be drawn from all subjects at Days 1, 31, 61, 91, Month 8 and Month 14 (Visits 1, 3, 4, 6, 7 and 8).
- Nasal/throat swabs: In case of RTI symptoms during the RSV season (approximately from October to March), the study participants will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab by qualified staff from the study team. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- **Type of study:** self-contained.
- **Data collection:** eCRF. Solicited symptoms will be collected using an electronic subject Diary (eDiary). Unsolicited symptoms will be collected using a paper subject Diary.
- **Safety monitoring:** The study will be conducted in 2 parts with oversight by an IDMC. The investigator is not permitted to start vaccinating the subjects in the next step in each part until receipt of the favorable outcome of the respective safety evaluations by the IDMC.
  - Part A: Approximately 48 young adults aged 18-40 years will be enrolled and vaccinated with the first dose. If the IDMC evaluation on data up to 30 days post Dose 1 is favorable, the Part A study participants will be vaccinated with the second dose and Part B of the study will be initiated.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Part B: This part will be conducted in a 2-step staggered design to ensure maximum safety of the participating subjects. In Step 1, approximately 100 subjects will be enrolled and vaccinated. Safety evaluations based on unblinded data from those first 100 subjects will be performed by the IDMC to allow the start of Step 2. In Step 2, the remaining study participants (N≅900) will be recruited and vaccinated.

In total, 6 IDMC meetings for safety evaluation are foreseen in the vaccination phase of the study (Epoch 002), i.e., 2 meetings in Part A and 4 meetings in Part B.

During the persistence phase of Part B (Epoch 003), 2 IDMC meetings will be planned with an interval of approximately 6 months.

If any safety concern is identified by the investigator or the sponsor, *ad-hoc* safety evaluations by the IDMC may be performed.

Analysis planned for IDMC evaluations are described in a separate document (SAP for IDMC).

### • Group description for analysis:

For analysis based on subjects in Part A and Part B Step 1 (B1), the group labels listed in table below will be used in the TFLs.

For final analysis based on subjects from Part B Steps 1 and 2, the groups will be pooled (B1 and B2) and the Pooled group labels will be used in the TFLs.

Table 1 Groups description

| Group label in tables | Group definition for footnote | Pooled<br>Group label<br>in tables | Pooled Group definition for footnote |
|---|---|---|---|
| 30-PLAIN_A | subjects receiving<br>unadjuvanted 30 mcg<br>RSVPreF3 in Part A | NA | |
| 60-PLAIN_A | subjects receiving<br>unadjuvanted 60 mcg<br>RSVPreF3 in Part A | NA | |
| 120-<br>PLAIN_A | subjects receiving<br>unadjuvanted 120 mcg<br>RSVPreF3 in Part A | NA | |
| Placebo_A | subjects receiving Placebo in Part A | NA | |
| 30-<br>PLAIN_B1 | subjects receiving<br>unadjuvanted 30 mcg<br>RSVPreF3 in Part B Step 1 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |
| 30-<br>PLAIN_B2 | subjects receiving<br>unadjuvanted 30 mcg<br>RSVPreF3 in Part B Step 2 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| 0 | Statistical Analysis Plan Amendment | | |
|---|---|---|---|
| Group label in tables | Group definition for footnote | Pooled<br>Group label<br>in tables | Pooled Group definition for footnote |
| 60-<br>PLAIN_B1 | subjects receiving<br>unadjuvanted 60 mcg<br>RSVPreF3 in Part B Step 1 | 60-PLAIN_B | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B |
| 60-<br>PLAIN_B2 | subjects receiving<br>unadjuvanted 60 mcg<br>RSVPreF3 in Part B Step 2 | 60-PLAIN_B | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B |
| 120-<br>PLAIN_B1 | subjects receiving<br>unadjuvanted 120 mcg<br>RSVPreF3 in Part B Step 1 | 120-<br>PLAIN_B | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B |
| 120-<br>PLAIN_B2 | subjects receiving<br>unadjuvanted 120 mcg<br>RSVPreF3 in Part B Step 2 | 120-<br>PLAIN_B | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B |
| 30-<br>AS01E_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 1 | 30-AS01E_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 30-<br>AS01E_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 2 | 30-AS01E_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 60-<br>AS01E_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 1 | 60-AS01E_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 60-<br>AS01E_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 2 | 60-AS01E_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 120-<br>AS01E_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 1 | 120-<br>AS01E_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 120-<br>AS01E_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B Step 2 | 120-<br>AS01E_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01E in Part B |
| 30-<br>AS01B_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 1 | 30-AS01B_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |
| 30-<br>AS01B_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 2 | 30-AS01B_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |
| 60-<br>AS01B_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 1 | 60-AS01B_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |
| 60-<br>AS01B_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 2 | 60-AS01B_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| Group label in tables | Group definition for footnote | Pooled<br>Group label<br>in tables | Pooled Group definition for footnote |
|---|---|---|---|
| 120-<br>AS01B_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 1 | 120-<br>AS01B_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |
| 120-<br>AS01B_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B Step 2 | 120-<br>AS01B_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with<br>AS01B in Part B |
| Placebo_B1 | subjects receiving Placebo in Part B Step 1 | Placebo_B | subjects receiving Placebo in Part B |
| Placebo_B2 | subjects receiving Placebo in Part B Step 2 | Placebo_B | subjects receiving Placebo in Part B |

For some of the comparison analyses in Part B, the RSV vaccine groups will be pooled according to their adjuvant content and the following group names will be used in the TFLs:

| Pooled Group label in tables | Pooled Group definition for footnote | Groups to be pooled |
|---|---|---|
| PLAIN_B | subjects receiving unadjuvanted RSVPreF3 in Part B (30, 60 or 120 μg) | 30_PLAIN_B1, 30_PLAIN_B2,<br>60_PLAIN_B1, 60_PLAIN_B2,<br>120_PLAIN_B1, 120_PLAIN_B2 |
| AS01E_B | subjects receiving RSVPreF3 adjuvanted with AS01E in Part B (30, 60 or 120 μg) | 30_AS01E_B1, 30_ AS01E _B2, 60_<br>AS01E _B1, 60_ AS01E _B2, 120_<br>AS01E _B1, 120_ AS01E _B2 |
| AS01B_B | subjects receiving RSVPreF3 adjuvanted with AS01B in Part B (30, 60 or 120 μg) | 30_AS01B_B1, 30_ AS01B_B2, 60_<br>AS01B_B1, 60_ AS01B_B2, 120_<br>AS01B_B1, 120_ AS01B_B2 |

For the analysis by age category, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 60-69Y | 60-69 years old subjects |
| 2 | 70-80Y | 70-80 years old subjects |

For the analysis by CMV status before vaccination, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | CMV+ | Subjects CMV positive before vaccination |
| 2 | CMV- | Subjects CMV negative before vaccination |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 3. OBJECTIVES/ENDPOINTS

# 3.1. Objectives

### 3.1.1. Primary objective

#### For Part A and Part B:

• To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccine administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

### 3.1.2. Secondary objectives

#### For Part A and Part B:

- To characterize the humoral immune responses (including dose-response) in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).
- To characterize the cell-mediated immune responses in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

#### For Part B:

- To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccines administered IM according to a 0, 2 month schedule, up to the end of follow-up (Month 14, Visit 8).
- To evaluate the occurrence of RSV-associated respiratory tract infections (RTI) during the RSV season in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.

### 3.1.3. Tertiary objectives

#### For Part A and Part B:

To further characterize the cell-mediated immune responses to investigational RSV vaccine formulations.

#### For Part B:

- To further characterize immune responses to investigational RSV vaccine formulations.
- To characterize persistence of immune responses to the investigational RSV vaccine formulations at Month 8 (Visit 7) and Month 14 (Visit 8).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- To further evaluate the occurrence of RSV-associated RTI (including co-infections with other respiratory viruses) during the RSV seasons in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.
- To evaluate the occurrence of RSV-associated RTI during the RSV season using self-collected nasal swabs.

### 3.2. Endpoints

### 3.2.1. Primary endpoints

#### For Part A and Part B:

- Occurrence of AEs from first vaccination up to 30 days after the second vaccination (Day 91):
  - Occurrence of each solicited local and general AE during a 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) after each vaccination.
  - Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.
  - Occurrence of any hematological (erythrocytes, WBC and differential count, platelets count and hemoglobin level) and biochemical (ALT, AST, creatinine, BUN and uric acid) laboratory abnormalities at Days 1, 8, 61 and 68.
  - Occurrence of all Grade 3 non-serious AEs (solicited and unsolicited) during the 30-day follow-up period after each vaccination.
  - Occurrence of SAEs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

#### For Part B only:

 Occurrence of pIMDs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

### 3.2.2. Secondary endpoints

#### For Part A and Part B:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), on the day of second vaccination (Day 61) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least
     2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro.

### For Part B only:

- Occurrence of RSV-associated RTI (as measured by qRT-PCR in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons, up to the end of follow-up.
- Occurrence of SAEs from Dose 1 up to the end of follow-up.
- Occurrence of pIMDs from Dose 1 up to the end of follow-up.

### 3.2.3. Tertiary endpoints

#### For Part A and Part B:

- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro.

# For Part B only:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype B in all subjects.
  - RSVPreF3 site 0 specific antibody concentrations in a subset of subjects who
    received the selected vaccine formulation or placebo.
- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific memory B-cells in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Persistence of the humoral immune response with respect to components of the investigational vaccine at Months 8 and 14:
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- Persistence of the cell-mediated immune response profile with respect to components of the investigational vaccine:
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro, in all subjects (Month 8) and in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo (Month 14).
  - Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least
     2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro, in all subjects (Month 8) and in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo (Month 14).
  - Frequency of RSVPreF3-specific memory B-cells at Month 14 in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Any further exploratory immunology to detect RSV-related immune responses, such as but not limited to:
  - Antibodies against specific protein F epitopes.
  - Potential new immunological markers for protection.
  - Cross-reactive neutralizing antibody titers against hMPV
- Occurrence of RSV-associated RTI, including co-infections with other respiratory viruses (as measured by multiplex PCR in self-collected nasal swab samples and nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons.
- Occurrence of RSV-associated RTI as measured by qRT-PCR in self-collected nasal swab samples during the RSV seasons, up to the end of follow-up.

#### 4. ANALYSIS SETS

# 4.1. Definition

### 4.1.1. Exposed Set

The Exposed Set (ES) will include all subjects with study vaccine administration documented

A safety analysis based on the ES will include all vaccinated subjects.

An immunogenicity analysis based on ES will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at Dose 1.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 4.1.2. Per-Protocol Set for analysis of immunogenicity

The Per-Protocol set (PPS) for analysis of immunogenicity will be defined by time point (and this to include all eligible subjects' data up to the time of important protocol deviations). The PPS will include all evaluable subjects in the ES:

- Meeting all eligibility criteria.
- For whom the administration route of the vaccine was as according to protocol.
- For whom the study vaccine was administered as per protocol.
- Who did not receive a concomitant medication/ product leading to exclusion from a PP analysis, as described in Section 6.6.2 of the protocol, up to the considered time point.
- Who did not present with a medical condition leading to exclusion from a PP analysis, as described in Section 6.7 of the protocol, up to the considered time point.
- Who complied with the vaccination schedule, as specified in the protocol.
- Who complied with the timings of the post-vaccination blood sampling for immune response evaluation, as specified in the protocol.
- For whom post-vaccination immunogenicity results are available for at least one assay component at the corresponding time points.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES.

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

### 4.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions.

For codes 1040, 1070, 1080, 1090, 2040, 2060, 2080: subjects will be eliminated from the time at which the condition is met onwards.

For codes 2090, 2100, 2120: subjects will be eliminated at the specific visit at which the condition is met.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

When applicable, codes will be allocated to subjects as long as they are included in the study. For example, withdrawals before the second dose will not be attributed a code 1070 because they missed a dose.

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 900 | Invalid informed consent or fraudulent data | All | All |
| 1030 | Study vaccine not administered at all | All | All |
| 1040 | <ul> <li>Administration of concomitant vaccine(s) forbidden in the protocol:</li> <li>Any investigational or non-registered vaccine other than the study vaccine used during the study period</li> <li>A vaccine not foreseen by the study protocol administered during the period starting 30 days before the first dose and ending 30 days after the last vaccine dose, except for inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after each vaccination.</li> </ul> | All | Immunology |
| 1050 | Randomisation failure | All | Immunology |
| 1060 | Randomisation code was broken | All | Immunology |
| 1070 | <ul> <li>Vaccination not according to protocol:</li> <li>Incomplete vaccination course</li> <li>Subject was vaccinated with the correct vaccine but containing a lower volume</li> <li>Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number)</li> <li>Route of the study vaccine is not intramuscular</li> <li>Wrong reconstitution of administered vaccine</li> </ul> | Vaccination<br>Visits 1 and 4 | Immunology |
| 1080 | Vaccine temperature deviation → vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation | Vaccination visits 1 and 4 | Immunology |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| | Statistical Analysis Flati American | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable<br>for analysis<br>set |
| 1090 | Expired vaccine administered | Vaccination visits 1 and 4 | Immunology |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | Immunology |
| 2040 | <ul> <li>Administration of any medication forbidden by the protocol</li> <li>Any investigational or non-registered medication used during the study period</li> <li>Immunosuppressants or other immune-modifying drugs administered chronically (i.e., more than 14 consecutive days in total) during the study period</li> <li>Long-acting immune-modifying drugs administered at any time during the study period</li> <li>Immunoglobulins and/or any blood products administered during the study period</li> </ul> | All | Immunology |
| 2060 | Intercurrent medical condition • Subjects may be eliminated from the PPS if, during the study, they incur a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status (other than RSV infection). | All | Immunology |
| 2080 | Subjects did not comply with vaccination schedule: • Part A: number of days between dose 1 and dose 2 is outside [55-80 days] • Part B: number of days between dose 1 and dose 2 is outside [55-75 days] | Visit 4 | Immunology |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| Statistical Analysis Plan Amend | | | |
|---|---|---|---|
| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable<br>for analysis<br>set |
| 2090 | <ul> <li>Subjects did not comply with blood sample schedule at a specific visit:</li> <li>Number of days between dose 1 and visit 3 blood sample is outside [30-37 days]</li> <li>Number of days between dose 1 and visit 4 blood sample is outside [55-80 days] for Part A or [55-75 days] for Part B</li> <li>Number of days between dose 2 and visit 6 blood sample is outside [30-37 days]</li> <li>Part B only:</li> <li>Number of days between dose 2 and visit 7 blood sample is outside [170-190 days]</li> <li>Number of days between dose 2 and visit 8 blood sample is outside [350-395 days]</li> </ul> | Visits 3, 4, 6, 7 and 8 | Immunology |
| 2100 | <ul> <li>Immunological results not available post-vaccination</li> <li>No immunological result at visit x for all 3 following tests: RSV A Neutralising antibody titer, RSVPreF3-specific IgG antibody concentration and RSVPreF3-specific CD4+ T cells frequency </li> </ul> | Visits 3, 4, 6, 7, 8 | Immunology |
| 2120 | Obvious incoherence or abnormality or error in data • Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at lab | Visits 1, 3, 4, 6, 7, 8 | Immunology |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 5. STATISTICAL ANALYSES

Note that standard data derivation rules and stat methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and stat methods will be described in section 9.

## 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at first vaccination in years, gender, race and ethnicity) will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (60-69 years and 70-80 years in Part B only).

Withdrawal status will be summarized by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PP analyses will be tabulated.
- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal.

### 5.1.2. Additional considerations

The analysis of demographic characteristics by group will be performed on the ES and on the PPS.

Demography and baseline characteristics will also be summarized by country.

Vital signs (heart rate, respiratory rate, systolic/diastolic blood pressure, pulse oximetry) and pre-vaccination temperature reported at visit 1 (Part A and Part B) will be summarized by group using descriptive statistics.

Subject disposition in the ES and PPS will be reported as a whole and per group, and for each age category (60-69 years and 70-80 years in Part B only).

Distribution of hematology and biochemistry parameters at baseline with respect to normal laboratory ranges will be tabulated by group.

For Part B only, the follow-up time in the study (in days) up to DLP for analysis or up to last contact will be described overall and by group using descriptive statistics.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# 5.2. Exposure

### 5.2.1. Analysis of exposure planned in the protocol

NA

#### 5.2.2. Additional considerations

The number of doses of study vaccines administered will be tabulated by group and by vaccine.

# 5.3. Immunogenicity

# 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be performed on the PPS for immunogenicity in Part A and Part B.

In Part B only: if in any study group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is at least 10%, a second analysis will be performed on the ES.

### 5.3.1.1. Within groups evaluation - humoral immune response

For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified):

### In Part A and Part B:

- Percentage of subjects above pre-defined threshold and their exact 95% CI will be tabulated.
- GMCs/GMTs and their 95% CI will be tabulated and represented graphically.
- Geometric mean of ratios of antibody titer/concentrations at each post-vaccination time point over pre-vaccination (Day 1) will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves.
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will be computed and tabulated using descriptive statistics.

### In Part B only:

• Individual post-vaccination results (at Days 31 and 91) versus pre-vaccination results (Day 1) will be plotted using scatter plots. Results of the placebo group will be used as a reference.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- Distribution of the fold increase of the antibody titers/concentrations (post- over prevaccination titers) will be tabulated.
- The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points.

The immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

The humoral immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

### 5.3.1.2. Within groups evaluation - Cell-mediated immune response

The following parameters will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI:

#### In Part A and Part B:

- Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, upon in vitro stimulation and background substracted, measured by ICS using PBMCs.
- Frequency of CD4+ and/or CD8+ T-cells expressing any combination of immune marker(s) among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs (see details in section 5.3.2.2).
- Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.

### In Part B only:

- Frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.
- Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

This will be displayed overall and by pre-vaccination category: <Q1, Q1-Q3, >Q3, where Q1/Q3 are respectively the 25<sup>th</sup> and the 75<sup>th</sup> percentiles of the results at pre-vaccination computed on pooled groups.

In addition, vaccine response in terms of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , will be explored and summarised by group.

The descriptive immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

The cell-mediated immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

### 5.3.1.3. Between groups evaluation (Part B only)

Statistical analyses will be performed to compare the 9 RSV investigational vaccine formulations in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

The between-groups analysis will be performed using an ANCOVA model, in several steps as follows:

- 1. The 9 RSV formulations will be first compared to the Placebo in order to identify groups whose means are significantly higher from the mean of the Placebo group, in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells at Day 31 and Day 91 (One-sided alpha=2.5%, Dunnett's adjustment test for multiplicity).
- 2. The effect of the second vaccination will be evaluated by comparing the means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31), of the groups pooled according to their adjuvant content (AS01<sub>B</sub>, AS01<sub>E</sub> and Plain), in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibody titers (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose).
  - Based on the results of this test, the next comparisons will be performed either at Day 91 or at Day 31.
- 3. Appropriate contrasts will be implemented to compare the RSV formulations as follows:
  - To demonstrate the adjuvant effect (on pooled groups according to their adjuvant content: AS01<sub>B</sub>, AS01<sub>E</sub>, Plain), by testing sequentially AS01<sub>B</sub> and AS01<sub>E</sub> versus Plain (One-sided alpha=2.5% for each superiority test: Adjuvant >Plain) in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibodies and, if applicable, by comparing AS01<sub>B</sub> vs AS01<sub>E</sub>.
  - To demonstrate linearity of increase in immune response when increasing the antigen dose in each adjuvanted group in terms of RSV-A neutralizing antibody and/or RSVPreF3-specific CD4+ T-cells.
  - Further ANCOVA t-tests would demonstrate superiority of 120 μg or 60 μg, should a quadratic effect be demonstrated.

Similar exploratory comparisons might also be performed on the RSVPreF3 ELISA antibody concentrations if deemed necessary.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 5.3.2. Additional considerations

# 5.3.2.1. Within groups – humoral immune response

- Correlations between assays of the humoral response will be investigated using scatter plots generated on pooled RSV groups in Part B:
  - RSVPreF3-specific IgG versus RSV A neutralizing antibody titer at each timepoint,
  - RSV A versus RSV B neutralizing antibody titer at Pre-vaccination and Day 91
  - RSVPreF3-specific IgG versus RSV-B neutralizing antibody titer at Prevaccination and Day 91

The same analysis will be performed on the fold increase post over pre-vaccination.

For each assay, values strictly below the cut-off and values strictly greater than the upper limit of quantification (ULOQ) will not be used for the scatter plots neither for the evaluation of the coefficients of correlation.

- The fold increase (post over pre-vaccination) of the RSVPreF3 IgG antibody concentrations versus the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will also be displayed graphically <u>by group</u> using scatter plots.
- The hMPV neutralizing antibody titers will also be tested at Day 1 and Day 91, on all subjects in Part A and on a subset of 40 subjects per group in Part B. The following analysis will be performed for each hMPV subtypes (A1, B1, A2, B2):
  - Percentage of subjects above pre-defined threshold and their exact 95% CI will be tabulated.
  - GMTs and their 95% CI will be tabulated and represented graphically.
  - Geometric mean of ratios of antibody titer at post-vaccination time point (Day 91) over pre-vaccination (Day 1) will be tabulated with 95% CI.
  - Antibody titer will be displayed using reverse cumulative curves.
  - Distribution of the fold increase of the antibody titers (post- over pre-vaccination titers) will be tabulated.
  - Individual post-vaccination results (Day 91) versus pre-vaccination results (Day 1) will be plotted using scatter plots for the selected RSV formulation and the placebo group as a reference.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 5.3.2.2. Within groups – Cell-mediated immune response

**Descriptive statistics** of the cell-mediated immune response will be tabulated and displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.

The RSVPreF3-specific CD4+/CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+/CD8+ T cells.

More specifically, the frequencies of RSVPreF3-specific CD4+ T cells expressing at least 2 cytokines [ $Freq^{2+}$ ] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}}$ 

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with medium only (background)

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with a pool of peptides covering RSVPreF3 (induction)

 $N_{Back/Ind}^{CD4}$  = Total number of CD4 T cells involved in the assay (background or induction)

Same computations will be done for all CMI responses that will be analysed, i.e.:

- Frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least 2 markers including at least 1 cytokine\* among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs.
  - \* cytokines are IL-2, TNF-\alpha, IFN-\gamma, IL-13, and IL-17
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IFN-γ (Th1-like response), as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IL-13 (Th2-like response), as measured by ICS using PBMCs.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- Frequency of RSVPreF3-specific CD4+/ CD8+ T-cells expressing at least IL-17 (Th17-like response), as measured by ICS using PBMCs.
- Co-expression profile: Frequency of RSVPreF3-specific CD4+ T-cells expressing any combination of marker(s) among CD40L, IL-2, TNF-α, IFN-γ, as measured by ICS using PBMCs, at Day 31 and Day 91 (→15 combinations).

**Vaccine response** in terms of RSVPreF3-specific CD4+ T cells frequencies expressing at least 2 markers among CD40L, IL-2, TNF-α, IFN-γ will be explored as follows:

Distribution of the fold increase: the percentage of subjects with at least a 2-fold,
 4-fold, 6-fold, 8-fold, 10-fold increase post-vaccination as compared to prevaccination (Post over Pre) will be tabulated by timepoint and by group.

For the computation of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 marker(s)** among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

#### 5.3.2.3. Between groups analysis

Statistical comparisons will be performed on the logarithm base 10 transformed results, in terms of RSV-A neutralizing antibody titers and frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

### a. Comparisons versus Placebo:

The 9 RSV formulations will be compared to the Placebo (control group) at Day 31 and Day 91 using an ANCOVA model with the Dunnett's adjustment method for multiplicity. The model will include the treatment group and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. Geometric mean ratios between groups and associated Dunnett's adjusted 95% CIs of the ratios will be tabulated.

The Dunnett's test is specifically designed for situations where all groups are to be compared against one "Reference" group. It is commonly used after ANCOVA has rejected the hypothesis of equality of the means of the distributions.

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test (where=(visit=D91));
CLASS treatmnt Adj agecat;
MODEL log(titer)=treatmnt baseline agecat / ddfm=KR DDFM=KR
outpm=pred_model cl;
REPEATED / group=Adj ; /* test homogeneity of variances and consider
different variance by adjuvant content if appropriate */
LSMEANS treatmnt / ALPHA=0.05 Adjust=Dunnett pdiff=control ("Placebo")
CL;
RUN;
```
208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### b. Comparisons between RSV groups:

The difference between RSV groups will be evaluated using an ANCOVA model including the adjuvant content (AS01B, AS01E, Plain), the antigen dose (30, 60, 120  $\mu$ g), the visit (Day 31, Day 91) and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. The adjuvant by antigen interaction will also be tested, and included in the model if significant at 10% (p-value <10%).

Based on this global model, appropriate contrasts will be used to perform the following comparisons:

1. Effect of the second vaccination:

The means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31) will be compared within each pooled group according to adjuvant content (AS01B, AS01E and Plain) (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose). Geometric mean ratios and associated 95% CIs will be tabulated.

## 2. Adjuvant effect:

The adjuvant effect will be tested sequentially as follow (One-sided alpha=2.5% for each superiority test):

- i. AS01B versus Plain
- ii. AS01E versus Plain
- iii. AS01B versus AS01E.

Geometric mean ratios and their 95% CIs will be computed for each comparison.

The same comparisons will also be performed by age category.

3. Antigen dose-response: test linear and quadratic effect of the antigen dose. Depending on significance of those 2 effects, ANCOVA t-tests might be done to demonstrate superiority of 120 µg or 60 µg.

Geometric mean ratios and their 95% CIs will be computed for each pairwise comparison within each adjuvant content family (120 µg vs 60 µg, 120 µg vs 30 µg, 60 µg vs 30 µg for Plain, AS01E and AS01B groups).

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test;
  class Adj(1B, 1E, PL) Ag(30, 60, 120) visit(PD1, PD2) subject agecat;
  model log(titer) = Adj Ag visit Adj*Ag Adj*visit Ag*visit Adj*Ag*visit
  baseline baseline*visit agecat / DDFM=KR S outpm=pred_model cl;
  REPEATED visit / SUBJECT=subject type=unr group=Adj;
  /* test homogeneity of variances and consider different variance by
  adjuvant content if appropriate */

  LSMEANS Adj*visit /E slice=visit CL PDIFF ALPHA=0.05; /*option E to see
  coefficients assigned to each effect */
  LSMEANS Adj*visit /E slice=Adj CL PDIFF ALPHA=0.05;
  LSMEANS Adj*Ag*visit / slice=visit CL PDIFF ALPHA=0.05;
  /* contrasts to be added for each comparison of interest */
  QUIT;
```

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

**The inferential analysis** on the RSVPreF3-specific CD4+ T cells will be performed on the log-transformation frequency of the CD4+ T cells expressing at least 2 markers (background or induction) computed by adding an offset of 0.5 cells to the number of activated CD4+ T cells (Delta method, see below). These transformations are deemed appropriate for further inferential analyses provided the incidence of activated CD4+ T-cells is below 4%.

Considering:

$$X_{ijk} = \log \left( \frac{n_{background}^{2+} + 0.5}{N_{Background}^{CD4}} \right), \text{ the log background frequency, and}$$

$$Y_{ijk} = \log \left( \frac{n_{lnduction}^{2+} + 0.5}{N_{lnduction}^{CD4}} \right), \text{ the log induction frequency}$$

As described for humoral response, the differences between RSV groups will be evaluated using an ANCOVA model including the adjuvant content (AS01B, AS01E, Plain), the antigen dose (30, 60, 120 µg), the visit (Day 31, Day 91) and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log-transformed CD4 T cell frequency following induction and the post-vaccination log-transformed CD4 T cell frequency under background condition as covariates.

All interactions will also be tested and included in the model if significant.

The following model will be used to analyse the log-transformed ratio between induction and background frequencies, and provide estimates of the RSVPreF3-specific CD4+ T cell frequency relative to background frequency. These estimates better represent the net effect of the vaccines over the CD4+ T cells frequency as the nuisance background frequency is subtracted from the induction frequency.

$$\begin{aligned} Y_{ijk} - x_{ijk} &= \mu_{jk} + \alpha_{j}.y_{i0k} + \beta.x_{ijk} + \varepsilon_{ijk}, \\ \widehat{Y}_{jk} - x_{ijk}\big|_{\bar{y}_0,\bar{x}} &= \mu_{jk} + \alpha_{j}.\bar{y}_0 + \beta.\bar{x}, \end{aligned}$$
 with

LS means conditional to  $\bar{y}_0$  and  $\bar{x}$ , where:

i, j, k=subject i, visit j, group k;  $\bar{y}_0$  = mean log induction frequency at pre-vaccination,

 $\bar{x}$  = mean log background after vaccination.

Note: This analysis is assuming that the background is the same for all groups and all timepoints. This assumption will be checked during the analysis.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

From that model, the least-squares means are then back-transformed into geometric means for the Induction / Background frequency ratio. The Background mean is then subtracted from the Induction mean and the fold-increase on that difference is calculated, as follows:

$$\hat{Z}_{jk} = 10^{\wedge} (\hat{Y}_{jk} - \overline{x}) - 1 = \frac{10^{\wedge} (\hat{Y}_{jk}) - 10^{\wedge} (\overline{x})}{10^{\wedge} (\overline{x})}$$
 and

$$Log(\hat{W}_{jk}) = Log\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right) = Log\left(\frac{10^{\wedge}(\hat{Y}_{jk_2}) - 10^{\wedge}(\bar{x})}{10^{\wedge}(\hat{Y}_{jk_1}) - 10^{\wedge}(\bar{x})}\right), \text{ where}$$

 $\hat{I}_{jk}$  = mean increase from background to induction frequency relative to background frequency at visit *j* for treatment *k*, and

 $\hat{W}_{jk}$  = vaccine effect on the antigen specific frequency following adjustment for background frequency.

The test and the 95% CIs for treatment comparisons will be calculated according to the delta method on the log-transformed ratio of RSVPref3-specific frequency relative to the background frequency estimates.

For each comparison, the covariance matrix of the means is pre multiplied and postmultiplied by the vector of partial derivative to provide the variance of the contrast:

$$Var\left(Log_{10}\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right)\right) = T\left(\nabla_{\hat{Y}_{jk_1},\hat{Y}_{jk_2}}(\bullet)\right) \cdot \sum \cdot \nabla_{\hat{Y}_{jk_1},\hat{Y}_{jk_2}}(\bullet)$$

Where

 $\sum$  is the covariance matrix, and

$$\nabla_{\hat{Y}_{jk}1,\hat{Y}_{jk2}}(\bullet) = \nabla_{\hat{Y}_{jk1},\hat{Y}_{jk2}}\left(Log_{10}\left(\frac{\hat{Z}_{jk2}}{\hat{Z}_{jk1}}\right)\right) = \begin{pmatrix} -1 - \frac{1}{\hat{Z}_{jk1}} \\ 1 + \frac{1}{\hat{Z}_{jk2}} \end{pmatrix}$$

The  $Log10(W_{jk})$  confidence interval is calculated based on the T-student percentile using the degrees of freedom provided by the MIXED procedure for the difference of means under consideration (eg  $Y_{jk2}$  and  $Y_{jk1}$ ) and the standard error calculated above.

$$Log_{10}\left(LowerCI\left(W_{jk}\right)\right) = Log_{10}\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right) - TINV(1 - alpha/2, df) \bullet \left[Var\left(Log_{10}\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right)\right) + TINV\left(\frac{1}{2} - alpha/2\right)\right]$$

The confidence intervals are then back-transformed to the original units to provide the confidence intervals for  $W_{jk}$ . (Amendment 2 – 17 MAR 2020).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 5.4. Analysis of safety and reactogenicity

## 5.4.1. Analysis of safety and reactogenicity planned in the protocol

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for Grade 3 non-serious AEs.

The percentage of subjects with any AE (solicited and unsolicited) resulting in a medically attended visit during the 30-day follow-up period will also be tabulated after each dose and overall.

The percentage of subjects reporting each individual solicited local AE (any grade and Grade 3) and solicited general AE (any grade, Grade 3, any related and Grade 3 related) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.

For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall. Similar tabulations will be performed for any fever with a causal relationship to vaccination and for Grade 3 (> 39.0°C/102.2°F) causally related fever.

For each group and for each hematology and biochemistry parameter:

- The percentage of subjects having hematology and biochemistry results below or above the laboratory normal ranges will be tabulated by time point.
- The summary of grading post-vaccination will be tabulated versus baseline. (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX C in the protocol. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

The percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

The percentage of subjects with at least one report of SAE classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. SAEs will also be described in detail.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

For Part A only, pregnancy and pregnancy outcomes will be listed (if applicable).

For Part B only, the percentage of subjects with at least one pIMD classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. PIMDs will also be described in detail.

The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall.

The analysis of safety will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years in Part B only).

#### 5.4.2. Additional considerations

All analyses will be descriptive and will be based on the Exposed Set (ES).

Compliance in completing solicited adverse events information will be tabulated after each dose and overall.

The percentage of subjects with at least **one local solicited** AE, with at least **one general solicited** AE and with **any solicited** AE during the 7-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, and for Grade 3 AEs considered related to vaccination.

The number of days with solicited symptoms reported during the **7-day follow-up period** will be tabulated for each solicited adverse event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).

The same tabulation will be done for Grade 3 symptoms, and also during **the whole post-vaccination period** (to include the total number of days for symptoms ongoing beyond the follow-up period).

The incidence of each solicited symptom (any grade and grade 3) will also be represented graphically per group and per dose.

Analysis of solicited symptoms will also be done:

- on the **pooled groups according to adjuvant content** (AS01B, AS01E, Plain), overall and by age category.
- On symptoms reported during the 4-day period, i.e. on the day of vaccination and 3 subsequent days, for each group after each dose and overall.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### 5.4.2.1. Solicited Adverse Events

Solicited adverse events will be reported daily during the 7-day (from Day 1 to Day 7) follow up period after each vaccination, using structured diaries. Missing or non-evaluable measurements will not be replaced.

In order to summarize the data, the maximum intensity of local injection site redness/swelling (in mm) and fever (in °C) will be categorized as follows:

| Grading | Redness/swelling | Fever |
|---------|------------------|-----------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C (100.4°F) - ≤ 38.5°C (101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C (101.3°F) - ≤ 39.0°C (102.2°F) |
| 3: | > 100 mm | > 39.0°C (102.2°F) |

Fever is defined as temperature  $\geq 38.0^{\circ}\text{C} / 100.4^{\circ}\text{F}$  (regardless of the location of measurement). The preferred location for measuring temperature in this study will be the oral cavity. Body temperature will also be summarized by 0.5°C increments as follows:  $\geq 38.0, >38.5, >39.0, >39.5, >40.0$ °C.

Each subject's data will be summarized according to the maximal severity observed during the follow-up period for each adverse event and each dose, followed by a summary across subjects and across doses.

#### 5.4.2.2. Unsolicited Adverse Events

When an unsolicited adverse event occurs more than once for a subject, the maximal severity and strongest relationship to the vaccine group will be counted. The selection of unsolicited AEs reported during the follow-up period will be done using the day of onset.

The analysis of unsolicited adverse events includes the following categories:

- Any unsolicited adverse event.
- Possibly related unsolicited adverse events.
- Grade 3 unsolicited adverse events
- Grade 3 possibly related unsolicited adverse events.
- Serious adverse events (SAEs)
- Possibly related SAEs.
- Potential Immune-Mediated disease (pIMDs, in Part B only)
- Medically attended adverse events

SAEs and pIMDs reported during the entire study period will be tabulated.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

In addition, the following time periods will be considered to report SAEs/pIMDs at the first and second analyses (E1 02 and E1 03, see section 7.1):

- from Dose 1 up to 30 days post dose 2 (or up to 90 days post dose 1 for subjects who did not received the second dose)
- from Dose 1 up to 6 months\* post dose 2 (or up to 8 months\* post dose 1 for subjects who did not received the second dose).
- From Dose 1 up to Data lock point, in order to report all SAEs/pIMDs reported at the time of analysis.

Listing of AEs/SAEs leading premature withdrawal from study or to interruption of vaccination will be described in detail.

#### 5.4.2.3. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes:

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10015150 | Erythema |
| Swelling | 10053425 | Swelling at injection site |
| Fatigue | 10016256 | Fatigue |
| Fever | 10016558 | Fever |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Headache | 10019211 | Headache |
| Myalgia | 10028411 | Myalgia |
| Shivering | 10040558 | Shivering |
| Arthralgia | 10003239 | Arthralgia |

For clintrial gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

<sup>\*</sup> months will be converted in days in order to select the events for the output tables.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 5.4.2.4. Clinical Safety Laboratory Investigations

In case of invalid or missing results or clinically significant grade 3 and above abnormal laboratory findings, a repeat testing may be done to confirm the first result (see Protocol section 7.1.4). For the analysis, the following rules will be applied:

- In general, the first result will be considered, except if this result is missing.
- In case of retesting for a grade 3 at pre-vaccination, the retesting will be considered if the result is < grade 3.</li>
- If result at Visit 1 is missing, the result of the screening will be used as baseline in the analysis.

#### 5.4.2.5. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

## 5.5. Analysis of RTI for Part B

## 5.5.1. Analysis of RTI planned in the protocol

The analysis will be performed on the ES.

Any RTI episode for which a visit for the assessment of potential RSV-RTI has been performed (with nasal/throat swab sampling) will be considered for the analysis. The assessment of RSV infection will be performed using qRT-PCR on nasal/throat swabs separately for samples collected by the subject and those collected by an appropriately qualified person (i.e., medical or nursing) at the assessment visit.

The proportion of subjects with at least one RSV-associated RTI (with 95 % CI) will be calculated by group.

Descriptive analyses (mean, median, min, max) of viral load assessed by quantitative PCR (RSV-A/B) of RSV-RTI will be performed by study group.

The incidence rate of all-cause RTI (with 95% CI) will be calculated by group. These will also be presented by co-infection identified by multiplex PCR.

#### 5.5.2. Additional considerations

The mean viral load of the RSV positive-RTI samples will also be reported by collection method (at assessment visit or at home) and by collection time (0-2, 3-4, >4 days between RTI onset date of symptoms and collection date).

Information collected at assessment visit will be described for RSV RTI episodes versus Non-RSV RTI episodes, as tested by qRT-PCR on nasal/throat swabs collected at assessment visit. It will include: vital signs, clinical symptoms, self-collected nasal swab result, medically attended visit and SAE related to the episode.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

RTI episodes will be described in detail in a listing. In addition, baseline RSV A Neutralizing antibody titer (GMT and 95% CIs) will be presented graphically by RTI episode status (RSV-RTI vs Non RSV-RTI vs No RTI).

## 6. ANALYSIS INTERPRETATION

All analyses will be descriptive with the aim to characterize the difference in safety/reactogenicity or immunogenicity between groups.

All comparisons will be exploratory. They should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons, except for the comparisons of all RSV formulations vs Placebo (Dunnett's adjustment).

## 7. CONDUCT OF ANALYSES

## 7.1. Sequence of analyses

The analyses will be performed stepwise:

- A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints up to Day 91 are available (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). This will include results from all subjects in Part A and Part B. This analysis will be considered as final for those endpoints. A clinical study report will be written.
  - At this point, the statistician will be unblinded (i.e., individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblind some specific subjects, the study will be considered as single-blind from this point onwards, with subjects remaining blinded up to study end (Visit 8, Month 14). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.
- A second analysis will be performed when all safety data up to Month 8 (Visit 7) are available (data as clean as possible). At this time, the following analyses will be performed:
  - The safety analysis of data up to 6 months post-Dose 2.
  - The analysis of all qPCR data available at that time.
  - The analysis of laboratory results that may become available at that time.
- A third immunogenicity analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 8 are available, to evaluate the persistence up to 6 months post-Dose 2 in Part B.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

• A fourth analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 14 (Visit 8) are available for the subjects enrolled in Step 1 of Part B. This analysis will include any additional laboratory results that may become available at that time.

No individual listings will be provided before the final end of study analysis.

• The final end of study analysis will be performed when all data for at least primary and secondary endpoints up to study conclusion are available (Month 14). All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage. An integrated clinical study report containing all available data will be written and made available to the investigators.

If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These data will be documented in annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=public posting, SR=study<br>report, internal) | Reference for TFL<br>TOC |
|---|---|---|---|
| Final analysis | E1_01 | SR, CTRS | See column A in TFL<br>TOC |
| Analysis up to<br>Day 91 | E1_02 | SR, CTRS | See column B in TFL<br>TOC |
| Analysis up to<br>Month 8 (safety<br>and PCR) | E1_03 | Internal | See column C in TFL<br>TOC |
| Analysis up to<br>Month 8<br>(immuno) | E1_04 | Internal | See column D in TFL<br>TOC |
| Analysis up to<br>Month 14 (Part B<br>Step 1) | E1_05 | Internal | See column E in TFL<br>TOC |

## 7.2. Statistical considerations for interim analyses

All confirmatory analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 8. CHANGES FROM PLANNED ANALYSES

## Statistical analyses

The fold-increase parameter for CMI (post over pre-vaccination) that will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI has been adapted as follows:

• *Fold increase (Post over pre-vaccination)* of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, *as measured by ICS using PBMCs*.

This analysis was also added for the Memory B cells:

• Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

All additional analysis planned compared to protocol are described in the "Additional considerations sections". The mains ones to be included in the CSR are also described below (changes indicated in bold):

- Demography and baseline characteristics will be summarized *by country*.
- Vital signs at baseline will be described by group using descriptive statistics.
- Exposure to study vaccine will be tabulated by group and by vaccine
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV neutralizing antibody titers will be reported for RSV-A *and RSV B*.
- Comparisons with Placebo will be done at Day 31 and Day 91, for both RSV A
  Neutralizing antibody and CD4+ T cells expressing at least 2 markers.
- Analyses of solicited symptoms were added: incidence of any/local/general solicited AEs, number of days with solicited AEs, analysis on pooled groups according to adjuvant content.
- RTI episodes: analysis of viral load by collection method and collection time was added, as well as the description of signs and symptoms for RSV-RTI vs Non-RSV RTI cases.
- Analysis of hMPV neutralizing antibody titers on all subjects in Part A and on a subset of subjects in Part B.

## Sequence of analyses

The wording of the 2<sup>nd</sup> analysis have been adapted as follows to allow the descriptive analysis of any additional immunogenicity results available for all subjects or for part of them:

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

- A second analysis will be performed when all safety data up to Month 8 (Visit 7) are available (data as clean as possible). At this time, the following analyses will be performed:
  - The safety analysis of data up to 6 months post-Dose 2.
  - The analysis of all qPCR data available at that time.
  - The analysis of laboratory results that may become available at that time.

## Sensitivity analysis

An issue in the randomization was identified on 23<sup>rd</sup> of July, and was identified as Significant Quality Issue (SQI) on the 6<sup>th</sup> of November 2019.

Randomization were performed in SBIR to create "placeholders"

- 1. For subjects whose eligibility was not yet confirmed
- 2. For subjects who were identified and whose ICF was not yet signed
- 3. For subjects not yet identified

This was not allowed neither based on the protocol, nor by consulting the central team.

As this issue might have an impact on the randomization, a sensitivity analysis will be performed excluding subjects who were randomized after the 23<sup>rd</sup> of July (randomization date >= 23JUL2019), for immunogenicity secondary endpoints at the time of first analysis (table template 17 and 22).

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1.

## 9.1. Handling of missing data

### 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - o If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - o If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.

- Adverse event start dates with missing day and month:
  - o If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - o If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 9.2. Duration of events

When a solicited AE is ongoing at the end of the solicited follow up period (Day 7), the following rules will be applied:

- If the event is present at Day 7 and information is available at each day up to the end of the event: count number of days with event up to last day reported
- If information is missing at several days between the first day with the event and the end of event: count missing days as days with an event (worst case scenario)
- For Grade 3 AEs: take into account the grading of the last day with AE reported (last observation carried forward)

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

## 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

## 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in section 9.1.

#### 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

## 10.1.2.3. Daily recording of solicited symptoms

#### 10.1.2.3.1. Studies with electronic diaries

For studies using electronic diaries for the collection of solicited symptoms, symptoms will be considered present only when a daily recording of grade 1 or more is present.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

#### 10.1.3. Data derivation

## 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

### 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) = 
$$((Temperature (Fahrenheit) - 32) \times 5)/9$$

Conversion of temperature from °Fahrenheit to °C will be performed according to SDTM specifications.

## 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | missing |

<sup>\*</sup>This rule will be used to computed descriptive statistics (GMTs, fold increase,etc). All values might be displayed in RCCs and scatter plots with individual results.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 10.1.3.4. Geometric mean titers (GMTs) and concentrations (GMCs)

Geometric Mean Titer (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Antibody titers or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the symptom reported at grade 1 or higher.

See also specific rules for ongoing symptoms in section 9.2.

## 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

#### 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal.

Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22.2% |
| 1/45 | 2.2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.

Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minima of transformed body temperatures will be displayed with one decimal.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 10.1.4.3. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

## 10.1.5. Statistical methodology

### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

## 10.1.5.2. Adjusted GMT or GMC ratios

When between-group GMT or GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

#### 10.2. TFL ToC

The TFL TOC provides the list of tables/figures/listings that will be generated at each analysis. It can be found in eTMF folder section 11.01.01.

The mock tables/figures referred under column named 'layout' can be found in section 12.

## 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 12. STUDY MOCK TFLS

The following drafted standard and study specific mocks will be used. Note that standard templates might be updated based on the last version of the standard catalogue used at the time of analysis. Titles and footnotes will be adapted accordingly.

The data display, title and footnotes are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

## 12.1. Demography

Template Table 1 Summary of demography and baseline characteristics (Exposed Set)

| | <each group=""></each> | | | Total |
|---|---|---|---|---|
| | N=XX | N=XXXX | | (XX |
| | Value or n | % | Value or n | % |
| Age (years) at first vaccination | | | | |
| N | XXX | | XXX | |
| Mean | XXX.X | | XXX.X | |
| Standard Deviation | XXX.X | | XXX.X | |
| Median | XXX.X | | XXX.X | |
| Minimum | XXX | | XXX | |
| Maximum | XXX | | XXX | |
| Sex | | | | |
| Male | XXX | XX.X | XXX | XX.X |
| Female | XXX | XX.X | XXX | XX.X |
| Ethnicity | | | | |
| <each ethnicity=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Race | | | | |
| <each race=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Age category | | | | |
| <each age="" category=""></each> | XXX | XX.X | XXX | XX.X |
| CMV status | | | | |
| Positive | XXX | XX.X | XXX | XX.X |
| Equivocal | XXX | XX.X | XXX | XX.X |
| Negative | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 2 Number of subjects by country and center (Exposed Set)

| | | <each group=""><br/>N=XXXX</each> | | Total<br>N=XXXX | |
|---|---|---|---|---|---|
| Country | Center-Investigator Name | n | % | n | % |
| <each country=""></each> | <each center-investigator="" name=""></each> | XXX | XX.X | XXX | XX.X |
| | All | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given center or country

 $% = (n/N) \times 100$ 

## Template Table 3 Number of subjects by study steps (Exposed Set)

| | | <each group=""><br/>N=XXXX</each> | | Total<br>N=XXXX |
|---------------|---|-----------------------------------|---|-----------------|
| Steps | n | % | n | % |
| Part A | | | | |
| Part B Step 1 | | | | |
| Part B Step 2 | | | | |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given category

 $% = (n/N) \times 100$ 

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 4 Summary of vital signs (Exposed Set)

| | | | <each group=""> N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| EACH VISIT> | Heart rate ( <unit>)</unit> | n | XXX | XXX |
| | , | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Respiratory rate ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Systolic Blood pressure ( <unit>)</unit> | n | XXX | XXX |
| | , , , | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Diastolic blood pressure ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Pulse oximetry ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Pre-vaccination Temperature (C) | n | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |

Short group label = long group label

N = total number of subjects

Value = value of the considered parameter

n = number of subjects in a given category

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 5 Summary of study completion with reason for withdrawal (Exposed Set)

| | <each group=""><br/>N=XXXX</each> | | Total<br>N=XXXX | |
|---|---|---|---|---|
| | n | % | n | % |
| Completed the study | XXX | XX.X | XXX | XX.X |
| Withdrawn from the study | XXX | XX.X | XXX | XX.X |
| Primary reason for withdrawal : | | | | |
| <each reason=""></each> | XXX | XX.X | XXX | XX.X |

Short group label = long group label

### Template Table 6 Summary of visit attendance (Exposed Set)

| | | | <each group=""><br/>N=XXXX</each> | | otal<br>XXXX |
|---|---|---|---|---|---|
| Visit | Status | n | % | n | % |
| <each visit=""></each> | Attended | XX | XX.X | XX | XX.X |
| | Did not attend yet | XX | XX.X | XX | XX.X |
| | Withdrawal at visit or earlier | XX | XX.X | XX | XX.X |
| | Did not attend | XX | XX.X | XX | XX.X |

Short group label = long group label

N = Number of subjects in each group or in total

n/% = number / percentage of subjects in a given category

## Template Table 7 Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set)

| Category | <each group=""><br/>N=XXX</each> | | | | Total<br>N=XXX | |
|---|---|---|---|---|---|---|
| Sub-category | Осс | n | % | Осс | n | % |
| At least one Important Protocol Deviation | | | | | | |
| < Each category > | | | | | | |
| <each sub-category=""></each> | | | | | | |

Short group label = long group label

N = Total number of subjects

Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects with important protocol deviations

# Template Table 8 Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set)

| | | Total<br>N= |
|-----------------------------------------------|---|-------------|
| | n | % |
| Withdrawals prior to randomization | | |
| <withdrawal 1="" reason=""></withdrawal> | | |
| <withdrawal 2="" reason=""></withdrawal> | | |
| Number of subjects included in randomized set | | |

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 9 Summary of subject disposition from Randomized Set to Exposed set (Randomized set)

| | | <each group=""><br/>N=XXXX</each> | | otal<br>XXXX |
|---|---|---|---|---|
| | n | % | n | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Exposed set | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

# Template Table 10 Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set)

| | | | | otal<br>XXXX |
|---|---|---|---|---|
| | n | % | n | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Per Protocol set at visit x | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 11 Summary of subject disposition from Exposed Set to End of study (Exposed set)

| | <each group=""> N=XXXX</each> | | | otal<br>XXXX |
|---|---|---|---|---|
| | n | % | n | % |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Number of subjects who completed the study | | | | |
| Completed with 1 dose | | | | |
| Completed with 2 doses | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

# Template Table 12 Deviations from protocol for age and intervals between study visits (Exposed set)

| Type of interval | | | <eacl< th=""><th>n group&gt;</th><th><each g<="" th=""><th>roup&gt;</th></each></th></eacl<> | n group> | <each g<="" th=""><th>roup&gt;</th></each> | roup> |
|---|---|---|---|---|---|---|
| | Interval range | | Value or n | % | Value or n | % |
| Age | <age range=""></age> | N | XXX | | XXX | |
| | | n | XXX | XX.X | XXX | XX.X |
| | | Minimum | XXX | | XXX | |
| | | Maximum | XXX | | XXX | |
| <each between<="" interval="" td=""><td><interval< td=""><td>N</td><td>XXX</td><td></td><td>XXX</td><td></td></interval<></td></each> | <interval< td=""><td>N</td><td>XXX</td><td></td><td>XXX</td><td></td></interval<> | N | XXX | | XXX | |
| study visit> | range> | | | | | |
| | | n | XXX | XX.X | XXX | XX.X |
| | | Minimum | XXX | | XXX | |
| | | Maximum | XXX | | XXX | |

## Template Table 13 Number of enrolled subjects by country

| | | <each group=""> N = XXX</each> | Total<br>N = XXX |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Country | <each country=""></each> | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 14 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults [18-64 years] | | |
| | Adults [65-84 years] | | |
| | Missing | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at study vaccination unknown

## Template Table 15 Minimum and maximum visit dates <analysis set name>

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit Description | Parameter | Date | Date | Date |
| < each informed consent> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| [Randomization] | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| <each visit=""></each> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |

Short group label = long group label

## 12.2. Exposure

## Template Table 16 Exposure to study vaccines by vaccine (Exposed Set)

| | | | group> | <each group<="" th=""></each> | |
|---|---|---|---|---|---|
| Vaccine administered | Number of subjects receiving | n | % | n | % |
| < Vaccine A> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Total number of doses | XXX | | XXX | |
| | administered during the study | | | | |
| < Each vaccine> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Total number of doses administered during the study | XXX | | XXX | |

Short group label = long group label

N = number of subjects in each group or in total included in the considered analysis set

n = number of subjects/doses in the given category

<sup>% =</sup> percentage of subjects in the given category

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## 12.3. Immunogenicity

## 12.3.1. Within groups

Template Table 17 Number and percentage of subjects with <antibody titer /concentration> equal to or above <cut-off unit> and <GMT/Cs> <analysis set name>

| | | | | >= | off u | nit | | GMT/C | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | 95% | 6 CI | | | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| <each antibody=""></each> | <each<br>group&gt;</each<br> | <each timing=""></each> | | | | | | | | | | |

Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

N = Number of subjects with available results

n/% = number/percentage of subjects with titer/concentration equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

MIN/MAX = Minimum/Maximum

Short timing label = long timing label

Template Figure 1 <GMT/Cs> and their 95% Cls for <antibody titers/concentrations> <analysis set name>



Short group label = long group label GMT/C = geometric mean antibody titer/concentration 95% CI = 95% confidence interval Short timing label = long timing label

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Note: This graph is provided as an example.

For RSV A Nab and RSVPreF3- specific IgG Ab, it will be adapted to display: all the groups (4 groups for Part A, 10 groups for Part B) and all available timepoints (4 TPs up to Day 91, 6 TPs up to study end for Part B). If needed for Part B, this graph might be split in several graphs: either by adjuvant content vs Placebo or by antigen content vs Placebo.

Same graph will be generated for RSV B NAb with 2 timepoints (10 groups, at Days 1 and 91), for RSVPreF3 site 0 Ab with 2 groups and 2 timepoints (selected formulation and Placebo groups, at Days 1 and 91), and for hMPV Nab (10 groups, at Days 1 and 91).

Template Table 18 Geometric mean of the individual ratio of <a href="fatters/concentrations">antibody titers/concentrations (units)> post-vaccination compared to pre-vaccination <Per Protocol Set></a>

| | | | | | | <gmt,c></gmt,c> | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 6 CI |
| Group | N | Time point | <gmt,c></gmt,c> | Time point | <gmt,c></gmt,c> | Ratio order | Value | LL | UL |
| | | description | | description | | | | | |
| <each< td=""><td>XXX</td><td>PI(D31)</td><td></td><td>PRE</td><td></td><td>PI(D31) / PRE</td><td></td><td></td><td></td></each<> | XXX | PI(D31) | | PRE | | PI(D31) / PRE | | | |
| group> | | , , | | | | , , | | | |
| | | <each point="" time=""></each> | | PRE | | <time point=""> / PRE</time> | | | |

Short group label = long group label

<GMT,C> = geometric mean antibody <titer,concentration>

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

Template Table 19 Distribution of <antibody titers/concentrations> fold increase post-vaccination compared to pre-vaccination <Per Protocol Set>

| | | | | <e< th=""><th>ach gr</th><th>oup&gt;</th><th></th><th></th><th><e< th=""><th>ach gr</th><th>oup&gt;</th><th></th></e<></th></e<> | ach gr | oup> | | | <e< th=""><th>ach gr</th><th>oup&gt;</th><th></th></e<> | ach gr | oup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95 | % CI | | | Ĭ | 95 | % CI |
| Antibody | Timing | FI | N | n | % | LL | UL | N | n | % | LL | UL |
| <each antibody=""></each> | <each timing=""></each> | < 1 | xx | xx | XX.X | xx.x | XX.X | xx | xx | XX.X | XX.X | XX.X |
| | | >= 1 | xx | xx | xx.x | xx.x | xx.x | xx | xx | XX.X | xx.x | xx.x |
| | | >= 2 | xx | xx | XX.X | xx.x | XX.X | xx | xx | XX.X | XX.X | XX.X |
| | | >= 4 | xx | XX | XX.X | XX.X | XX.X | xx | xx | XX.X | XX.X | XX.X |
| | | >= 6 | xx | ХХ | XX.X | xx.x | XX.X | хх | xx | XX.X | XX.X | XX.X |
| | | >= 8 | xx | ХХ | XX.X | xx.x | XX.X | хх | XX | XX.X | XX.X | XX.X |
| | | >= 10 | xx | XX | XX.X | xx.x | XX.X | XX | xx | xx.x | XX.X | XX.X |

Short group label = long group label

FI= Fold Increase post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with <titer, concentration> fold change meeting the specified criterion

95% CI = 95% confidence interval: LL = Lower Limit, UL = Upper Limit

Short timing label = long timing label

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 2 Reverse cumulative distribution curve of <antibody titers/concentrations> in the <group label> group <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: this graph is provided as an example. It will be generated by group, and will be adapted to display the 4 timepoints (PRE, D31, D61, D91) for the considered group. For Part B, same graphs will also be generated at Day 91 with groups according to adjuvant content or antigen content vs Placebo. If applicable, the upper limit of quantification will be presented (similarly to the cut-off).

For RSV B Nab ,RSVPreF3 site 0 specific Ab and hMPV NAb, the figure will display only 2 timepoints (Days 1 and 91).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 3 Kinetics of < antibody GMT/Cs> on subjects with results available at all timepoints up to <Day 91, Month 14> <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. Template will be adapted to display all the groups (10 groups for Part B) and all the timepoints (4 TPs up to Day 91, 6 TPs up to study end).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 4 Individual results of <RSV A Neutralizing antibody titer> at <time point> versus pre-vaccination in <group label> and Placebo B groups <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated as follows:

- RSV A Nab at Day 31 and Day 91, for each RSV groups (18 graphs)
- RSVPref3 IgG at Day 31 and Day 91, for each RSV groups (18 graphs)
- RSV B Nab at Day 91, for the selected formulation (1 graph)

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 5 Individual results of <RSV A versus RSV B Neutralizing antibody titer> at <time point> , on pooled RSV groups <Per protocol set>



Note: this graph is provided as an example. It will be generated on pooled RSV groups as follows:

- RSV A Nab vs RSVPreF3 IgG at each timepoint
- RSV A Nab vs RSV B Nab at Pre and Day 91
- RSV B Nab vs RSVPreF3 IgG at Pre and Day 91

Correlation coefficient will be computed on Log10 transformed data.

Raw data will be presented on Log10 axes.

The same graphs will be generated on fold increase Post over Pre.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 20 Geometric mean ratios of the fold increase (Pre to Post - vaccination) between RSVPreF3 IgG antibody concentrations and <RSV-A, RSV-B> neutralising antibody titers <Per protocol set>

| | | | | | | | | | GM | GM ratio of FI | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Timepoint | Group | N | RSVPref3 | 95 | % CI | <rsv-a, b=""></rsv-a,> | 9 | 5% | Value | LL | UL |
| - | - | | IgG GMF | LL | UL | Nab GMF | LL | UL | | | |
| PI(D31)/PRE | <each group=""></each> | | | | | | | | | | |
| <each timepoint=""></each> | | | | | | | | | | | |
| umepomiz | | | | | | | | | | | |

Short group label = long group label

N = Number of subjects with available results at the two considered time points (post and pre) for both RSVPreF3 IgG and <RSV-A, B> Nab

GMF = Geometric mean fold increase Pre to Post-vaccination

GM ratio of FI=Geometric mean ratio of fold increase (Pre to Post)

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

Template Figure 6 Individual results of the fold increase (post over prevaccination) of RSVPreF3 IgG antibody concentrations versus <RSV A, RSV B> neutralizing antibody titers at <time point> in <group label> <Per protocol set>



Short group label = long group label

Note: This graph is provided as an example. It will be generated as follows:

- Y axis=RSVPreF3 lgG vs X axis=RSV A Nab, at Days 31 and 91, for each RSV group (18 graphs)
- Y axis= RSVPreF3 IgG vs X axis=RSV B Nab at Day 91, for the selected formulation (1 graph)
- Axes will be in Log10.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 21 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immune Marker | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></at> | <each timing=""></each> | N | XXXX | XXXX |
| markers> | | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Note: this table will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC).

Template Table 22 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by pre-vaccination category <Per Protocol Set>

| | | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|---|
| Immune | Pre-vaccination status | | | | |
| Marker | | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<></td></at> | <q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<> | <each timing=""></each> | N | XXXX | XXXX |
| markers> | | | GM xx.x SD Minimum xx.x | XX.X | XX.X |
| | | | | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X |
| | | | Median | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X |
| | [Q1-Q3] | <each timing=""></each> | <each< td=""><td></td><td></td></each<> | | |
| | | | parameter> | | |
| | >Q3 | | | | |
| | Total | | | | |

Short group label = long group label

<Q1= subjects with pre-vaccination frequency < Q1 of the frequencies at pre-vaccination computed on pooled groups Q1-Q3= subjects with pre-vaccination frequency within [Q1-Q3] of the frequencies at pre-vaccination computed on pooled groups

>Q3=subjects with pre-vaccination frequency < Q3 of the frequencies at pre-vaccination computed on pooled groups N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25<sup>th</sup> and 75<sup>th</sup> percentiles

Short timing label = long timing label

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 7 Boxplots with individual data of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. Depending on the analysis, it will display groups and timepoints as follows:

- Part A: 1 graph with 4 groups and 3 (D1, D31, D91) or 4 timepoints (D1, D31, D61, D91)
- Part B: 3 graphs with 4 groups (either by adjuvant content or by antigen content vs Placebo), and 3 timepoints (D1, D31, D91) or 5 timepoints (up to Month 8) or 6 timepoints (up to Month 14, only for selected Ag dose and Placebo)

This graph will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC).

For Part B, the same graph will be generated for memory B-cells, with 4 groups (selected Ag dose with Plain/AS01E/AS01B, and Placebo) and 4 timepoints (PRE, D31, D91, M14).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 8 Frequency of RSVPreF3 specific CD4+ T-cells expressing any combination of markers among IL-2, CD40L, TNFa, IFNg in <group label> group at Day 31 and Day 91 (per million of CD4+ T cells, by ICS) <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated by group and will be adapted to display Q1-Median-Q3 for each combination of the markers (15) at Day 31 and Day 91.

Template Table 23 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immune Marker | Timing | Statistic | value | Value |
| <at 2<="" least="" td=""><td><each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each></td></at> | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each> | N | XXXX | Xxxx |
| markers> | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results at both timepoints (pre and post)

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 24 Descriptive statistics of the frequency of RSVPreF3 specificmemory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| Immuno assay | Timing | Statistic | <each group=""> value</each> | <each group=""> value</each> |
|---|---|---|---|---|
| | | Otatistic | value | value |
| Memory B cells | <each timing=""></each> | N | XXXX | XXXX |
| | | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Template Table 25 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| Immuno assay | Timing | Statistic | <each group=""> value</each> | <each group=""> value</each> |
|---|---|---|---|---|
| Memory B cells | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>XXXX</td></each> | N | XXXX | XXXX |
| , | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25<sup>th</sup> and 75<sup>th</sup> percentiles

Short timing label = long timing label
208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 26 Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | | <e< th=""><th>ach gr</th><th>oup&gt;</th><th></th><th></th><th><e< th=""><th>ach gr</th><th>oup&gt;</th><th></th></e<></th></e<> | ach gr | oup> | | | <e< th=""><th>ach gr</th><th>oup&gt;</th><th></th></e<> | ach gr | oup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | % CI | | | _ | | % CI |
| Assay | Timing | FI | N | n | % | LL | UL | N | n | % | LL | UL |
| <assay name=""></assay> | <each timing=""></each> | < 2 | xx | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 2 | xx | хх | XX.X | XX.X | XX.X | xx | xx | XX.X | XX.X | XX.X |
| | | >= 4 | xx | xx | XX.X | xx.x | xx.x | xx | xx | xx.x | XX.X | XX.X |
| | | >= 6 | xx | хх | XX.X | xx.x | xx.x | XX | XX | xx.x | XX.X | xx.x |
| | | >= 8 | xx | xx | XX.X | XX.X | XX.X | XX | xx | xx.x | XX.X | XX.X |
| | | >= 10 | xx | xx | XX.X | XX.X | XX.X | xx | xx | xx.x | XX.X | XX.X |

Short group label = long group label

FI= Fold increase Post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with fold increase meeting the specified criterion

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Short timing label = long timing label

#### 12.3.2. Between groups

Template Table 27 Comparisons of the 9 RSV formulations versus Placebo in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at one month post <dose 1 (Day 31), dose 2 (Day 91)> (ANCOVA model, Dunnett's test) – Part B <Per Protocol set>

| Assay | Timepoint | RSV group | N | GM <t,f> ratio</t,f> | Dunne | ett's 95% CI | Dunnett's |
|---|---|---|---|---|---|---|---|
| | | | | (RSV over Placebo) | LL | UL | p-value |
| <assay name=""></assay> | <day 31,="" 91="" day=""></day> | 30-PLAIN_B | | | | | |
| , | | 60-PLAIN_B | | | | | |
| | | 120-PLAIN_B | | | | | |
| | | 30-AS01E_B | | | | | |
| | | 60-AS01E_B | | | | | |
| | | 120-AS01E_B | | | | | |
| | | 30-AS01B_B | | | | | |
| | | 60-AS01B_B | | | | | |
| | | 120-AS01B_B | | | | | |

Short group label = long group label

N= Number of subjects with both pre- and post-vaccination results available

GM<T.F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

RSV Vaccine is considered superior to Placebo if one-sided p-value < 0.025

Dunnett's 95% CI = 95% confidence interval based on Dunnett's adjustment, LL = lower limit, UL = upper limit ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed

<titer,frequency> as covariate, and the treatment and age category as fixed effects

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 28 Comparisons of the mean responses post dose 2 (Day 91) versus post dose 1 (Day 31) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> on pooled groups according to adjuvant content (ANCOVA model) – Part B <Per Protocol set >

| Assay | RSV group | N | GM <t,f> ratio</t,f> | 95% | CI | p-value |
|---|---|---|---|---|---|---|
| | | | (D91/D31) | LL | UL | |
| <assay name=""></assay> | PLAIN_B | | | | | |
| | AS01E_B | | | | | |
| | AS01B_B | | | | | |

Short pooled group label = long pooled group label

N= Number of subjects with results available at both timepoints

GM<T,F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

PII D91 is considered as significantly higher to PI D31 if one-sided p-value <0.025

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance); LL = lower limit. UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the adjuvant content, antigen dose and age category as fixed effects

Template Table 29 Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) - Part B <Per Protocol set>

| | | | Group 1 | | | | | G | roup 2 | | | GM <t,f> ratio<br/>(Group 1 /<br/>Group 2)</t,f> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 5%<br>CI | | | | | 5%<br>CI | | 95% | CI | |
| | | Group 1 | N | GM <t,f></t,f> | LL | UL | Group 2 | N | GM <t,f></t,f> | | | Value | LL | UL | p- |
| Assay | Timepoint | - | | | | | | | | LL | UL | | | | value |
| <assay< td=""><td><each< td=""><td>AS01B_B</td><td></td><td></td><td></td><td></td><td>PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<></td></assay<> | <each< td=""><td>AS01B_B</td><td></td><td></td><td></td><td></td><td>PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | AS01B_B | | | | | PLAIN_B | | | | | | | | |
| name> | timing> | AS01E_B | | | | | PLAIN_B | | | | | | | | |
| | | AS01B B | | | | | AS01E B | | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance);

LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and adjuvant content, antigen dose and age category as fixed effects Group 1 is considered superior to Group 2 if one-sided p-value <0.025

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 30 Comparisons of the RSV groups (by antigen dose level) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) – Part B <Per Protocol set >

| | | | Group 1 | | | Gı | roup 2 | | GM <t,f<br>(Grou</t,f<br> | ) | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 5%<br>CI | | | | 5%<br>CI | | 95% | CI | |
| Assay | Timepoint | Group 1 | N | GM <t,f></t,f> | | Group 2 | N | GM <t,f></t,f> | | Value | | UL | p-value |
| <assay< td=""><td><each< td=""><td>120-</td><td></td><td></td><td></td><td></td><td>60-</td><td></td><td></td><td></td><td></td><td></td><td></td><td>_</td></each<></td></assay<> | <each< td=""><td>120-</td><td></td><td></td><td></td><td></td><td>60-</td><td></td><td></td><td></td><td></td><td></td><td></td><td>_</td></each<> | 120- | | | | 60- | | | | | | | _ |
| name> | timing> | PLAIN_B | | | | PLAIN_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | PLAIN_B | | | | PLAIN_B | | | | | | | |
| | | 60-PLAIN_B | | | | 30- | | | | | | | |
| | | | | | | PLAIN_B | | | | | | | |
| | | 120- | | | | 60- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 60- | | | | 30- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 120- | | | | 60- | | | | | | | |
| | | AS01B_B | | | | AS01B_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | AS01B_B | | | | AS01B_B | | | | | | | |
| | | 60- | | | | 30- | | | | | | | |
| | | AS01B_B | | | | AS01B_B | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance);

LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the treatment, age category and gender as fixed effects Group 1 is considered superior to Group 2 if one-sided p-value <0.025

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 31 Parameters of the ANCOVA model for the comparison between RSV groups in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg>- Part B <analysis set name>

| Timepoint | Variable | DF | <b>Fvalue</b> | p-value |
|---|---|---|---|---|
| <each timepoint=""></each> | Pre-vaccination log <titer, frequency=""></titer,> | | | |
| | Age category | | | |
| | Adjuvant | | | |
| | Antigen | | | |
| | Visit | | | |
| | Linear effect of antigen | | | |
| | Quadratic effect of antigen | | | |
| | Antigen*Adjuvant | | | |

Antigen = Antigen dose (3 levels: 30, 60, 120 mcg)

Adjuvant = Adjuvant content (3 levels: no adjuvant, AS01E, AS01B)

Antigen\*Adjuvant = interaction between antigen dose and adjuvant

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and adjuvant content, antigen dose and age category as fixed effects

DF = degrees of freedom

Interaction (Antigen \* Adjuvant) considered as statistically significant if p-value <0.100

Main factors (Pre-vaccination, antigen, adjuvant) considered as statistically significant if p-value <0.050 (model including interaction)

#### **12.4.** Safety

### Template Table 32 Compliance in completing solicited adverse events information (Exposed Set)

| | | <each group=""></each> | |
|------------------------|-----|------------------------|----------------|
| DOSE | N | n | Compliance (%) |
| Vaccination at Visit 1 | XXX | XXX | XX.X |
| Vaccination at Visit 4 | XXX | XXX | XX.X |
| TOTAL | XXX | XXX | XX.X |

Short group label = long group label

N=Number of administered vaccinations

n = number of vaccinations with solicited symptom information completed

Compliance (%) =  $(n / N) \times 100$ 

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 33 Incidence and nature of <grade 3> symptoms (solicited and unsolicited) <with causal relationship to vaccination> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis set name>

| | | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th></th><th></th><th>&lt;</th><th>Each g</th><th>roup&gt;</th><th></th></ea<> | ch gro | up> | | | < | Each g | roup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 6 CI | | | | 95 | % CI |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

#### For overall/subject:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

<sup>95%</sup> CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 34 Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <analysis set name>

| | | | <each group=""></each> | | | | | <each group=""></each> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | 6 CI | | | | 95 | 5% CI |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

#### Template Table 35 Incidence of solicited local symptoms reported during the 7day (Days 1-7) post-vaccination period following each dose and overall <analysis set name>

| | | | | | <e< th=""><th>ach g</th><th>roup&gt;</th></e<> | ach g | roup> |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| DOSE 1 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| DOSE 2 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/DOSE | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/SUBJECT | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### Template Table 36 Incidence of solicited general symptoms reported during the 7day (Days 1-7) post-vaccination period following each dose and overall <cohort name>

| | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|
| <b>D</b> | 0 | T | A.I | | 0/ | | 95 % CI |
| Oose 1 | Symptom | Type | N | n | % | LL | UL |
| OOSE 1 | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | iever> | Crada >0 | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OSE 2 | <each except<="" symptom="" td="" –=""><td>All</td><td></td><td></td><td></td><td></td><td></td></each> | All | | | | | |
| | fever> | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | - (0.2) | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| VERALL/DOSE | <each except<="" symptom="" td="" –=""><td>All</td><td></td><td></td><td></td><td></td><td></td></each> | All | | | | | |
| | fever> | Crade >2 | | | | | |
| | | Grade ≥2 | | - | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| | | | | | <e< th=""><th>ach gi</th><th>roup&gt;</th></e<> | ach gi | roup> |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OVERALL/SUBJECT | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | , | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 37 Number of days with < local/general > solicited symptoms during < the 7-day (Days 1-7), the whole > post-vaccination period < analysis set name >

| | | | <each group=""></each> |
|---|---|---|---|
| Dose | Symptom | Statistic | Value |
| DOSE 1 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| DOSE 2 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| OVERALL/DOS | E <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |

Short group label = long group label n = number of doses with the symptom

Q1 = 25th percentile

Q3= 75th percentile

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 9 Incidence of solicited <local, general> adverse events reported during the 7-day (Days 1-7) post-vaccination period following each dose <Exposed set>



Short group label = long group label

Note: this graph is provided as an example. It will be adapted to display the percentage of subjects reporting each local or general symptom, any grade and grade 3, by group and by dose. Template will be discussed at the time of the dry-run.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Table 38 Percentage of subjects reporting the occurrence of <grade 3> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> within the 30-day (Days 1-30) post-vaccination period <analysis set name>

| | | | | nch gro<br>N=XXX | - | | | ı | Total | X | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | - | | | | 95% | 6 CI | | | | 95% | 6 CI |
| Primary System Organ Class (CODE) | Preferred Term<br>(CODE) | n* | n | % | LL | UL | n* | N | % | LL | UL |
| | At least one symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XX.X | XX.X | XXX | Ххх | XX.X | XX.X | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

### Template Table 39 List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <Exposed set>

| Grou<br>p | Sub<br>. No | Countr<br>y | AE<br>Descriptio | SA<br>E | Causalit<br>y | Vaccinatio<br>n and visit | Type of discontinuation |
|---|---|---|---|---|---|---|---|

Short group label = long group label

## Template Table 40 Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment <analysis set name>

| | | | Age<br>at | |
|---|---|---|---|---|
| Group | Sub.<br>No. | Country | onset | Primary System<br>Organ Class |
| <each< td=""><td></td><td></td><td></td><td></td><td></td></each<> | | | | |
| group> | | | | |

| | Sub. | | | Day<br>of | | | | | 0.40.0 | pIMD<br>source |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | No. | Medical visit type | Dose | onset | Duration | Intensity | Causality | Outcome | | |
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | |
| group> | | | | | | | | | | |

Short group label = long group label

<sup>\*</sup> type of discontinuation refers to whether the discontinuation is a treatment discontinuation or study follow-up discontinuation

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### Template Table 41 Listing of SAEs <analysis set name>

| Group | Sub.<br>No. | Gender | Country | Race | Age at onset (Year) | Verbatim | Preferred Term |
|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | |
| group> | | | | | | | |

| Group | Primary System<br>Organ Class | Medical visit ty | pe Dose | Day<br>of<br>onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | |
| group> | | _ | | | | | | |

Short group label = long group label

### Template Table 42 Listing of pregnancies reported during the study period in Part A <analysis set name>

| Gro | Su | Count | Rac | Age at | Previo | LM | Days | Age | Date | Pregna | Date | Gestational |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| up | b. | ry | е | vaccinat | us | Р | betwe | at | of | ncy | of | weeks at |
| | No. | | | ion | Dose | dat | en | delive | delive | Outcom | outco | birth/miscarr |
| | | | | | | е | LMP- | ry | ry | е | me | iage |
| | | | | | | | vacc | (Year) | | | | /termination |

Short group label = long group label LMP=Last Mentrual Period

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 43 Number and percentage of subjects taking concomitant medication during the <XX>-day (Days 1-<XX>) post-vaccination period by dose and overall <analysis set name>

| | | <each group=""> <eacl< th=""><th><each< th=""><th colspan="3">h group&gt;</th></each<></th></eacl<></each> | | | | | <each< th=""><th colspan="3">h group&gt;</th></each<> | h group> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | <95 | >% CI | | | | <95 | >% CI |
| Dose | | N | n | % | LL | UL | N | N | % | LL | UL |
| DOSE x | Any | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = total number of subjects with the corresponding administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified type of concomitant medication was taken at least once during the considered period

For overall/subject:

N = total number of subjects with at least one administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

### Template Table 44 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges, 7 days post dose <1, 2> <analysis set name>

| | | | <ea< th=""><th>ach gro</th><th>up&gt;</th><th colspan="4"><each group=""></each></th></ea<> | ach gro | up> | <each group=""></each> | | |
|---|---|---|---|---|---|---|---|---|
| Laboratory parameter | Range indicator at<br>Baseline (PRE) | Range<br>indicator at<br>post-<br>vaccination | N | n | % | N | n | % |
| <each parameter=""></each> | UNKNOWN | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | BELOW | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | WITHIN | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | ABOVE | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |

Short group label = long group label

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

Baseline= Pre-vaccination at <Day 1, Day 61>

Post-vaccination= Post vaccination at <Day 8, Day 68>

## Template Table 45 Summary of hematology and biochemistry results by grade at 7 days post dose <1, 2 > versus baseline (<Day 1, Day 61>) <analysis set name>

| | | | <ea< th=""><th>ch gro</th><th>oup &gt;</th></ea<> | ch gro | oup > |
|---|---|---|---|---|---|
| Laboratory parameter | Baseline | Post-vaccination | N | n | % |
| <each parameter=""></each> | Unknown | Unknown | | | |
| | | <each grade=""></each> | | | |
| | <each grade=""></each> | Unknown | | | |
| | | <each grade=""></each> | | | |
| | Total | Unknown | | | |
| | | <each grade=""></each> | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Baseline= Pre-vaccination at <Day 1, Day 61>

Post-vaccination = Post vaccination at <Day 8, Day 68>

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Note: Templates 45 and 46 will be generated post dose 1 with results at Visit 2 (Day 8) versus baseline at Day 1, and post dose 2 with results at Visit 5 (Day 68) versus baseline at Day 61.

Template Table 46 Summary of hemoglobin change from baseline at 7 days postdose <1, 2> (Exposed set)

| | | <ea< th=""><th colspan="4"><each gro<="" th=""></each></th></ea<> | <each gro<="" th=""></each> | |
|---|---|---|---|---|
| Laboratory parameter | | N | n | % |
| Hemoglobin - change from baseline | UNKNOWN | | | |
| Ç Ç | GRADE 0 | | | |
| | GRADE 1 | | | |
| | GRADE 2 | | | |
| | GRADE 3 | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period

n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Note: This table will be generated post dose 1 with results at Visit 2 (Day 8) and Day 1 as baseline, and post dose 2 with results at Visit 5 (Day 68) and Day 61 as baseline.

Template Figure 10 Boxplot of <each hematology/biochemistry parameter> (Exposed Set)



Note: This graph is given as an example. It will be adapted to display one boxplot per group and per timepoint, all timepoints available (5 TPs: Screening, Days 1, 8, 61, 68). For Part A, one graph will be generated displaying the 4 groups. For Part B, 3 graphs will be generated displaying 4 groups: 3 RSV groups (30/60/120 -Plain, - AS01E or - AS01B) and the Placebo group.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 47 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis set name>

| | | | ch gr<br>N=XX) | - | <each group<br="">N=XXXX</each> | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

## Template Table 48 Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis set name>

| | | | <eacl< th=""><th>n group</th><th>&gt;</th><th><each< th=""><th>n group&gt;<br/>XX</th><th>•</th></each<></th></eacl<> | n group | > | <each< th=""><th>n group&gt;<br/>XX</th><th>•</th></each<> | n group><br>XX | • |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System<br>Organ Class (CODE) | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Fatal SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related Fatal | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| SAE | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

N = number of subjects with administered dose

n/% = number/percentage of subjects reporting the symptom at least once

n\* = Number of events reported

Related = assessed by the investigator as related

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### 12.5. Analysis of RTI

Template Table 49 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis set name>

| | | | <each group=""></each> | | | ıp> | Tota | | | al | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI | | | | | 95% | 6 CI | | | |
| Samples | RSV status | N | ı | n % | 6 | LL | UL | N | n | % | LL | UL |
| Nasal/throat swab at assessment visit | RSV+ | | | | | | | | | | | |
| | RSV- | | | | | | | | | | | |
| | All | | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by qRT-PCR at least once

RSV-= subjects tested as RSV negative by qRT-PCR

All= subjects with at least one gRT-PCR result available

N = number of subjects in each group or in Total

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template Table 50 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis set name>

| | | | <ea< th=""><th>ach</th><th>gro</th><th>up&gt;</th><th colspan="3">Tota</th><th>ıl</th><th></th></ea<> | ach | gro | up> | Tota | | | ıl | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95% | δCI |
| Samples | RSV status | N | n | % | LL | UL | N | n | % | LL | UL |
| Nasal swab at home | RSV+ | | | | | | | | | | |
| | RSV- | | | | | | | | | | |
| | All | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by qRT-PCR at least once

RSV-= subjects tested as RSV negative by qRT-PCR

All= subjects with at least one qRT-PCR result available

N = number of subjects in each group

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

## Template Table 51 Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <Exposed set>

| | | | RSV A + | | | | RS | V B + | |
|---|---|---|---|---|---|---|---|---|---|
| Days after<br>RTI onset | Swab | N | n | % | mean | N | n | % | mean |
| 0-2 | Nasal swab at home<br>Nasal/throat swab at assessment<br>visit | | | | | | | | |
| 3-4 | Nasal swab at home<br>Nasal/throat swab at assessment<br>visit | | | | | | | | |
| >4 | Nasal swab at home<br>Nasal/throat swab at assessment<br>visit | | | | | | | | |

Days after RTI onset = number of days between start of RTI symptoms and collection date

N=Number of swabs with gRT-PCR results available

n/%= number/percentage of swabs tested as RSV A/B positive by qRT-PCR

mean= mean of the viral load computed on RSV A/B positive swabs

Template Table 52 Descriptive statistics of the viral load of the RSV- confirmed RTI episodes, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <at home> <Exposed Set>

| | | <each group=""><br/>N=</each> | Total<br>N= |
|---------|------------|-------------------------------|-------------|
| Туре | Parameters | Value | Value |
| RSV A + | n | | |
| | Mean | | |
| | Min | | |
| | Q1 | | |
| | Median | | |
| | Q3 | | |
| | Max | | |
| RSV B + | | | |
| All RSV | | | |
| + | | | |

Short group label = long group label

RSV A+= RSV A positive samples by gRT-PCR

RSV B+-= RSV B positive samples by qRT-PCR

All RSV += All RSV positive samples by qRT-PCR

N = Number of swabs with qRT-PCR results available

n= number/percentage of samples in each category

Q1 and Q3 = 25th and 75th percentiles

Min/Max = Minimum/Maximum

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

# Template Table 53 Number and percentage of subjects reporting co-infections with respiratory viruses, as measured by multiplex PCR on RSV A/B positive RTI samples collected <at assessment visit, at home> <Exposed Set>

| | | R | RSV<br>N = | |
|------------------------|---|---|------------|-------|
| | | | 9 | 5% CI |
| Categories | n | % | LL | UL |
| Influenza A Virus | | | | |
| Influenza B Virus | | | | |
| <each virus=""></each> | | | | |
| Total | | | | |

N = number of swabs tested RSV positive by qRT-PCR

### Template Table 54 Clinical signs and symptoms associated with RTI episodes (Exposed set)

| | | _ | V RTI | _ | n RSV RTI<br>I=XXXX | | otal |
|---|---|---|---|---|---|---|---|
| Characteristics | Categories | n | % | n | % | n | % |
| Heart Rate increase | 10-20 | | | | | | |
| (beats/min) | | | | | | | |
| | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Respiratory rate increase (breaths/min) | 5-10 | | | | | | |
| (breatis/iiii) | 10-15 | | | | | | |
| | 15-20 | | | | | | |
| | 20-25 | | | | | | |
| | 20 20 | | | | | | |
| Systolic blood pressure increase (mmHg) | 10-20 | | | | | | |
| , J | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Diastolic blood pressure increase (mmHg) | 10-20 | | | | | | |
| 3, | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Oxygen saturation decrease (%) | 1-2 | | | | | | |
| | 3-4 | | | | | | |
| | 5-6 | | | | | | |
| | 7-8 | | | | | | |

n/% = number/percentage of swabs tested positive by multiplex in a given category

Total= number of swabs tested positive for at least one virus

LL, UL= Exact 95% Lower and Upper confidence limits

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

| | | | V RTI | Non RSV RTI<br>N=XXXX | | | otal<br>XXXX |
|---|---|---|---|---|---|---|---|
| Characteristics | Categories | n | % | n | % | n | % |
| Upper respiratory symptoms | <each symptom=""></each> | | | | | | |
| Lower respiratory symptoms | <each symptom=""></each> | | | | | | |
| qPCR result | RSV A+ | | | | | | |
| • | RSV B+ | | | | | | |
| | RSV - | | | | | | |
| Self-collected Nasal swab | RSV+ | | | | | | |
| | RSV- | | | | | | |
| | NA | | | | | | |
| Medically attended visit | Emergency room | | | | | | |
| • | Hospitalisation | | | | | | |
| | Medical personnel | | | | | | |
| | None | | | | | | |
| SAE associated to the episode | Yes | | | | | | |
| • | No | | | | | | |

RSV RTI= RTI episode tested as RSV positive by qRT-PCR on nasal/throat swab collected at assessment visit Non-RSV RTI= RTI episode tested as RSV negative by qRT-PCR on nasal/throat swab collected at assessment visit N = number of RTI episodes in each category or in total

n = number of RTI episodes in the corresponding category

For vital signs, change from baseline (increase/decrease) will be displayed by category: category of 10 units increase for heart rate, systolic and diastolic BP, 5 units increase for respiratory rate, and 1% decrease for oxygen saturation (to be adapted at the time of dry run if needed)

### Template Table 55 Listing of RTI episodes reported during RTI surveillance in Part B (Exposed set)

| Gro | Su | Age | Se | Episo | Start | End | Date of | Nb of | Dat | RSV | RSV | Dat | RSV- | RSV- | Medica | SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| up | b. | at | X | de nb | date | date | assessm | signs | е | Α | В | е | Α | В | lly | relate |
| | No. | Dos | | | of | of | ent visit | and | nas | positi | positi | nas | positi | positi | attende | d to |
| | | e 1 | | | episo | episo | | sympto | al | ve | ve | al | ve | ve | d visit | RTI |
| | | | | | de | de | | ms | swa | (site) | (site) | swa | (hom | (hom | | episo |
| | | | | | | | | | b | | | b at | e) | e) | | de |
| | | | | | | | | | on | | | hom | | | | |
| | | | | | | | | | site | | | е | | | | |
| | | | | | | | | | | Yes/N | Yes/N | | Yes/N | Yes/N | | Yes/N |
| | | | | | | | | | | 0 | 0 | | 0 | 0 | | 0 |

Short group label = long group label

 $<sup>% =</sup> n / N \times 100$ 

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

Template Figure 11 GMTs and 95% Cls of RSV A Neutralizing antibody titer at baseline for subjects reporting RTI episodes (RSV RTI vs or non RSV RTI vs No RTI), by groups pooled according to the adjuvant content <Exposed Set>



This graph is provided as an example, template will be finalized at the time of the dry-run. It will display the GMTs and 95% CIs for subjects reporting confirmed RSV RTI episodes vs subjects reporting Non-RSV RTI episodes vs subjects who did not report any RTI episode (NON RTI), in the RSV groups pooled according to the adjuvant content (Plain, AS01E, AS01B).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### 12.6. Additional templates (Amendment 1)

### Template Table 56 Distribution of hematology and biochemistry parameters at baseline with respect to normal laboratory ranges <analysis set name>

| | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th><ea< th=""><th>ach gro</th><th>up&gt;</th></ea<></th></ea<> | ch gro | up> | <ea< th=""><th>ach gro</th><th>up&gt;</th></ea<> | ach gro | up> |
|---|---|---|---|---|---|---|---|
| Laboratory parameter | Range<br>indicator at<br>baseline | N | n | % | N | n | % |
| <each parameter=""></each> | UNKNOWN | | | | | | |
| | BELOW | | | | | | |
| | WITHIN | | | | | | |
| | ABOVE | | | | | | |

Short group label = long group label

N = number of subjects with available results for the specified laboratory parameter in a given baseline category n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

### Template Table 57 Summary of follow-up time (in days) up to <DLP or last contact> (Exposed Set)

| | <each group=""> N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|
| | Value | Value |
| Number of days in the study | | |
| N | xxx | XXX |
| Mean | XXX.X | XXX.X |
| Median | XXX.X | XXX.X |
| Minimum | xxx | XXX |
| Maximum | xxx | XXX |

Short group label = long group label

N = total number of subjects

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Amendment 2

#### Template Table 58 Summary of subjects by unsolicited adverse event category

| | | <each group=""><br/>N=XXXX</each> |
|---|---|---|
| t least one unsolicited adverse event within 30-day of any vaccination | n* | XXX |
| , , | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one related unsolicited adverse event within 30-day of any vaccination | n* | XXX |
| • | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one medically attended unsolicited adverse event within 30-day of any | n* | XXX |
| accination | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one serious unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | n* | XXX |
| · · · · · · | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one serious related unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | n* | XXX |
| | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one potential immune-mediated disorder (pIMD) <up dlp="" or="" study<="" td="" to=""><td>n*</td><td>XXX</td></up> | n* | XXX |
| nd> | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one related potential immune-mediated disorder (pIMD) <up dlp="" or<="" td="" to=""><td>n*</td><td>XXX</td></up> | n* | XXX |
| udy end> | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| t least one fatal unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | n* | XXX |
| | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once 95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
|---|---|
| Detailed Title: | A Phase I/II, randomized, placebo-controlled, observer-blind, multicenter study to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' investigational respiratory syncytial virus (RSV) vaccine (adjuvanted with AS01 <sub>E</sub> or AS01 <sub>B</sub> or unadjuvanted) when administered intramuscularly according to a 0, 2 month schedule in adults aged 18-40 or 60-80 years. |
| eTrack study number and<br>Abbreviated Title | 208851 (RSV OA=ADJ-002) |
| Scope: | All data pertaining to the above study (except IDMC analyses) |
| Date of Statistical Analysis<br>Plan | Amendment 1 Final: 27 January 2020 |
| Co-ordinating author: | PPD (Statistician) |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead) PPD , PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) PPD (Scientific writer) PPD (Stat Peer Reviewer) PPD (Regulatory Affairs) PPD (SERM physician) PPD (Safety scientist) PPD (Public disclosure representative) PPD (CLS – Clinical Read-outs) PPD (CMI Expert representative) |
| Approved by: | PPD (Clinical and Epidemiology Project Lead) PPD (Lead statistician) PPD (Statistician) PPD (Lead Scientific writer) PPD (Lead stat Analyst) |

APP 9000058193 Statistical Analysis Plan Template V4 (Effective date: 3 June 2019)

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### **TABLE OF CONTENTS**

| | | | PAGE |
|---|---|---|---|
| TAE | BLE OF | F CONTENTS | 2 |
| LIS | T OF T | TABLES | 4 |
| LIS | T OF F | FIGURES | 5 |
| LIS | T OF T | ΓΕΜΡLATE TABLES | 6 |
| LIS | T OF T | TEMPLATE FIGURES | 11 |
| LIS | T OF A | ABBREVIATIONS | 12 |
| 1. | DOCL | JMENT HISTORY | 14 |
| 2. | STUD | DY DESIGN | 14 |
| 3. | | ECTIVES/ENDPOINTS | |
| | 3.1. | Objectives | |
| | | 3.1.1. Primary objective | |
| | | 3.1.2. Secondary objectives | |
| | 2.2 | 3.1.3. Tertiary objectives | |
| | 3.2. | Endpoints | |
| | | 3.2.1. Primary endpoints | |
| | | 3.2.3. Tertiary endpoints | |
| 4. | ANAL | YSIS SETS | 24 |
| | 4.1. | Definition | 24 |
| | | 4.1.1. Exposed Set | 24 |
| | | 4.1.2. Per-Protocol Set for analysis of imr | |
| | 4.2. | Criteria for eliminating data from Analysis Se | |
| | | 4.2.1. Elimination from Exposed Set (ES) | |
| | | 4.2.2. Elimination from Per-protocol analy | sis Set (PPS)25 |
| <b>5</b> . | STAT | ISTICAL ANALYSES | 28 |
| | 5.1. | Demography | 28 |
| | | 5.1.1. Analysis of demographics/baseline in the protocol | characteristics planned |
| | | 5.1.2. Additional considerations | |
| | 5.2. | Exposure | |
| | 0.2. | 5.2.1. Analysis of exposure planned in the | |
| | | 5.2.2. Additional considerations | |
| | 5.3. | Immunogenicity | |
| | | 5.3.1. Analysis of immunogenicity planned | |
| | | 5.3.2. Additional considerations | |
| | 5.4. | Analysis of safety and reactogenicity | |
| | | 5.4.1. Analysis of safety and reactogenicit | ty planned in the |
| | | protocol | 38 |

| | | 5.4.2. | Additional considerations | 39 |
|---|---|---|---|---|
| | 5.5. | <b>Analysis</b> | of RTI for Part B | |
| | | 5.5.1. | Analysis of RTI planned in the protocol | |
| | | 5.5.2. | Additional considerations | 42 |
| 6. | ANALY | YSIS INTE | ERPRETATION | 43 |
| 7. | COND | LICT OF A | ANALYSES | 43 |
| ٠. | 7.1. | | e of analyses. | |
| | 7.2. | | al considerations for interim analyses | |
| 0 | CLIANI | | • | |
| 8. | CHAN | GES FRU | M PLANNED ANALYSES | 45 |
| 9. | | | RD DATA DERIVATION RULES AND STATISTICAL | |
| | METH | | | |
| | 9.1. | Handling | of missing data | |
| | | 9.1.1. | Dates | 47 |
| | 9.2. | Duration | of events | 48 |
| 10 | ANNE | XES | | 49 |
| 10. | 10.1. | | rules for standard data derivations and statistical methods | |
| | 10.1. | 10.1.1. | Attributing events to vaccine doses | |
| | | 10.1.2. | Handling of missing data | |
| | | 10.1.3. | Data derivation | |
| | | 10.1.4. | Display of decimals | |
| | | 10.1.5. | Statistical methodology | |
| | 10.2. | | - Catalogod Motifology | |
| 11. | REFE | RENCES. | | 53 |
| 10 | CTLID | V MOCK | TFLS | ΕΛ |
| 12. | 12.1. | | | |
| | 12.1. | | aphy | |
| | 12.2. | | egenicity | |
| | 12.3. | | Within groups | |
| | | | · | |
| | 12.4. | | Between groups | |
| | 12.4.<br>12.5. | | of DTI | |
| | 12.5.<br>12.6 | • | of RTIltemplates (Amendment 1) | |
| | 1/0 | Audinona | acientolales (Amenoment I) | 97 |

#### 208851 | Statistical Analysis Plan Amendment 1 27 Jan 2020 | TMF-1608921 | 2.0


208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### LIST OF TABLES

| | | PAGE |
|---------------|----------------|------|
| Table 1 Group | ps description | 18 |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### LIST OF FIGURES

| | | PAGE |
|----------|--------------|------|
| Figure 1 | Study design | 14 |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### LIST OF TEMPLATE TABLES

| | | PAGE |
|---|---|---|
| | e 1 Summary of demography and baseline characteristics (Exposed Set) | 54 |
| Template Table | e 2 Number of subjects by country and center (Exposed Set) | 55 |
| Template Table | e 3 Number of subjects by study steps (Exposed Set) | 55 |
| Template Table | e 4 Summary of vital signs (Exposed Set) | 55 |
| • | e 5 Summary of study completion with reason for withdrawal (Exposed Set) | 56 |
| Template Table | e 6 Summary of visit attendance (Exposed Set) | 56 |
| | e 7 Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set) | 57 |
| | e 8 Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set) | 57 |
| Template Table | e 9 Summary of subject disposition from Randomized Set to Exposed set (Randomized set) | 57 |
| | e 10 Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set) | 58 |
| • | e 11 Summary of subject disposition from Exposed Set to End of study (Exposed set) | 58 |
| | e 12 Deviations from protocol for age and intervals between study visits (Exposed set) | 59 |
| Template Table | e 13 Number of enrolled subjects by country | 59 |
| Template Table | e 14 Number of enrolled subjects by age category | 59 |
| Template Table | e 15 Minimum and maximum visit dates <analysis name="" set=""></analysis> | 60 |
| Template Table | e 16 Exposure to study vaccines by vaccine (Exposed Set) | 60 |
| | e 17 Number and percentage of subjects with <antibody concentration="" titer=""> equal to or above <cut-off unit=""> and <gmt cs=""> <analysis name="" set=""></analysis></gmt></cut-off></antibody> | 61 |
| · · | e 18 Geometric mean of the individual ratio of <antibody (units)="" concentrations="" titers=""> post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | 63 |

| • | e 20 Distribution of <antibody concentrations="" titers=""> fold increase post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | 63 |
|---|---|---|
| · | e 21 Geometric mean ratios of the fold increase (Pre to Post - vaccination) between RSVPreF3 IgG antibody concentrations and <rsv-a, rsv-b=""> neutralising antibody titers <per protocol="" set=""> 67</per></rsv-a,> | |
| · | e 22 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL- 2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 68 |
| • | e 23 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by pre-vaccination category <per protocol="" set=""></per> | 69 |
| · | e 24 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | 71 |
| • | e 25 Descriptive statistics of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <per protocol="" set=""></per> | 72 |
| · | e 26 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <per protocol="" set=""></per> | 72 |
| · | e 27 Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | <b>7</b> 3 |
| | e 28 Comparisons of the 9 RSV formulations versus Placebo in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at one month post <dose (day="" 1="" 2="" 31),="" 91)="" dose=""> (ANCOVA model, Dunnett's test) – Part B <per protocol="" set=""> 73</per></dose></rsv> | |
| | e 29 Comparisons of the mean responses post dose 2 (Day 91) versus post dose 1 (Day 31) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> on pooled groups according to adjuvant content (ANCOVA model) – Part B <per protocol="" set=""></per></rsv> | 74 |

| Template Tab | le 30 Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) - Part B <per protocol="" set=""></per></rsv> | 75 |
|---|---|---|
| Template Tab | le 31 Comparisons of the RSV groups (by antigen dose level) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) – Part B <per protocol="" set=""> 76</per></rsv> | |
| Template Tab | le 32 Parameters of the ANCOVA model for the comparison between RSV groups in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,="">- Part B <analysis name="" set=""></analysis></rsv> | 77 |
| Template Tab | le 33 Compliance in completing solicited adverse events information (Exposed Set) | 77 |
| Template Tab | le 34 Incidence and nature of <grade 3=""> symptoms (solicited and unsolicited) <with causal="" relationship="" to="" vaccination=""> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis name="" set=""></analysis></with></grade> | 78 |
| Template Tab | le 35 Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <analysis name="" set=""></analysis> | 79 |
| Template Tab | le 36 Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <analysis name="" set=""></analysis> | 79 |
| Template Tab | le 37 Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <cohort name=""></cohort> | 80 |
| Template Tab | le 38 Number of days with < local/general> solicited symptoms during < the 7-day (Days 1-7), the whole> post-vaccination period < analysis set name> | 82 |
| Template Tab | le 39 Percentage of subjects reporting the occurrence of <grade 3=""> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> within the 30-day (Days 1-30) post-vaccination period <analysis name="" set=""></analysis></with></grade> | 84 |
| Template Tab | le 40 List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <exposed set=""></exposed> | 84 |

| Template Tab | e 41 Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or | 0.5 |
|---|---|---|
| | by investigator assessment <analysis name="" set=""></analysis> | 65 |
| Template Tab | e 42 Listing of SAEs <analysis name="" set=""></analysis> | 85 |
| Template Tab | e 43 Listing of pregnancies reported during the study period in Part A <analysis name="" set=""></analysis> | 86 |
| Template Tab | e 44 Number and percentage of subjects taking concomitant medication during the <xx>-day (Days 1-<xx>) post-vaccination period by dose and overall <analysis name="" set=""></analysis></xx></xx> | 86 |
| Template Tab | e 45 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges, 7 days post dose <1, 2> <analysis name="" set=""></analysis> | 88 |
| Template Tab | le 46 Summary of hematology and biochemistry results by grade at 7 days post dose <1, 2 > versus baseline ( <day 1,="" 61="" day="">) <a href="mailto:analysis set name">analysis set name</a>&gt;</day> | 88 |
| Template Tab | e 47 Summary of hemoglobin change from baseline at 7 days post-dose <1, 2> (Exposed set) | 89 |
| Template Tab | e 48 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis name="" set=""></analysis> | 90 |
| Template Tab | e 49 Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis name="" set=""></analysis> | 90 |
| Template Tab | e 50 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis name="" set=""></analysis> | 91 |
| Template Tab | le 51 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis name="" set=""></analysis> | 91 |
| Template Tab | le 52 Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <exposed set=""></exposed> | 92 |
| Template Tab | le 53 Descriptive statistics of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <at home=""> <exposed set=""></exposed></at> | Q? |
| | Homes styloged dets | 52 |

| | • | |
|---|---|---|
| infecti<br>PCR ( | Number and percentage of subjects reporting coons with respiratory viruses, as measured by multiplex on RSV A/B positive RTI samples collected <at assessment="" at="" home=""> <exposed set=""></exposed></at> | 93 |
| | Clinical signs and symptoms associated with RTI episodes sed set) | 93 |
| | Listing of RTI episodes reported during RTI surveillance in (Exposed set) | 95 |
| baseli | Distribution of hematology and biochemistry parameters at ne with respect to normal laboratory ranges <analysis set=""></analysis> | 97 |
| | Summary of follow-up time (in days) up to <dlp ct="" last="" or=""> (Exposed Set)</dlp> | 97 |
| | Summary of subjects by unsolicited adverse event ory | 98 |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### LIST OF TEMPLATE FIGURES

| | | | PAGE |
|---|---|---|---|
| Template Figu | | > and their 95% CIs for <antibod <analysis="" name="" set=""></antibod> | |
| Template Figu | | cumulative distribution curve of <- ons> in the <group label=""> group</group> | |
| Template Figu | available at all tir | f < antibody GMT/Cs> on subject<br>mepoints up to <day 1<="" 91,="" month="" td=""><td>4&gt; <per< td=""></per<></td></day> | 4> <per< td=""></per<> |
| Template Figu | <time point=""> vers</time> | results of <rsv a="" a<br="" neutralizing="">sus pre-vaccination in <group lab<br="">ps <per protocol="" set=""></per></group></rsv> | el> and |
| Template Figu | antibody titer> at | results of <rsv <time="" a="" et="" point="" rsv="" versus="">, on pooled RSV g</rsv> | roups <per< td=""></per<> |
| Template Figu | vaccination) of R <rsv a,="" b="" rsv=""></rsv> | results of the fold increase (post<br>RSVPreF3 IgG antibody concentre<br>> neutralizing antibody titers at <<br>Per protocol set> | ations versus<br>time point> in |
| Template Figu | RSVPreF3 speciments among IL-2, CD4 | with individual data of the frequer<br>ific-CD4+ T cells expressing at le<br>40L, TNFa, IFNg (per million of C<br>col set> | ast 2 markers<br>D4+ T cells, by |
| Template Figu | any combination <group label=""> group</group> | y of RSVPreF3 specific CD4+ T-<br>of markers among IL-2, CD40L,<br>oup at Day 31 and Day 91 (per n<br><per protocol="" set=""></per> | TNFa, IFNg in<br>nillion of CD4+ |
| Template Figu | reported during the | of solicited <local, general=""> adverbe 7-day (Days 1-7) post-vaccina ose <exposed set=""></exposed></local,> | ation period |
| Template Figu | | Boxplot of <each b<="" hematology="" td=""><td>•</td></each> | • |
| Template Figu | antibody titer at b<br>(RSV RTI vs or n | GMTs and 95% CIs of RSV A No baseline for subjects reporting Ronon RSV RTI vs No RTI), by grou | ΓI episodes<br>ps pooled |
| | according to the | adjuvant content < Exposed Set> | •96 |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### LIST OF ABBREVIATIONS

AE Adverse event

ALT Alanine Aminotransferase
ANCOVA Analysis of Covariance
ANOVA Analysis of Variance

AST Aspartate Aminotransferase

BUN Blood Urea Nitrogen

CD40L Cluster of Differentiation 40 Ligand

CI Confidence Interval

CMI Cell-Mediated Immunity

CMV Cytomegalovirus

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

DLP Data Lock Point

eCRF electronic Case Report Form

eDiary electronic Diary

ELISA Enzyme-linked immunosorbent assay

ELU/ml ELISA unit per milliliter

EoS End of Study
ES Exposed Set

FDA Food and Drug Administration

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICS Intracellular Cytokine Staining

IDMC Independent Data Monitoring Committee

IFN-γ Interferon Gamma
IgG Immunoglobulin G

IL Interleukin

LL Lower Limit of the confidence interval

LLOQ Lower Limit Of Quantification

Mcg or µg Microgram

MedDRA Medical Dictionary for Regulatory Activities

#### 208851 | Statistical Analysis Plan Amendment 1 27 Jan 2020 | TMF-1608921 | 2.0


208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

PBMC Peripheral Blood Mononuclear Cells

PCR Polymerase Chain Reaction

PD Protocol Deviation

pIMD Potential Immune-Mediated Disease

PPS Per Protocol Set
PT Preferred Term

qRT-PCR Quantitative Reverse Transcription Polymerase Chain Reaction

RSV Respiratory Syncitial Virus
RTI Respiratory Tract Infection

SAE Serious adverse event SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

TFL Tables Figures and ListingsTNF-α Tumor Necrosis Factor alpha

TOC Table of Content

UL Upper Limit of the confidence interval

WBC White Blood cells
208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|---|---|---|
| 14-JAN-2019 | first version | Final: 11 SEP 2018 |
| 27-JAN-2020 | Amendment 1: implement changes discussed at | Final: 11 SEP 2018 |
| | the KOM Dry-run and progress meetings | |

## 2. STUDY DESIGN

Figure 1 Study design



BS S: Blood sample for safety (hematology/biochemistry)

BS H: Blood sample for humoral immune responses

BS C: Blood sample for cell-mediated immune responses (for CD4+/CD8+ and/or memory B-cell testing)

FU: Follow-up; PCR: Polymerase Chain Reaction

<sup>\*</sup> Visit 1 should take place no longer than 30 days after the Screening Visit. In case Visit 1 occurs more than 30 days after the Screening Visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection for safety laboratory assessment must be repeated (maximum one re-screening per subject is allowed). Only laboratory results from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. The subject can only be randomized once the investigator receives the results and confirms the eligibility criteria.

- \*\* In Part A, a first IDMC evaluation of safety data up to Day 31 based on all subjects (~12 per group or at least 8 per group in case of slow recruitment) will be performed before proceeding with administration of Dose 2 in Part A and Dose 1 in Part B. A second IDMC evaluation will be performed based on safety data up to Day 68 for all subjects. Part B of the study can only be initiated upon favorable outcome of the first IDMC safety evaluation in Part A.
- \*\*\* In Part B, a third and fourth IDMC evaluation of safety data up to Day 8 and Day 68, respectively, for the first enrolled and vaccinated subjects (~10 per group or at least 8 per group in case of slow recruitment) will be performed. Additional IDMC evaluations will happen during the conduct of the study.
- <sup>†</sup> In case of RTI symptoms during the RSV seasons (approximately from October to March), the subject will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab at the site. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- <sup>£</sup> Analysis 1 will be performed on all data collected up to Day 91 for at least primary and secondary endpoints based on both study parts (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). Analysis 2 will be performed when all safety data up to Month 8 (Visit 7) are available. The analyses will be based on data as clean as possible.
- **Experimental design:** Phase I/II, observer-blind, randomized, controlled, multicountry study with 2 parts (i.e., Part A in young adults aged 18-40 years with 4 parallel groups and Part B in older adults aged 60-80 years with 10 parallel groups).
- **Primary Completion Date (PCD):** last visit of the vaccination phase in Part B (Visit 6 [Day 91]).
- End of Study (EoS): Last testing results released of samples collected up to Visit 8 in Part B (Month 14) (for assays related to primary and secondary endpoints only).
- **Treatment allocation:** Subjects will be randomized using a centralised randomization system on internet (SBIR) on Day 1.

In Part A, the aim is to enrol approximately 48 subjects (~12 per group) aged 18-40 years. The randomization algorithm will use a minimisation procedure accounting for center and gender.

In Part B, the aim is to enrol approximately 700 subjects (~70 per group) aged 60-69 years and approximately 300 subjects (~30 per group) aged 70-80 years. The randomization algorithm will use a minimisation procedure accounting for age, center and gender in each step.

# • Study groups:

For the investigational RSV vaccines in Part A and Step 1 in Part B, the RSVPreF3 high-dose formulation containing 120  $\mu$ g RSVPreF3 will be used to prepare the vaccines for all dose groups (i.e., 30  $\mu$ g, 60  $\mu$ g and 120  $\mu$ g dose groups). For Step 2 in Part B, the RSVPreF3 low-dose and mid-dose formulations (containing 30  $\mu$ g and 60  $\mu$ g RSVPreF3, respectively) will be used for the groups receiving 30  $\mu$ g and 60  $\mu$ g of RSVPreF3, respectively, and the RSVPreF3 high-dose formulation will be used for the 120  $\mu$ g dose groups. As the reconstitution methods for the vaccines administered to subjects enrolled in Step 1 and 2 of Part B will be different, separate study groups have been identified (referred to as B1 and B2). Throughout this

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

document, the combined groups for Steps 1 and 2 are mentioned when referring to the number of groups in Part B (10 groups).

- Control: placebo.
- **Vaccination schedule:** Two vaccine doses administered intramuscularly at Day 1 and Day 61.
- **Blinding**: observer-blind.

The vaccination phases of each study part (Epoch 002) will be observer-blind. A first statistical analysis will be performed on data available up to one month post-Dose 2 (Visit 6, Day 91). Given that summary safety results may unblind some specific subjects, the persistence phase of Part B (Epoch 003) will be considered as single-blind with subjects remaining blinded up to study end (Visit 8 [Month 14]). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

- RTI surveillance in Part B: Active and passive surveillance will only be carried out during RSV seasons (approximately from October to March) throughout the entire Part B of the study:
  - Active surveillance: study participants will be contacted by the investigator/study staff every 2 weeks to identify if they experience an RTI.
  - Passive surveillance: study participants are instructed to contact the investigator/study staff as soon as they experience an RTI.

At the beginning of RSV seasons, study participants will be reminded of the start of the RTI surveillance.

## • Sampling schedule:

## In Part A:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the electronic Case Report Form (eCRF). The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for cytomegalovirus (CMV) status determination will be drawn from all subjects.
- **Blood samples for safety assessment** (hematology/biochemistry) will be drawn from all subjects on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Blood samples for humoral immunogenicity and cell-mediated immunity
 (CMI) testing will be drawn from all subjects at Days 1, 31, 61 and 91 (Visits 1, 3, 4 and 6).

### In Part B:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF. The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for CMV status determination will be drawn from all subjects.
- **Blood samples for safety assessment** (hematology/biochemistry) will be drawn from all subjects and on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).
- **Blood samples for humoral immunogenicity and CMI** testing will be drawn from all subjects at Days 1, 31, 61, 91, Month 8 and Month 14 (Visits 1, 3, 4, 6, 7 and 8).
- Nasal/throat swabs: In case of RTI symptoms during the RSV season (approximately from October to March), the study participants will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab by qualified staff from the study team. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- Type of study: self-contained.
- **Data collection:** eCRF. Solicited symptoms will be collected using an electronic subject Diary (eDiary). Unsolicited symptoms will be collected using a paper subject Diary.
- **Safety monitoring:** The study will be conducted in 2 parts with oversight by an IDMC. The investigator is not permitted to start vaccinating the subjects in the next step in each part until receipt of the favorable outcome of the respective safety evaluations by the IDMC.
  - Part A: Approximately 48 young adults aged 18-40 years will be enrolled and vaccinated with the first dose. If the IDMC evaluation on data up to 30 days post Dose 1 is favorable, the Part A study participants will be vaccinated with the second dose and Part B of the study will be initiated.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Part B: This part will be conducted in a 2-step staggered design to ensure maximum safety of the participating subjects. In Step 1, approximately 100 subjects will be enrolled and vaccinated. Safety evaluations based on unblinded data from those first 100 subjects will be performed by the IDMC to allow the start of Step 2. In Step 2, the remaining study participants (N≅900) will be recruited and vaccinated.

In total, 6 IDMC meetings for safety evaluation are foreseen in the vaccination phase of the study (Epoch 002), i.e., 2 meetings in Part A and 4 meetings in Part B.

During the persistence phase of Part B (Epoch 003), 2 IDMC meetings will be planned with an interval of approximately 6 months.

If any safety concern is identified by the investigator or the sponsor, *ad-hoc* safety evaluations by the IDMC may be performed.

Analysis planned for IDMC evaluations are described in a separate document (SAP for IDMC).

## • Group description for analysis:

For analysis based on subjects in Part A and Part B Step 1 (B1), the group labels listed in table below will be used in the TFLs.

For final analysis based on subjects from Part B Steps 1 and 2, the groups will be pooled (B1 and B2) and the Pooled group labels will be used in the TFLs.

Table 1 Groups description

| Group label in tables | Group definition for footnote | Pooled Group label in tables | Pooled Group definition for footnote |
|---|---|---|---|
| 30-PLAIN_A | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part A | NA | |
| 60-PLAIN_A | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part A | NA | |
| 120-PLAIN_A | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part A | NA | |
| Placebo_A | subjects receiving Placebo in Part A | NA | |
| 30-PLAIN_B1 | subjects receiving unadjuvanted<br>30 mcg RSVPreF3 in Part B Step<br>1 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |
| 30-PLAIN_B2 | subjects receiving unadjuvanted<br>30 mcg RSVPreF3 in Part B Step<br>2 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |
| 60-PLAIN_B1 | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B Step<br>1 | 60-PLAIN_B | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part B |
| 60-PLAIN_B2 | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B Step<br>2 | 60-PLAIN_B | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part B |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| Group label in | Group definition for footnote | Pooled Group | Pooled Group definition for footnote |
|---|---|---|---|
| tables | | label in tables | • |
| 120-PLAIN_B1 | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B Step<br>1 | 120-PLAIN_B | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part B |
| 120-PLAIN_B2 | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B Step<br>2 | 120-PLAIN_B | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part B |
| 30-AS01E_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 30-AS01E_B | subjects receiving 30 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 30-AS01E_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 30-AS01E_B | subjects receiving 30 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 60-AS01E_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 60-AS01E_B | subjects receiving 60 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 60-AS01E_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 60-AS01E_B | subjects receiving 60 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 120-AS01E_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 120-AS01E_B | subjects receiving 120 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 120-AS01E_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 120-AS01E_B | subjects receiving 120 mcg RSVPreF3 adjuvanted with AS01E in Part B |
| 30-AS01B_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 30-AS01B_B | subjects receiving 30 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| 30-AS01B_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 30-AS01B_B | subjects receiving 30 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| 60-AS01B_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 60-AS01B_B | subjects receiving 60 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| 60-AS01B_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 60-AS01B_B | subjects receiving 60 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| 120-AS01B_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 120-AS01B_B | subjects receiving 120 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| 120-AS01B_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 120-AS01B_B | subjects receiving 120 mcg RSVPreF3 adjuvanted with AS01B in Part B |
| Placebo_B1 | subjects receiving Placebo in Part<br>B Step 1 | Placebo_B | subjects receiving Placebo in Part B |
| Placebo_B2 | subjects receiving Placebo in Part B Step 2 | Placebo_B | subjects receiving Placebo in Part B |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

For some of the comparison analyses in Part B, the RSV vaccine groups will be pooled according to their adjuvant content and the following group names will be used in the TFLs:

| Pooled Group label in tables | Pooled Group definition for footnote | Groups to be pooled |
|---|---|---|
| PLAIN_B | subjects receiving unadjuvanted RSVPreF3 in Part B (30, 60 or 120 μg) | 30_PLAIN_B1, 30_PLAIN_B2,<br>60_PLAIN_B1, 60_PLAIN_B2,<br>120_PLAIN_B1, 120_PLAIN_B2 |
| AS01E_B | subjects receiving RSVPreF3 adjuvanted with AS01E in Part B (30, 60 or 120 μg) | 30_AS01E_B1, 30_ AS01E_B2, 60_ AS01E<br>_B1, 60_ AS01E_B2, 120_ AS01E_B1,<br>120_ AS01E_B2 |
| AS01B_B | subjects receiving RSVPreF3 adjuvanted with AS01B in Part B (30, 60 or 120 μg) | 30_AS01B_B1, 30_ AS01B_B2, 60_ AS01B<br>_B1, 60_ AS01B_B2, 120_ AS01B_B1,<br>120_ AS01B_B2 |

For the analysis by age category, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sin-droin lane in tables Sin-droin definition for footnot | |
|---|---|---|
| 1 60-69Y | | 60-69 years old subjects |
| 2 | 70-80Y | 70-80 years old subjects |

For the analysis by CMV status before vaccination, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 CMV+ | | Subjects CMV positive before vaccination |
| 2 | CMV- | Subjects CMV negative before vaccination |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 3. OBJECTIVES/ENDPOINTS

# 3.1. Objectives

# 3.1.1. Primary objective

## For Part A and Part B:

• To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccine administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

## 3.1.2. Secondary objectives

## For Part A and Part B:

- To characterize the humoral immune responses (including dose-response) in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).
- To characterize the cell-mediated immune responses in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

#### For Part B:

- To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccines administered IM according to a 0, 2 month schedule, up to the end of follow-up (Month 14, Visit 8).
- To evaluate the occurrence of RSV-associated respiratory tract infections (RTI) during the RSV season in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.

# 3.1.3. Tertiary objectives

## For Part A and Part B:

• To further characterize the cell-mediated immune responses to investigational RSV vaccine formulations.

#### For Part B:

- To further characterize immune responses to investigational RSV vaccine formulations.
- To characterize persistence of immune responses to the investigational RSV vaccine formulations at Month 8 (Visit 7) and Month 14 (Visit 8).
- To further evaluate the occurrence of RSV-associated RTI (including co-infections with other respiratory viruses) during the RSV seasons in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

• To evaluate the occurrence of RSV-associated RTI during the RSV season using self-collected nasal swabs.

# 3.2. Endpoints

## 3.2.1. Primary endpoints

#### For Part A and Part B:

- Occurrence of AEs from first vaccination up to 30 days after the second vaccination (Day 91):
  - Occurrence of each solicited local and general AE during a 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) after each vaccination.
  - Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.
  - Occurrence of any hematological (erythrocytes, WBC and differential count, platelets count and hemoglobin level) and biochemical (ALT, AST, creatinine, BUN and uric acid) laboratory abnormalities at Days 1, 8, 61 and 68.
  - Occurrence of all Grade 3 non-serious AEs (solicited and unsolicited) during the 30-day follow-up period after each vaccination.
  - Occurrence of SAEs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

## For Part B only:

 Occurrence of pIMDs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

## 3.2.2. Secondary endpoints

## For Part A and Part B:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), on the day of second vaccination (Day 61) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.
- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least
     2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## For Part B only:

- Occurrence of RSV-associated RTI (as measured by qRT-PCR in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons, up to the end of follow-up.
- Occurrence of SAEs from Dose 1 up to the end of follow-up.
- Occurrence of pIMDs from Dose 1 up to the end of follow-up.

# 3.2.3. Tertiary endpoints

## For Part A and Part B:

- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro.

## For Part B only:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype B in all subjects.
  - RSVPreF3 site 0 specific antibody concentrations in a subset of subjects who received the selected vaccine formulation or placebo.
- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific memory B-cells in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Persistence of the humoral immune response with respect to components of the investigational vaccine at Months 8 and 14:
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.
- Persistence of the cell-mediated immune response profile with respect to components of the investigational vaccine:
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro, in all subjects (Month 8) and in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo (Month 14).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least
   2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro, in all subjects (Month 8)
   and in a subset of subjects who received the selected level of antigen dose (3
   RSV vaccine formulations) or placebo (Month 14).
- Frequency of RSVPreF3-specific memory B-cells at Month 14 in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Any further exploratory immunology to detect RSV-related immune responses, such as but not limited to:
  - Antibodies against specific protein F epitopes.
  - Potential new immunological markers for protection.
  - Cross-reactive neutralizing antibody titers against hMPV
- Occurrence of RSV-associated RTI, including co-infections with other respiratory viruses (as measured by multiplex PCR in self-collected nasal swab samples and nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons.
- Occurrence of RSV-associated RTI as measured by qRT-PCR in self-collected nasal swab samples during the RSV seasons, up to the end of follow-up.

## 4. ANALYSIS SETS

#### 4.1. Definition

## 4.1.1. Exposed Set

The Exposed Set (ES) will include all subjects with study vaccine administration documented

A safety analysis based on the ES will include all vaccinated subjects.

An immunogenicity analysis based on ES will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at Dose 1.

# 4.1.2. Per-Protocol Set for analysis of immunogenicity

The Per-Protocol set (PPS) for analysis of immunogenicity will be defined by time point (and this to include all eligible subjects' data up to the time of important protocol deviations). The PPS will include all evaluable subjects in the ES:

- Meeting all eligibility criteria.
- For whom the administration route of the vaccine was as according to protocol.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- For whom the study vaccine was administered as per protocol.
- Who did not receive a concomitant medication/ product leading to exclusion from a PP analysis, as described in Section 6.6.2 of the protocol, up to the considered time point.
- Who did not present with a medical condition leading to exclusion from a PP analysis, as described in Section 6.7 of the protocol, up to the considered time point.
- Who complied with the vaccination schedule, as specified in the protocol.
- Who complied with the timings of the post-vaccination blood sampling for immune response evaluation, as specified in the protocol.
- For whom post-vaccination immunogenicity results are available for at least one assay component at the corresponding time points.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES.

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

## 4.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions.

For codes 1040, 1070, 1080, 1090, 2040, 2060, 2080: subjects will be eliminated from the time at which the condition is met onwards.

For codes 2090, 2100, 2120: subjects will be eliminated at the specific visit at which the condition is met.

When applicable, codes will be allocated to subjects as long as they are included in the study. For example, withdrawals before the second dose will not be attributed a code 1070 because they missed a dose.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 900 | Invalid informed consent or fraudulent data | All | All |
| 1030 | Study vaccine not administered at all | All | All |
| 1040 | <ul> <li>Administration of concomitant vaccine(s) forbidden in the protocol: <ul> <li>Any investigational or non-registered vaccine other than the study vaccine used during the study period</li> <li>A vaccine not foreseen by the study protocol administered during the period starting 30 days before the first dose and ending 30 days after the last vaccine dose, except for inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after each vaccination.</li> </ul> </li> </ul> | All | Immunology |
| 1050 | Randomisation failure | All | Immunology |
| 1060 | Randomisation code was broken | All | Immunology |
| 1070 | Vaccination not according to protocol: Incomplete vaccination course Subject was vaccinated with the correct vaccine but containing a lower volume Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) Route of the study vaccine is not intramuscular Wrong reconstitution of administered vaccine | Vaccination<br>Visits 1 and 4 | Immunology |
| 1080 | Vaccine temperature deviation vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation | Vaccination visits 1 and 4 | Immunology |
| 1090 | Expired vaccine administered | Vaccination visits 1 and 4 | Immunology |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | Immunology |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 2040 | <ul> <li>Administration of any medication forbidden by the protocol</li> <li>Any investigational or non-registered medication used during the study period</li> <li>Immunosuppressants or other immune-modifying drugs administered chronically (i.e., more than 14 consecutive days in total) during the study period</li> <li>Long-acting immune-modifying drugs administered at any time during the study period</li> <li>Immunoglobulins and/or any blood products administered during the study period</li> </ul> | All | Immunology |
| 2060 | Intercurrent medical condition • Subjects may be eliminated from the PPS if, during the study, they incur a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status (other than RSV infection). | All | Immunology |
| 2080 | Subjects did not comply with vaccination schedule: • Part A: number of days between dose 1 and dose 2 is outside [55-80 days] • Part B: number of days between dose 1 and dose 2 is outside [55-75 days] | Visit 4 | Immunology |
| 2090 | Subjects did not comply with blood sample schedule at a specific visit: Number of days between dose 1 and visit 3 blood sample is outside [30-37 days] Number of days between dose 1 and visit 4 blood sample is outside [55-80 days] for Part A or [55-75 days] for Part B Number of days between dose 2 and visit 6 blood sample is outside [30-37 days] Part B only: Number of days between dose 2 and visit 7 blood sample is outside [170-190 days] Number of days between dose 2 and visit 8 blood sample is outside [350-395 days] | Visits 3, 4, 6, 7 and 8 | Immunology |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 2100 | Immunological results not available post-vaccination No immunological result at visit x for all 3 following tests: RSV A Neutralising antibody titer, RSVPreF3-specific IgG antibody concentration and RSVPreF3-specific CD4+ T cells frequency | Visits 3, 4, 6, 7, 8 | Immunology |
| 2120 | Obvious incoherence or abnormality or error in data Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at lab | Visits 1, 3, 4, 6, 7, 8 | Immunology |

## 5. STATISTICAL ANALYSES

Note that standard data derivation rules and stat methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and stat methods will be described in section 9

# 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at first vaccination in years, gender, race and ethnicity) will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (60-69 years and 70-80 years in Part B only).

Withdrawal status will be summarized by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PP analyses will be tabulated.
- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### 5.1.2. Additional considerations

The analysis of demographic characteristics by group will be performed on the ES and on the PPS.

Demography and baseline characteristics will also be summarized by country.

Vital signs (heart rate, respiratory rate, systolic/diastolic blood pressure, pulse oximetry) and pre-vaccination temperature reported at visit 1 (Part A and Part B) will be summarized by group using descriptive statistics.

Subject disposition in the ES and PPS will be reported as a whole and per group, and for each age category (60-69 years and 70-80 years in Part B only).

Distribution of hematology and biochemistry parameters at baseline with respect to normal laboratory ranges will be tabulated by group.

For Part B only, the follow-up time in the study (in days) up to DLP for analysis or up to last contact will be described overall and by group using descriptive statistics.

# 5.2. Exposure

# 5.2.1. Analysis of exposure planned in the protocol

NA

#### 5.2.2. Additional considerations

The number of doses of study vaccines administered will be tabulated by group and by vaccine.

# 5.3. Immunogenicity

# 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be performed on the PPS for immunogenicity in Part A and Part B.

In Part B only: if in any study group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is at least 10%, a second analysis will be performed on the ES.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 5.3.1.1. Within groups evaluation - humoral immune response

For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified):

## In Part A and Part B:

- Percentage of subjects above pre-defined threshold and their exact 95% CI will be tabulated.
- GMCs/GMTs and their 95% CI will be tabulated and represented graphically.
- Geometric mean of ratios of antibody titer/concentrations at each post-vaccination time point over pre-vaccination (Day 1) will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves.
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will be computed and tabulated using descriptive statistics.

## In Part B only:

- Individual post-vaccination results (at Days 31 and 91) versus pre-vaccination results (Day 1) will be plotted using scatter plots. Results of the placebo group will be used as a reference.
- Distribution of the fold increase of the antibody titers/concentrations (post- over prevaccination titers) will be tabulated.
- The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points.

The immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

The humoral immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

#### 5.3.1.2. Within groups evaluation - Cell-mediated immune response

The following parameters will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI:

30

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## In Part A and Part B:

- Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, upon in vitro stimulation and background substracted, measured by ICS using PBMCs.
- Frequency of CD4+ and/or CD8+ T-cells expressing **any combination of immune marker(s)** among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs (see details in section 5.3.2.2).
- Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.

## In Part B only:

- Frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.
- Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

This will be displayed overall and by pre-vaccination category: <Q1, Q1-Q3, >Q3, where Q1/Q3 are respectively the 25<sup>th</sup> and the 75<sup>th</sup> percentiles of the results at pre-vaccination computed on pooled groups.

In addition, vaccine response in terms of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , will be explored and summarised by group.

The descriptive immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

The cell-mediated immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

# 5.3.1.3. Between groups evaluation (Part B only)

Statistical analyses will be performed to compare the 9 RSV investigational vaccine formulations in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

The between-groups analysis will be performed using an ANCOVA model, in several steps as follows:

1. The 9 RSV formulations will be first compared to the Placebo in order to identify groups whose means are significantly higher from the mean of the Placebo group, in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells at Day 31 and Day 91 (One-sided alpha=2.5%, Dunnett's adjustment test for multiplicity).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- 2. The effect of the second vaccination will be evaluated by comparing the means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31), of the groups pooled according to their adjuvant content (AS01<sub>B</sub>, AS01<sub>E</sub> and Plain), in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibody titers (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose).
  - Based on the results of this test, the next comparisons will be performed either at Day 91 or at Day 31.
- 3. Appropriate contrasts will be implemented to compare the RSV formulations as follows:
  - To demonstrate the adjuvant effect (on pooled groups according to their adjuvant content: AS01<sub>B</sub>, AS01<sub>E</sub>, Plain), by testing sequentially AS01<sub>B</sub> and AS01<sub>E</sub> versus Plain (One-sided alpha=2.5% for each superiority test: Adjuvant >Plain) in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibodies and, if applicable, by comparing AS01<sub>B</sub> vs AS01<sub>E</sub>.
  - To demonstrate linearity of increase in immune response when increasing the antigen dose in each adjuvanted group in terms of RSV-A neutralizing antibody and/or RSVPreF3-specific CD4+ T-cells.
  - Further ANCOVA t-tests would demonstrate superiority of 120 μg or 60 μg, should a quadratic effect be demonstrated.

Similar exploratory comparisons might also be performed on the RSVPreF3 ELISA antibody concentrations if deemed necessary.

## 5.3.2. Additional considerations

#### 5.3.2.1. Within groups – humoral immune response

- Correlations between assays of the humoral response will be investigated using scatter plots generated on pooled RSV groups in Part B:
  - RSVPreF3-specific IgG versus RSV A neutralizing antibody titer at each timepoint,
  - RSV A versus RSV B neutralizing antibody titer at Pre-vaccination and Day 91
  - RSVPreF3-specific IgG versus RSV-B neutralizing antibody titer at Prevaccination and Day 91

The same analysis will be performed on the fold increase post over pre-vaccination.

For each assay, values strictly below the cut-off and values strictly greater than the upper limit of quantification (ULOQ) will not be used for the scatter plots neither for the evaluation of the coefficients of correlation.

• The fold increase (post over pre-vaccination) of the RSVPreF3 IgG antibody concentrations versus the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will also be displayed graphically <u>by group</u> using scatter plots.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- The hMPV neutralizing antibody titers will also be tested at Day 1 and Day 91, on all subjects in Part A and on a subset of 40 subjects per group in Part B. The following analysis will be performed for each hMPV subtypes (A1, B1, A2, B2):
  - Percentage of subjects above pre-defined threshold and their exact 95% CI will be tabulated.
  - GMTs and their 95% CI will be tabulated and represented graphically.
  - Geometric mean of ratios of antibody titer at post-vaccination time point (Day 91) over pre-vaccination (Day 1) will be tabulated with 95% CI.
  - Antibody titer will be displayed using reverse cumulative curves.
  - Distribution of the fold increase of the antibody titers (post- over pre-vaccination titers) will be tabulated.
  - Individual post-vaccination results (Day 91) versus pre-vaccination results (Day 1) will be plotted using scatter plots for the selected RSV formulation and the placebo group as a reference.

## 5.3.2.2. Within groups – Cell-mediated immune response

**Descriptive statistics** of the cell-mediated immune response will be tabulated and displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.

The RSVPreF3-specific CD4+/CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+/CD8+ T cells.

More specifically, the frequencies of RSVPreF3-specific CD4+ T cells expressing at least 2 cytokines [ $Freq^{2+}$ ] will be computed as follows:

$$Freq_{Background}^{2+} = \frac{n_{background}^{2+}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2+} = \frac{n_{Induction}^{2+}}{N_{Induction}^{CD4}}$ ,

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with medium only (background)

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with a pool of peptides covering RSVPreF3 (induction)

 $N_{Back/Ind}^{CD4}$  = Total number of CD4 T cells involved in the assay (background or induction)

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Same computations will be done for all CMI responses that will be analysed, i.e.:

- Frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least 2 markers including at least 1 cytokine\* among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs.
- \* cytokines are IL-2, TNF-α, IFN-γ, IL-13, and IL-17
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IFN-γ (Th1-like response), as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IL-13 (Th2-like response), as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/ CD8+ T-cells expressing at least IL-17 (Th17-like response), as measured by ICS using PBMCs.
- Co-expression profile: Frequency of RSVPreF3-specific CD4+ T-cells expressing any combination of marker(s) among CD40L, IL-2, TNF-α, IFN-γ, as measured by ICS using PBMCs, at Day 31 and Day 91 (→15 combinations).

**Vaccine response** in terms of RSVPreF3-specific CD4+ T cells frequencies expressing at least 2 markers among CD40L, IL-2, TNF-α, IFN-γ will be explored as follows:

• Distribution of the fold increase: the percentage of subjects with at least a 2-fold, 4-fold, 6-fold, 8-fold, 10-fold increase post-vaccination as compared to pre-vaccination (Post over Pre) will be tabulated by timepoint and by group.

For the computation of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 marker(s)** among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

## 5.3.2.3. Between groups analysis

Statistical comparisons will be performed on the logarithm base 10 transformed results, in terms of RSV-A neutralizing antibody titers and frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

## a. Comparisons versus Placebo:

The 9 RSV formulations will be compared to the Placebo (control group) at Day 31 and Day 91 using an ANCOVA model with the Dunnett's adjustment method for multiplicity. The model will include the treatment group and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. Geometric mean ratios between groups and associated Dunnett's adjusted 95% CIs of the ratios will be tabulated.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

The Dunnett's test is specifically designed for situations where all groups are to be compared against one "Reference" group. It is commonly used after ANCOVA has rejected the hypothesis of equality of the means of the distributions.

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test (where=(visit=D91));
CLASS treatmnt Adj agecat;
MODEL log(titer)=treatmnt baseline agecat / ddfm=KR DDFM=KR
outpm=pred_model cl;
REPEATED / group=Adj ; /* test homogeneity of variances and consider
different variance by adjuvant content if appropriate */
LSMEANS treatmnt / ALPHA=0.05 Adjust=Dunnett pdiff=control ("Placebo")
CL;
RUN;
```

# b. Comparisons between RSV groups:

The difference between RSV groups will be evaluated using an ANCOVA model including the adjuvant content (AS01B, AS01E, Plain), the antigen dose (30, 60, 120  $\mu$ g), the visit (Day 31, Day 91) and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. The adjuvant by antigen interaction will also be tested, and included in the model if significant at 10% (p-value <10%).

Based on this global model, appropriate contrasts will be used to perform the following comparisons:

#### 1. Effect of the second vaccination:

The means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31) will be compared within each pooled group according to adjuvant content (AS01B, AS01E and Plain) (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose). Geometric mean ratios and associated 95% CIs will be tabulated

## 2. Adjuvant effect:

The adjuvant effect will be tested sequentially as follow (One-sided alpha=2.5% for each superiority test):

35

- 1. AS01B versus Plain
- 2 AS01E versus Plain
- 3. AS01B versus AS01E.

Geometric mean ratios and their 95% CIs will be computed for each comparison.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

The same comparisons will also be performed by age category.

3. Antigen dose-response: test linear and quadratic effect of the antigen dose. Depending on significance of those 2 effects, ANCOVA t-tests might be done to demonstrate superiority of 120 µg or 60 µg.

Geometric mean ratios and their 95% CIs will be computed for each pairwise comparison within each adjuvant content family (120 µg vs 60 µg, 120 µg vs 30 µg, 60 µg vs 30 µg for Plain, AS01E and AS01B groups).

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test;
  class Adj(1B, 1E, PL) Ag(30, 60, 120) visit(PD1, PD2) subject agecat;
  model log(titer) = Adj Ag visit Adj*Ag Adj*visit Ag*visit Adj*Ag*visit
baseline baseline*visit agecat / DDFM=KR S outpm=pred_model cl;
  REPEATED visit / SUBJECT=subject type=unr group=Adj;
  /* test homogeneity of variances and consider different variance by
  adjuvant content if appropriate */

  LSMEANS Adj*visit /E slice=visit CL PDIFF ALPHA=0.05; /*option E to see
  coefficients assigned to each effect */
  LSMEANS Adj*visit /E slice=Adj CL PDIFF ALPHA=0.05;
  LSMEANS Adj*ag*visit / slice=visit CL PDIFF ALPHA=0.05;
```

The inferential analysis on the RSVPreF3-specific CD4+ T cells will be performed on the log-transformation frequency of the CD4+ T cells expressing at least 2 markers (background or induction) computed by adding an offset of 0.5 cells to the number of activated CD4+ T cells (Delta method, see below). These transformations are deemed appropriate for further inferential analyses provided the incidence of activated CD4+ T-cells is below 4%.

Considering:

$$X_{ijk} = \log \left( \frac{n_{background}^{2+} + 0.5}{N_{Background}^{CD4}} \right), \text{ the log background frequency, and}$$

$$Y_{ijk} = \log \left( \frac{n_{lnduction}^{2+} + 0.5}{N_{lnduction}^{CD4}} \right), \text{ the log induction frequency}$$

The following model can be used to analyse the log-transformed ratio between induction and background frequencies, and provide estimates of the RSVPreF3-specific frequency (Delta Method- Inference on Induction/background data):

$$\begin{aligned} Y_{ijk} &= \mu_{jk} + \alpha_{j}.y_{i0k} + \beta.x_{ijk} + \varepsilon_{ijk}, \text{ with} \\ &(\overline{Y_{jk} - x_{jk}})\Big|_{\overline{y}_{0},\overline{x}} = \mu_{jk} + \alpha_{j}.\overline{y}_{0} + \beta.\overline{x}, \text{ LS means conditional to } \overline{y}_{0} \text{ and } \overline{x} \end{aligned}$$

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

where:

i, j, k=subject i, visit j, group k;  $\bar{y}_0$ = mean log induction frequency at pre-vaccination,

 $\bar{x}$  = mean log background after vaccination.

Note: This analysis is assuming that the background is the same for all groups and all timepoints. This assumption will be checked during the analysis.

Geometric means (GMs) of post-vaccination RSVPreF3-specific CD4+ T cell frequency and 95% CIs, will be calculated conditionally to the means of the pre-vaccination log-transformed CD4+ T cell frequency following induction with RSVPreF3 and the post-vaccination log-transformed CD4+ T cell frequency under background conditions.

The test and the 95% CIs for treatment comparisons will be calculated according to the delta method on the log-transformed ratio of RSVPref3-specific frequency relative to the background frequency estimates:

$$\hat{Z}_{jk} = 10^{\hat{}}(\hat{Y}_{jk} - \bar{x}) - 1 = \frac{10^{\hat{}}(\hat{Y}_{jk}) - 10^{\hat{}}(\bar{x})}{10^{\hat{}}(\bar{x})}$$
, and

$$Log(\hat{W}_{jk}) = Log\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right) = Log\left(\frac{10^{\wedge}(\hat{Y}_{jk_2}) - 10^{\wedge}(\bar{x})}{10^{\wedge}(\hat{Y}_{jk_1}) - 10^{\wedge}(\bar{x})}\right), \text{ where}$$

 $\hat{Z}_{jk}$  = mean increase from background to induction frequency relative to background frequency at visit j for treatment k, and

 $\hat{W}_{jk}$  = vaccine effect on the antigen specific frequency following adjustment for background frequency.

# Algorithm for calculations of Confidence Intervals of antigen-specific CMI response using the Delta-Method

Analysis results transformations:

- 1. The LSM and CI are back-transformed on the original scale to provide Geometric Mean Ratios of the induction frequency over background frequency. (Induction freq GM / Background freq GM)
- 2. Unity is removed from the Geometric Mean Ratios & CI ((Induction freq GM Background freq GM) / Background freq GM)
- 3. The result in 2 is multiplied by the geometric mean of background frequency used to calculate the LSM to provide the geometric means for the antigen-specific frequency.

(Induction freq GM – Background freq GM)

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- 4. The log-transformed of the result in 2 is calculated and the difference between test group and control group is calculated.
  Log(Induction\_freq GM\_test Background\_freq GM) Log(Induction\_freq GM\_control Background\_freq GM)
- 5. The confidence interval of the result in 4 is calculated through the delta-method, using student-t distribution and the number of degree of freedom provided by MIXED for the difference in LSM
- The result in 4 is back-transformed to original scale to provide the fold-increase in the frequency of antigen-specific frequency.
   (Induction\_freq GM\_t Background\_freq GM) /
   (Induction\_freq GM c Background\_freq GM)

# 5.4. Analysis of safety and reactogenicity

# 5.4.1. Analysis of safety and reactogenicity planned in the protocol

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for Grade 3 non-serious AEs.

The percentage of subjects with any AE (solicited and unsolicited) resulting in a medically attended visit during the 30-day follow-up period will also be tabulated after each dose and overall.

The percentage of subjects reporting each individual solicited local AE (any grade and Grade 3) and solicited general AE (any grade, Grade 3, any related and Grade 3 related) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.

For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall. Similar tabulations will be performed for any fever with a causal relationship to vaccination and for Grade 3 (> 39.0°C/102.2°F) causally related fever.

For each group and for each hematology and biochemistry parameter:

- The percentage of subjects having hematology and biochemistry results below or above the laboratory normal ranges will be tabulated by time point.
- The summary of grading post-vaccination will be tabulated versus baseline. (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX C in the protocol. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

The percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

The percentage of subjects with at least one report of SAE classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. SAEs will also be described in detail.

For Part A only, pregnancy and pregnancy outcomes will be listed (if applicable).

For Part B only, the percentage of subjects with at least one pIMD classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. PIMDs will also be described in detail.

The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall.

The analysis of safety will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years in Part B only).

## 5.4.2. Additional considerations

All analyses will be descriptive and will be based on the Exposed Set (ES).

Compliance in completing solicited adverse events information will be tabulated after each dose and overall.

The percentage of subjects with at least **one local solicited** AE, with at least **one general solicited** AE and with **any solicited** AE during the 7-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, and for Grade 3 AEs considered related to vaccination.

The number of days with solicited symptoms reported during the **7-day follow-up period** will be tabulated for each solicited adverse event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

The same tabulation will be done for Grade 3 symptoms, and also during **the whole post-vaccination period** (to include the total number of days for symptoms ongoing beyond the follow-up period).

The incidence of each solicited symptom (any grade and grade 3) will also be represented graphically per group and per dose.

Analysis of solicited symptoms will also be done:

- on the **pooled groups according to adjuvant content** (AS01B, AS01E, Plain), overall and by age category.
- On symptoms reported during the 4-day period, i.e. on the day of vaccination and 3 subsequent days, for each group after each dose and overall.

## 5.4.2.1. Solicited Adverse Events

Solicited adverse events will be reported daily during the 7-day (from Day 1 to Day 7) follow up period after each vaccination, using structured diaries. Missing or non-evaluable measurements will not be replaced.

In order to summarize the data, the maximum intensity of local injection site redness/swelling (in mm) and fever (in °C) will be categorized as follows:

| Grading | Redness/swelling | Fever |
|---------|------------------|-----------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C (100.4°F) - ≤ 38.5°C (101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C (101.3°F) - ≤ 39.0°C (102.2°F) |
| 3: | > 100 mm | > 39.0°C (102.2°F) |

Fever is defined as temperature  $\geq 38.0^{\circ}\text{C} / 100.4^{\circ}\text{F}$  (regardless of the location of measurement). The preferred location for measuring temperature in this study will be the oral cavity. Body temperature will also be summarized by 0.5°C increments as follows:  $\geq 38.0, >38.5, >39.0, >39.5, >40.0$ °C.

Each subject's data will be summarized according to the maximal severity observed during the follow-up period for each adverse event and each dose, followed by a summary across subjects and across doses.

## 5.4.2.2. Unsolicited Adverse Events

When an unsolicited adverse event occurs more than once for a subject, the maximal severity and strongest relationship to the vaccine group will be counted. The selection of unsolicited AEs reported during the follow-up period will be done using the day of onset.

The analysis of unsolicited adverse events includes the following categories:

- Any unsolicited adverse event.
- Possibly related unsolicited adverse events.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

- Grade 3 unsolicited adverse events
- Grade 3 possibly related unsolicited adverse events.
- Serious adverse events (SAEs)
- Possibly related SAEs.
- Potential Immune-Mediated disease (pIMDs, in Part B only)
- Medically attended adverse events
- SAEs and pIMDs reported during the entire study period will be tabulated.
- In addition, the following time periods will be considered to report SAEs/pIMDs at the first and second analyses (E1 02 and E1 03, see section 7.1):
- from Dose 1 up to 30 days post dose 2 (or up to 90 days post dose 1 for subjects who did not received the second dose)
- from Dose 1 up to 6 months\* post dose 2 (or up to 8 months\* post dose 1 for subjects who did not received the second dose).
- From Dose 1 up to Data lock point, in order to report all SAEs/pIMDs reported at the time of analysis.
  - \* months will be converted in days in order to select the events for the output tables.
- Listing of AEs/SAEs leading premature withdrawal from study or to interruption of vaccination will be described in detail.

## 5.4.2.3. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10015150 | Erythema |
| Swelling | 10053425 | Swelling at injection site |
| Fatigue | 10016256 | Fatigue |
| Fever | 10016558 | Fever |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Headache | 10019211 | Headache |
| Myalgia | 10028411 | Myalgia |
| Shivering | 10040558 | Shivering |
| Arthralgia | 10003239 | Arthralgia |

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 5.4.2.4. Clinical Safety Laboratory Investigations

In case of invalid or missing results or clinically significant grade 3 and above abnormal laboratory findings, a repeat testing may be done to confirm the first result (see Protocol section 7.1.4). For the analysis, the following rules will be applied:

- In general, the first result will be considered, except if this result is missing.
- In case of retesting for a grade 3 at pre-vaccination, the retesting will be considered if the result is < grade 3.
- If result at Visit 1 is missing, the result of the screening will be used as baseline in the analysis.

#### 5.4.2.5. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

## 5.5. Analysis of RTI for Part B

# 5.5.1. Analysis of RTI planned in the protocol

The analysis will be performed on the ES.

Any RTI episode for which a visit for the assessment of potential RSV-RTI has been performed (with nasal/throat swab sampling) will be considered for the analysis. The assessment of RSV infection will be performed using qRT-PCR on nasal/throat swabs separately for samples collected by the subject and those collected by an appropriately qualified person (i.e., medical or nursing) at the assessment visit.

The proportion of subjects with at least one RSV-associated RTI (with 95 % CI) will be calculated by group.

Descriptive analyses (mean, median, min, max) of viral load assessed by quantitative PCR (RSV-A/B) of RSV-RTI will be performed by study group.

The incidence rate of all-cause RTI (with 95% CI) will be calculated by group. These will also be presented by co-infection identified by multiplex PCR.

#### 5.5.2. Additional considerations

The mean viral load of the RSV positive-RTI samples will also be reported by collection method (at assessment visit or at home) and by collection time (0-2, 3-4, >4 days between RTI onset date of symptoms and collection date).

Information collected at assessment visit will be described for RSV RTI episodes versus Non-RSV RTI episodes, as tested by qRT-PCR on nasal/throat swabs collected at assessment visit. It will include: vital signs, clinical symptoms, self-collected nasal swab result, medically attended visit and SAE related to the episode.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

RTI episodes will be described in detail in a listing. In addition, baseline RSV A Neutralizing antibody titer (GMT and 95% CIs) will be presented graphically by RTI episode status (RSV-RTI vs Non RSV-RTI vs No RTI).

## 6. ANALYSIS INTERPRETATION

All analyses will be descriptive with the aim to characterize the difference in safety/reactogenicity or immunogenicity between groups.

All comparisons will be exploratory. They should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons, except for the comparisons of all RSV formulations vs Placebo (Dunnett's adjustment).

## 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The analyses will be performed stepwise:

- A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints up to Day 91 are available (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). This will include results from all subjects in Part A and Part B. This analysis will be considered as final for those endpoints. A clinical study report will be written.
  - At this point, the statistician will be unblinded (i.e., individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblind some specific subjects, the study will be considered as single-blind from this point onwards, with subjects remaining blinded up to study end (Visit 8, Month 14). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.
- A second analysis will be performed when all safety data up to Month 8 (Visit 7) are available (data as clean as possible). At this time, the following analyses will be performed:
  - The safety analysis of data up to 6 months post-Dose 2.
  - The analysis of all qPCR data available at that time.
  - The analysis of laboratory results that may become available at that time.
- A third immunogenicity analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 8 are available, to evaluate the persistence up to 6 months post-Dose 2 in Part B.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

• A fourth analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 14 (Visit 8) are available for the subjects enrolled in Step 1 of Part B. This analysis will include any additional laboratory results that may become available at that time.

No individual listings will be provided before the final end of study analysis.

• The final end of study analysis will be performed when all data for at least primary and secondary endpoints up to study conclusion are available (Month 14). All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage. An integrated clinical study report containing all available data will be written and made available to the investigators.

If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These data will be documented in annex(es) to the study report and will be made available to the investigators at that time.

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=public posting, SR=study<br>report, internal) | Reference for TFL TOC |
|---|---|---|---|
| Final analysis | E1_01 | SR, CTRS | See column A in TFL TOC |
| Analysis up to Day 91 | E1_02 | SR, CTRS | See column B in TFL TOC |
| Analysis up to Month 8 (safety and PCR) | E1_03 | Internal | See column C in TFL TOC |
| Analysis up to Month 8 (immuno) | E1_04 | Internal | See column D in TFL TOC |
| Analysis up to Month 14 (Part B Step 1) | E1_05 | Internal | See column E in TFL TOC |

# 7.2. Statistical considerations for interim analyses

All confirmatory analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 8. CHANGES FROM PLANNED ANALYSES

## Statistical analyses

The fold-increase parameter for CMI (post over pre-vaccination) that will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI has been adapted as follows:

• Geometric mean ratios *Fold increase (Post over pre-vaccination)* of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, at each post-vaccination time point over pre-vaccination (Day 1) will be tabulated with 95% CI as measured by ICS using *PBMCs*.

This analysis was also added for the Memory B cells:

• Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

All additional analysis planned compared to protocol are described in the "Additional considerations sections". The mains ones to be included in the CSR are also described below (changes indicated in bold):

- Demography and baseline characteristics will be summarized *by country*.
- Vital signs at baseline will be described by group using descriptive statistics.
- Exposure to study vaccine will be tabulated by group and by vaccine
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV neutralizing antibody titers will be reported for RSV-A *and RSV B*.
- Comparisons with Placebo will be done *at Day 31* and Day 91, for both RSV A Neutralizing antibody *and CD4+ T cells expressing at least 2 markers*.
- Analyses of solicited symptoms were added: incidence of any/local/general solicited AEs, number of days with solicited AEs, analysis on pooled groups according to adjuvant content.
- RTI episodes: analysis of viral load by collection method and collection time was added, as well as the description of signs and symptoms for RSV-RTI vs Non-RSV RTI cases.
- Analysis of hMPV neutralizing antibody titers on all subjects in Part A and on a subset of subjects in Part B.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Sequence of analyses

The wording of the 2<sup>nd</sup> analysis have been adapted as follows to allow the descriptive analysis of any additional immunogenicity results available for all subjects or for part of them:

- A second analysis will be performed when all safety data up to Month 8 (Visit 7) are available (data as clean as possible). At this time, the following analyses will be performed:
  - The safety analysis of data up to 6 months post-Dose 2.
  - The analysis of all qPCR data available at that time.
  - The analysis of laboratory results that may become available at that time.

## Sensitivity analysis

An issue in the randomization was identified on 23<sup>rd</sup> of July, and was identified as Significant Quality Issue (SQI) on the 6<sup>th</sup> of November 2019.

Randomization were performed in SBIR to create "placeholders"

- 1. For subjects whose eligibility was not yet confirmed
- 2. For subjects who were identified and whose ICF was not yet signed
- 3. For subjects not yet identified

This was not allowed neither based on the protocol, nor by consulting the central team.

As this issue might have an impact on the randomization, a sensitivity analysis will be performed excluding subjects who were randomized after the 23<sup>rd</sup> of July (randomization date >= 23JUL2019), for immunogenicity secondary endpoints at the time of first analysis (table template 17 and 22).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1 (Business rules for standard data derivations and statistical methods).

# 9.1. Handling of missing data

## 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- Adverse event start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1<sup>st</sup> of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
  - Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
  - Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

47

208851 | Statistical Analysis Plan Amendment 1 27 Jan 2020 | TMF-1608921 | 2.0

## CONFIDENTIAL

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 9.2. Duration of events

When a solicited AE is ongoing at the end of the solicited follow up period (Day 7), the following rules will be applied:

- If the event is present at Day 7 and information is available at each day up to the end of the event: count number of days with event up to last day reported
- If information is missing at several days between the first day with the event and the end of event: count missing days as days with an event (worst case scenario)
- For Grade 3 AEs: take into account the grading of the last day with AE reported (last observation carried forward)

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

# 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2. the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one.

## 10.1.2. Handling of missing data

## 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in section 9.1.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

#### 10.1.2.3. Daily recording of solicited symptoms

#### 10.1.2.3.1. Studies with electronic diaries

For studies using electronic diaries for the collection of solicited symptoms, symptoms will be considered present only when a daily recording of grade 1 or more is present.

49
208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

### 10.1.3. Data derivation

### 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

### 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) = 
$$((Temperature (Fahrenheit) - 32) \times 5)/9$$

Conversion of temperature from °Fahrenheit to °C will be performed according to SDTM specifications.

### 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off and value is <=ULOQ | value |
| "value" and value is > ULOQ | ULOQ* |
| All other cases | missing |

<sup>\*</sup>This rule will be used to computed descriptive statistics (GMTs, fold increase,etc). All values might be displayed in RCCs and scatter plots with individual results.

50

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 10.1.3.4. Geometric mean titers (GMTs) and concentrations (GMCs)

Geometric Mean Titer (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Antibody titers or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

### 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the symptom reported at grade 1 or higher.

See also specific rules for ongoing symptoms in section 9.2.

### 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

### 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 10.1.4. Display of decimals

### 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with one decimal.

Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22.2% |
| 1/45 | 2.2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.

Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

### 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minima of transformed body temperatures will be displayed with one decimal.

52

27-JAN-2020

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 10.1.4.3. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

### 10.1.5. Statistical methodology

### 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

### 10.1.5.2. Adjusted GMT or GMC ratios

When between-group GMT or GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

### 10.2. TFL ToC

The TFL TOC provides the list of tables/figures/listings that will be generated at each analysis. It can be found in eTMF folder section 11.01.01.

The mock tables/figures referred under column named 'layout' can be found in section 12.

### 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 12. STUDY MOCK TFLS

The following drafted standard and study specific mocks will be used. Note that standard templates might be updated based on the last version of the standard catalogue used at the time of analysis. Titles and footnotes will be adapted accordingly.

The data display, title and footnotes are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

### 12.1. Demography

Template Table 1 Summary of demography and baseline characteristics (Exposed Set)

| | _ | <each group=""><br/>N=XXXX</each> | | al<br>(XX |
|---|---|---|---|---|
| | Value or n | % | Value or n | % |
| Age (years) at first vaccination | | | | |
| N | XXX | | XXX | |
| Mean | XXX.X | | XXX.X | |
| Standard Deviation | XXX.X | | XXX.X | |
| Median | XXX.X | | XXX.X | |
| Minimum | XXX | | XXX | |
| Maximum | XXX | | XXX | |
| Sex | | | | |
| Male | XXX | XX.X | XXX | XX.X |
| Female | XXX | XX.X | XXX | XX.X |
| Ethnicity | | | | |
| <each ethnicity=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Race | | | | |
| <each race=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Age category | | | | |
| <each age="" category=""></each> | XXX | XX.X | XXX | XX.X |
| CMV status | | | | |
| Positive | XXX | XX.X | XXX | XX.X |
| Equivocal | XXX | XX.X | XXX | XX.X |
| Negative | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Table 2 Number of subjects by country and center (Exposed Set)

| | | <each group=""><br/>N=XXXX</each> | | To<br>N=X | tal<br>XXX |
|---|---|---|---|---|---|
| Country | Center-Investigator Name | n | % | n | % |
| <each country=""></each> | <each center-investigator="" name=""></each> | XXX | XX.X | XXX | XX.X |
| | All | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given center or country

 $% = (n/N) \times 100$ 

### Template Table 3 Number of subjects by study steps (Exposed Set)

| | <each group=""><br/>N=XXXX</each> | | | Total<br>=XXXX |
|---------------|-----------------------------------|---|---|----------------|
| Steps | n | % | N | % |
| Part A | | | | |
| Part B Step 1 | | | | |
| Part B Step 2 | | | | |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given category

 $% = (n/N) \times 100$ 

### Template Table 4 Summary of vital signs (Exposed Set)

| | | | <each group=""><br/>N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| EACH VISIT> | Heart rate ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Respiratory rate ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Systolic Blood pressure ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | Xxx |
| | | Maximum | XXX | Xxx |
| | Diastolic blood pressure ( <unit>)</unit> | n | XXX | Xxx |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | Xxx |
| | | Maximum | XXX | Xxx |

27-JAN-2020 55

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| Visit | Characteristics | Parameters | <each group=""> N=XXXX Value</each> | Total<br>N=XXXX<br>Value |
|---|---|---|---|---|
| | Pulse oximetry ( <unit>)</unit> | n | XXX | Xxx |
| | , , | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | Xxx |
| | | Maximum | XXX | Xxx |
| | Pre-vaccination Temperature (C) | n | | |
| | , , , | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |

Short group label = long group label

N = total number of subjects

Value = value of the considered parameter

n = number of subjects in a given category

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

### Template Table 5 Summary of study completion with reason for withdrawal (Exposed Set)

| | | <each group=""><br/>N=XXXX</each> | | tal<br>XXX |
|---|---|---|---|---|
| | n | % | n | % |
| Completed the study | XXX | XX.X | XXX | XX.X |
| Withdrawn from the study | XXX | XX.X | XXX | XX.X |
| Primary reason for withdrawal : | | | | |
| <each reason=""></each> | XXX | XX.X | XXX | XX.X |

Short group label = long group label

### Template Table 6 Summary of visit attendance (Exposed Set)

| | | | <each group=""><br/>N=XXXX</each> | | otal<br>XXXX |
|---|---|---|---|---|---|
| Visit | Status | n | % | n | % |
| <each visit=""></each> | Attended | XX | XX.X | XX | XX.X |
| | Did not attend yet | XX | XX.X | XX | XX.X |
| | Withdrawal at visit or earlier | XX | XX.X | XX | XX.X |
| | Did not attend | XX | XX.X | XX | XX.X |

Short group label = long group label

N = Number of subjects in each group or in total

n/% = number / percentage of subjects in a given category

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 7 Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set)

| Category | | <each group=""> N=XXX</each> | | | Total<br>N=XXX | |
|---|---|---|---|---|---|---|
| Sub-category | Осс | n | % | Осс | n | % |
| At least one Important Protocol Deviation | | | | | | |
| < Each category > | | | | | | |
| <each sub-category=""></each> | | | | | | |

Short group label = long group label

N = Total number of subjects

Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects with important protocol deviations

### Template Table 8 Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set)

| | Tota<br>N= | - |
|-----------------------------------------------|------------|---|
| | n | % |
| Withdrawals prior to randomization | | |
| <withdrawal 1="" reason=""></withdrawal> | | |
| <withdrawal 2="" reason=""></withdrawal> | | |
| Number of subjects included in randomized set | | |

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

### Template Table 9 Summary of subject disposition from Randomized Set to Exposed set (Randomized set)

| | < | <each group=""><br/>N=XXXX</each> | | Total<br>I=XXXX |
|---|---|---|---|---|
| | N | % | n | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Exposed set | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

27-JAN-2020 57

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 10 Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set)

| | <e< th=""><th>ach group&gt; N=XXXX</th><th></th><th colspan="2">Γotal<br/>=XXXX</th></e<> | ach group> N=XXXX | | Γotal<br>=XXXX |
|---|---|---|---|---|
| | n | % | n | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Per Protocol set at visit x | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

## Template Table 11 Summary of subject disposition from Exposed Set to End of study (Exposed set)

| | < | Each group> N=XXXX | N | Total |
|---|---|---|---|---|
| | n | % | n | % |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Number of subjects who completed the study | | | | |
| Completed with 1 dose | | | | |
| Completed with 2 doses | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 12 Deviations from protocol for age and intervals between study visits (Exposed set)

| | | | <eac< th=""><th>h group&gt;</th><th><each g<="" th=""><th>roup&gt;</th></each></th></eac<> | h group> | <each g<="" th=""><th>roup&gt;</th></each> | roup> |
|---|---|---|---|---|---|---|
| Type of interval | Interval<br>range | | Value or n | % | Value or n | % |
| | _ | NI | | 70 | | 70 |
| Age | <age range=""></age> | IN | XXX | | XXX | |
| | | n | XXX | XX.X | XXX | XX.X |
| | | Minimum | XXX | | XXX | |
| | | Maximum | XXX | | XXX | |
| <each between<="" interval="" td=""><td><interval< td=""><td>N</td><td>XXX</td><td></td><td>XXX</td><td></td></interval<></td></each> | <interval< td=""><td>N</td><td>XXX</td><td></td><td>XXX</td><td></td></interval<> | N | XXX | | XXX | |
| study visit> | range> | n | XXX | XX.X | XXX | XX.X |
| | | Minimum | XXX | | XXX | |
| | | Maximum | XXX | | XXX | |

### Template Table 13 Number of enrolled subjects by country

| | | <each group=""> N = XXX</each> | Total<br>N = XXX |
|---|---|---|---|
| Characteristics | Categories | N | n |
| Country | <each country=""></each> | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

### Template Table 14 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults [18-64 years] | | |
| | Adults [65-84 years] | | |
| | Missing | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at study vaccination unknown

59

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Table 15 Minimum and maximum visit dates <analysis set name>

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit Description | Parameter | Date | Date | Date |
| < each informed consent> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| [Randomization] | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| <each visit=""></each> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |

Short group label = long group label

### 12.2. Exposure

### **Template Table 16 Exposure to study vaccines by vaccine (Exposed Set)**

| | | | group><br>XXX | <each group=""> N=XXXX</each> | |
|---|---|---|---|---|---|
| Vaccine administered | Number of subjects receiving | n | % | n | % |
| < Vaccine A> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Total number of doses | XXX | | XXX | |
| | administered during the study | | | | |
| < Each vaccine> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Total number of doses administered during the study | XXX | | XXX | |

Short group label = long group label

N = number of subjects in each group or in total included in the considered analysis set

n = number of subjects/doses in the given category

<sup>% =</sup> percentage of subjects in the given category

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### 12.3. Immunogenicity

### 12.3.1. Within groups

## Template Table 17 Number and percentage of subjects with <antibody titer /concentration> equal to or above <cut-off unit> and <GMT/Cs> <antibody concentration> <antibody concentration> <antibody concentration> <a href="https://www.esample.com/concentration"> <a href="https://www.es

| Antibody Group | | | ; | >=cut- | off un | it | GMT/C | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | 95 | % CI | | 959 | % CI | |
| | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| <each<br>antibody&gt;</each<br> | <each<br>group&gt;</each<br> | <each timing=""></each> | | | | | | | | | | |

Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

N = Number of subjects with available results

n/% = number/percentage of subjects with titer/concentration equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

MIN/MAX = Minimum/Maximum

Short timing label = long timing label

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Figure 1 <GMT/Cs> and their 95% Cls for <antibody titers/concentrations> <analysis set name>



Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

95% CI = 95% confidence interval

Short timing label = long timing label

Note: This graph is provided as an example.

For RSV A Nab and RSVPreF3- specific IgG Ab, it will be adapted to display: all the groups (4 groups for Part A, 10 groups for Part B) and all available timepoints (4 TPs up to Day 91, 6 TPs up to study end for Part B).

If needed for Part B, this graph might be split in several graphs: either by adjuvant content vs Placebo or by antigen content vs Placebo.

Same graph will be generated for RSV B NAb with 2 timepoints (10 groups, at Days 1 and 91), for RSVPreF3 site 0 Ab with 2 groups and 2 timepoints (selected formulation and Placebo groups, at Days 1 and 91), and for hMPV Nab (10 groups, at Days 1 and 91).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 18 Geometric mean of the individual ratio of <a href="fatter: 1809">antibody titers/concentrations (units)</a> post-vaccination compared to pre-vaccination <Per Protocol Set>

| | | | | | | <gmt,c></gmt,c> | ratio | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | 95% | % CI |
| Group | N | Time point description | <gmt,c></gmt,c> | Time point description | <gmt,c></gmt,c> | Ratio order | Value | LL | UL |
| <each group=""></each> | XXX | PI(D31) | | PRE | | PI(D31) / PRE | | | |
| | | <each point="" time=""></each> | | PRE | | <time point=""> / PRE</time> | | | |

Short group label = long group label

<GMT,C> = geometric mean antibody <titer,concentration>

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

Template Table 19 Distribution of <antibody titers/concentrations> fold increase post-vaccination compared to pre-vaccination <Per Protocol Set>

| | | | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th></th><th></th><th><ea< th=""><th>ch gro</th><th>up&gt;</th><th></th></ea<></th></ea<> | ch gro | up> | | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th></th></ea<> | ch gro | up> | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 95% | 6 CI | | | | 95% | 6 CI |
| Antibody | Timing | FI | N | n | % | LL | UL | N | n | % | LL | UL |
| <each antibody=""></each> | <each timing=""></each> | < 1 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 1 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | | >= 2 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X |
| | | >= 4 | XX | XX | XX.X | xx.x | XX.X | XX | XX | XX.X | xx.x | XX.X |
| | | >= 6 | XX | XX | XX.X | xx.x | xx.x | XX | XX | XX.X | xx.x | XX.X |
| | | >= 8 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 10 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |

Short group label = long group label

FI= Fold Increase post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with <titer, concentration> fold change meeting the specified criterion

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Short timing label = long timing label

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 2 Reverse cumulative distribution curve of <antibody titers/concentrations> in the <group label> group <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: this graph is provided as an example. It will be generated by group, and will be adapted to display the 4 timepoints (PRE, D31, D61, D91) for the considered group. For Part B, same graphs will also be generated at Day 91 with groups according to adjuvant content or antigen content vs Placebo. If applicable, the upper limit of quantification will be presented (similarly to the cut-off).

For RSV B Nab ,RSVPreF3 site 0 specific Ab and hMPV NAb, the figure will display only 2 timepoints (Days 1 and 91).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 3 Kinetics of < antibody GMT/Cs> on subjects with results available at all timepoints up to <Day 91, Month 14> <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. Template will be adapted to display all the groups (10 groups for Part B) and all the timepoints (4 TPs up to Day 91, 6 TPs up to study end).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 4 Individual results of <RSV A Neutralizing antibody titer> at <time point> versus pre-vaccination in <group label> and Placebo\_B groups <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated as follows:

- RSV A Nab at Day 31 and Day 91, for each RSV groups (18 graphs)
- RSVPref3 IgG at Day 31 and Day 91, for each RSV groups (18 graphs)
- RSV B Nab at Day 91, for the selected formulation (1 graph)

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 5 Individual results of <RSV A versus RSV B Neutralizing antibody titer> at <time point> , on pooled RSV groups <Per protocol set>



Note: this graph is provided as an example. It will be generated on pooled RSV groups as follows:

- RSV A Nab vs RSVPreF3 lgG at each timepoint
- RSV A Nab vs RSV B Nab at Pre and Day 91
- RSV B Nab vs RSVPreF3 lgG at Pre and Day 91

Correlation coefficient will be computed on Log10 transformed data.

Raw data will be presented on Log10 axes.

The same graphs will be generated on fold increase Post over Pre.

Template Table 20 Geometric mean ratios of the fold increase (Pre to Post - vaccination) between RSVPreF3 IgG antibody concentrations and <RSV-A, RSV-B> neutralising antibody titers <Per protocol set>

| | | | | | | | | | GM | ratio c | f FI |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | | 95 | % CI |
| Timepoint | mepoint Group | N | RSVPref3 | 95 | % CI | <rsv-a, b=""></rsv-a,> | 9 | 5% | Value | LL | UL |
| - | | | IgG GMF | LL | UL | Nab GMF | LL | UL | | | |
| PI(D31)/PRE | <each group=""></each> | | | | | | | | | | |
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | | |
| timepoint> | | | | | | | | | | | |

Short group label = long group label

N = Number of subjects with available results at the two considered time points (post and pre) for both RSVPreF3 lgG and <RSV-A, B> Nab

GMF = Geometric mean fold increase Pre to Post-vaccination

GM ratio of FI=Geometric mean ratio of fold increase (Pre to Post)

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 6 Individual results of the fold increase (post over prevaccination) of RSVPreF3 IgG antibody concentrations versus <RSV A, RSV B> neutralizing antibody titers at <time point> in <group label> <Per protocol set>



Short group label = long group label

Note: This graph is provided as an example. It will be generated as follows:

- Y axis=RSVPreF3 IgG vs X axis=RSV A Nab, at Days 31 and 91, for each RSV group (18 graphs)
- Y axis= RSVPreF3 IgG vs X axis=RSV B Nab at Day 91, for the selected formulation (1 graph)
- Axes will be in Log10.

Template Table 21 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immune Marker | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></at> | <each timing=""></each> | N | XXXX | XXXX |
| markers> | | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Note: this table will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Table 22 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by pre-vaccination category <Per Protocol Set>

| | | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|---|
| Immune | Pre-vaccination status | | | | |
| Marker | | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<></td></at> | <q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<> | <each timing=""></each> | N | XXXX | XXXX |
| markers> | | | GM | XX.X | XX.X |
| | | | SD | | |
| | | | Minimum | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X |
| | | | Median | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X |
| | [Q1-Q3] | <each timing=""></each> | <each< td=""><td></td><td></td></each<> | | |
| | | _ | parameter> | | |
| | >Q3 | | | | |
| | Total | | | | |

Short group label = long group label

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

<sup>&</sup>lt;Q1= subjects with pre-vaccination frequency < Q1 of the frequencies at pre-vaccination computed on pooled groups Q1-Q3= subjects with pre-vaccination frequency within [Q1-Q3] of the frequencies at pre-vaccination computed on pooled groups

<sup>&</sup>gt;Q3=subjects with pre-vaccination frequency < Q3 of the frequencies at pre-vaccination computed on pooled groups N= Number of subjects with available results

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 7 Boxplots with individual data of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. Depending on the analysis, it will display groups and timepoints as follows:

- Part A: 1 graph with 4 groups and 3 (D1, D31, D91) or 4 timepoints (D1, D31, D61, D91)
- Part B: 3 graphs with 4 groups (either by adjuvant content or by antigen content vs Placebo), and 3 timepoints (D1, D31, D91) or 5 timepoints (up to Month 8) or 6 timepoints (up to Month 14, only for selected Ag dose and Placebo)

This graph will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC). For Part B, the same graph will be generated for memory B-cells, with 4 groups (selected Ag dose with Plain/AS01E/AS01B, and Placebo) and 4 timepoints (PRE, D31, D91, M14).

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 8 Frequency of RSVPreF3 specific CD4+ T-cells expressing any combination of markers among IL-2, CD40L, TNFa, IFNg in <group label> group at Day 31 and Day 91 (per million of CD4+ T cells, by ICS) <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated by group and will be adapted to display Q1-Median-Q3 for each combination of the markers (15) at Day 31 and Day 91.

Template Table 23 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immune Marker | Timing | Statistic | value | Value |
| <at 2<="" least="" td=""><td><each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each></td></at> | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each> | N | XXXX | Xxxx |
| markers> | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results at both timepoints (pre and post)

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Table 24 Descriptive statistics of the frequency of RSVPreF3 specificmemory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immuno assay | Timing | Statistic | value | value |
| Memory B cells | <each timing=""></each> | N | XXXX | XXXX |
| - | | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Template Table 25 Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immuno assay | Timing | Statistic | value | value |
| Memory B cells | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>XXXX</td></each> | N | XXXX | XXXX |
| • | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Table 26 Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | <each group=""></each> | | | | | | | | <each group=""></each> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | 6 CI | | | | 95% | 6 CI | |
| Assay | Timing | FI | N | n | % | LL | UL | N | n | % | LL | UL |
| <assay name=""></assay> | <each timing=""></each> | < 2 | Xx | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 2 | Xx | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 4 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 6 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 8 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | | >= 10 | XX | XX | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |

Short group label = long group label

FI= Fold increase Post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available n/% = number/percentage of subjects with fold increase meeting the specified criterion 95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit Short timing label = long timing label

### 12.3.2. Between groups

Template Table 27 Comparisons of the 9 RSV formulations versus Placebo in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at one month post <dose 1 (Day 31), dose 2 (Day 91)> (ANCOVA model, Dunnett's test) – Part B <Per Protocol set>

| Access | Timonoint | DCV group | N | GM <t,f> ratio</t,f> | Dunne | ett's 95% CI | Dunnett's |
|---|---|---|---|---|---|---|---|
| Assay | Timepoint | RSV group | IN | (RSV over Placebo) | LL | UL | p-value |
| <assay name=""></assay> | <day 31,="" 91="" day=""></day> | 30-PLAIN_B | | | | | |
| · | | 60-PLAIN_B | | | | | |
| | | 120-PLAIN_B | | | | | |
| | | 30-AS01E_B | | | | | |
| | | 60-AS01E_B | | | | | |
| | | 120-AS01E_B | | | | | |
| | | 30-AS01B_B | | | | | |
| | | 60-AS01B_B | | | | | |
| | | 120-AS01B_B | | | | | |

Short group label = long group label

N= Number of subjects with both pre- and post-vaccination results available

GM<T,F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

RSV Vaccine is considered superior to Placebo if one-sided p-value < 0.025

Dunnett's 95% CI = 95% confidence interval based on Dunnett's adjustment, LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed

<ti>titer, frequency> as covariate, and the treatment and age category as fixed effects</ti>

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Table 28 Comparisons of the mean responses post dose 2 (Day 91)
versus post dose 1 (Day 31) in terms of <RSV A Neutralizing
antibody titers, RSVPreF3-specific CD4 T cells expressing at
least 2 markers among IL-2, CD40L, TNFa, IFNg> on pooled
groups according to adjuvant content (ANCOVA model) – Part
B <Per Protocol set >

| Λοοον | DCV group | N | GM <t,f> ratio</t,f> | 95% ( | n volue | |
|---|---|---|---|---|---|---|
| Assay | RSV group | N | (D91/D31) | LL | UL | p-value |
| <assay name=""></assay> | PLAIN_B | | | | | |
| , | AS01E_B | | | | | |
| | AS01B_B | | | | | |

Short pooled group label = long pooled group label

N= Number of subjects with results available at both timepoints

GM<T,F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

PII D91 is considered as significantly higher to PI D31 if one-sided p-value <0.025

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance); LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the adjuvant content, antigen dose and age category as fixed effects

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 29 Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) - Part B <Per Protocol set>

| | | Group 1 | | Group 2 | | | | GM <t,f> ratio (Group 1 /<br/>Group 2)</t,f> | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95% | 6 CI | | 95% ( | CI | |
| Assay | Timepoint | Group 1 | N | GM <t,f></t,f> | LL | UL | Group 2 | N | GM <t,f></t,f> | LL | UL | Value | LL | UL | p-value |
| <assay name=""></assay> | <each timing=""></each> | AS01B_B | | | | | PLAIN_B | | | | | | | | |
| | | AS01E_B | | | | | PLAIN_B | | | | | | | | |
| | | AS01B_B | | | | | AS01E_B | | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance); LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and adjuvant content, antigen dose and age category as fixed effects

Group 1 is considered superior to Group 2 if one-sided p-value <0.025

27-JAN-2020 75

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Table 30 Comparisons of the RSV groups (by antigen dose level) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) – Part B <Per Protocol set >

| | | | Gı | roup 1 | | | | Group 2 | | | | GM <t,f> rat<br/>Gro</t,f> | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 959 | % CI | | | | 959 | % CI | | 95% | CI | |
| Assay | Timepoint | Group 1 | N | GM <t,f></t,f> | LL | UL | Group 2 | N | GM <t,f></t,f> | LL | UL | Value | LL | UL | p-value |
| <assay< td=""><td><each< td=""><td>120-PLAIN_B</td><td></td><td></td><td></td><td></td><td>60-PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<></td></assay<> | <each< td=""><td>120-PLAIN_B</td><td></td><td></td><td></td><td></td><td>60-PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | 120-PLAIN_B | | | | | 60-PLAIN_B | | | | | | | | |
| name> | timing> | 120-PLAIN_B | | | | | 30-PLAIN_B | | | | | | | | |
| | | 60-PLAIN_B | | | | | 30-PLAIN_B | | | | | | | | |
| | | 120-AS01E_B | | | | | 60-AS01E_B | | | | | | | | |
| | | 120-AS01E_B | | | | | 30-AS01E_B | | | | | | | | |
| | | 60-AS01E_B | | | | | 30-AS01E_B | | | | | | | | |
| | | 120-AS01B_B | | | | | 60-AS01B_B | | | | | | | | |
| | | 120-AS01B_B | | | | | 30-AS01B_B | | | | | | | | |
| | | 60-AS01B_B | | | | | 30-AS01B_B | | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance); LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the treatment, age category and gender as fixed effects

Group 1 is considered superior to Group 2 if one-sided p-value <0.025

27-JAN-2020 76

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# Template Table 31 Parameters of the ANCOVA model for the comparison between RSV groups in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg>- Part B <analysis set name>

| Timepoint | Variable | DF | Fvalue | p-value |
|---|---|---|---|---|
| <each timepoint=""></each> | Pre-vaccination log <titer, frequency=""></titer,> | | | |
| | Age category | | | |
| | Adjuvant | | | |
| | Antigen | | | |
| | Visit | | | |
| | Linear effect of antigen | | | |
| | Quadratic effect of antigen | | | |
| | Antigen*Adjuvant | | | |

Antigen = Antigen dose (3 levels: 30, 60, 120 mcg)

Adjuvant = Adjuvant content (3 levels: no adjuvant, AS01E, AS01B)

Antigen\*Adjuvant = interaction between antigen dose and adjuvant

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed

<ti>titer, frequency > as covariate, and adjuvant content, antigen dose and age category as fixed effects DF = degrees of freedom

Interaction (Antigen \* Adjuvant) considered as statistically significant if p-value <0.100

Main factors (Pre-vaccination, antigen, adjuvant) considered as statistically significant if p-value <0.050 (model including interaction)

### 12.4. Safety

### Template Table 32 Compliance in completing solicited adverse events information (Exposed Set)

| | | <each group=""></each> | |
|---|---|---|---|
| DOSE | N | n | Compliance (%) |
| Vaccination at Visit 1 | XXX | XXX | XX.X |
| Vaccination at Visit 4 | XXX | XXX | XX.X |
| TOTAL | XXX | XXX | XX.X |

77

Short group label = long group label

N=Number of administered vaccinations

n = number of vaccinations with solicited symptom information completed

Compliance (%) =  $(n / N) \times 100$ 

27-JAN-2020

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# Template Table 33 Incidence and nature of <grade 3> symptoms (solicited and unsolicited) <with causal relationship to vaccination> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis set name>

| | | | <ea< th=""><th>ach gro</th><th>up&gt;</th><th></th><th></th><th>&lt;</th><th>Each g</th><th>roup&gt;</th><th></th></ea<> | ach gro | up> | | | < | Each g | roup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | <del>-</del> | | 6 CI | | | | 95 | % CI |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General<br>symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

<sup>95%</sup> CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# Template Table 34 Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <analysis set name>

| | | <each group=""></each> | | | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | | | 95% CI | |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

### Template Table 35 Incidence of solicited local symptoms reported during the 7day (Days 1-7) post-vaccination period following each dose and overall <analysis set name>

| | | | | | <e< th=""><th>ach g</th><th>roup&gt;</th></e<> | ach g | roup> |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % CI |
| Dose | Symptom | Type | N | n | % | LL | UL |
| DOSE 1 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| DOSE 2 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/DOSE | <each symptom=""></each> | All | | | | | |
| | , | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/SUBJECT | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

27-JAN-2020 79

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

### Template Table 36 Incidence of solicited general symptoms reported during the 7day (Days 1-7) post-vaccination period following each dose and overall <cohort name>

| | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|
| Dose | Symptom | Туре | N | n | % | LL | UL |
| OOSE 1 | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | 10701 | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | 1 6461 ( 6) | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | - | | | | |
| | | Related | | 1 | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OOSE 2 | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | 1 6461 ( 6) | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OVERALL/DOSE | <pre><each except="" fever="" symptom="" –=""></each></pre> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | T | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | 1 5 7 5 7 | ≥38.0 | - | | | | |
| | | >38.5 | - | | | | |
| | | >39.0 | - | | | | |

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| | | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|
| | | | | | | | 95 % CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OVERALL/SUBJECT | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | , | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 37 Number of days with <*local/general>* solicited symptoms during <the 7-day (Days 1-7), the whole> post-vaccination period <analysis set name>

| | | | <each group=""></each> |
|---|---|---|---|
| Dose | Symptom | Statistic | Value |
| DOSE 1 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| DOSE 2 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| OVERALL/DOSI | E <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |

Short group label = long group label n = number of doses with the symptom Q1 = 25th percentile Q3= 75th percentile

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Template Figure 9 Incidence of solicited <local, general> adverse events reported during the 7-day (Days 1-7) post-vaccination period following each dose <Exposed set>



Short group label = long group label

Note: this graph is provided as an example. It will be adapted to display the percentage of subjects reporting each local or general symptom, any grade and grade 3, by group and by dose. Template will be discussed at the time of the dryrun.

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 38 Percentage of subjects reporting the occurrence of <grade 3> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> within the 30-day (Days 1-30) post-vaccination period <analysis set name>

| | | | <each group=""> N=XXXX</each> | | | | | | Total<br>N=XXXX | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | % CI | | | | 95% | % CI |
| Primary System Organ Class | | | | | | | | | | | |
| (CODE) | Preferred Term (CODE) | n* | n | % | LL | UL | n* | N | % | LL | UL |
| | At least one symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

### Template Table 39 List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <Exposed set>

| Group | Sub. No | Country | Gender | Race | AE Description | Preferred<br>Term | SAE | Causality | Outcome | Vaccination and visit | Type of discontinuation* |
|---|---|---|---|---|---|---|---|---|---|---|---|

Short group label = long group label

27-JAN-2020 84

<sup>\*</sup> type of discontinuation refers to whether the discontinuation is a treatment discontinuation or study follow-up discontinuation

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 40 Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment <analysis set name>

| Group | Sub. No. | Gender | Country | Race | Age at onset (Year) | Verbatim | Preferred Term | Primary System Organ Class |
|---|---|---|---|---|---|---|---|---|
| <each group=""></each> | > | | | | | | | |

| Group | Sub. No. | Medical visit type | Dose | Day of onset | Duration | Intensity | Causality | Outcome | SAE (Y/N) | pIMD source |
|---|---|---|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | |
| group> | | | | | | | | | | |

Short group label = long group label

### Template Table 41 Listing of SAEs <analysis set name>

| Group | Sub. No. | Gender | Country | Race | Age at onset<br>(Year) | Verbatim | Preferred Term |
|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | |
| group> | | | | | | | |

| _ | | | | | Day of | | | _ | |
|---|---|---|---|---|---|---|---|---|---|
| Group | Sub. No. | Primary System Organ Class | Medical visit type | Dose | onset | Duration | Intensity | Causality | Outcome |
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | |
| group> | | | | | | | | | |

Short group label = long group label

27-JAN-2020 85
208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### Template Table 42 Listing of pregnancies reported during the study period in Part A <analysis set name>

| ( | iralin | Sub.<br>No. | Country | IKACA | Age at vaccination | Previous<br>Dose | between | Age at<br>delivery<br>(Year) | Date of outcome | Gestational<br>weeks at<br>birth/miscar<br>riage<br>/termination |
|---|---|---|---|---|---|---|---|---|---|---|

Short group label = long group label

LMP=Last Mentrual Period

### Template Table 43 Number and percentage of subjects taking concomitant medication during the <XX>-day (Days 1-<XX>) post-vaccination period by dose and overall <analysis set name>

| | | | | <each< th=""><th>group&gt;</th><th></th><th></th><th></th><th><eac< th=""><th>h group&gt;</th><th></th></eac<></th></each<> | group> | | | | <eac< th=""><th>h group&gt;</th><th></th></eac<> | h group> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | <9 | 5>% CI | | | | <9: | 5>% CI |
| Dose | | N | n | % | LL | UL | N | N | % | LL | UL |
| OOSE x | Any | XX | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | xx | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any | XX | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any | XX | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | xx | XX | XX.X | XX.X | XX.X | XX | Xx | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

27-JAN-2020 86

N = total number of subjects with the corresponding administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified type of concomitant medication was taken at least once during the considered period For overall/subject:

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

N = total number of subjects with at least one administered dose n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period 95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

87 27-JAN-2020

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 44 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges, 7 days post dose <1, 2> <analysis set name>

| | | | <ea< th=""><th>ach gro</th><th>up&gt;</th><th><ea< th=""><th>ach gro</th><th>up&gt;</th></ea<></th></ea<> | ach gro | up> | <ea< th=""><th>ach gro</th><th>up&gt;</th></ea<> | ach gro | up> |
|---|---|---|---|---|---|---|---|---|
| Laboratory parameter | Range indicator at<br>Baseline (PRE) | Range<br>indicator at<br>post-<br>vaccination | N | n | % | N | n | % |
| <each parameter=""></each> | UNKNOWN | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | BELOW | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | WITHIN | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |
| | ABOVE | UNKNOWN | | | | | | |
| | | BELOW | | | | | | |
| | | WITHIN | | | | | | |
| | | ABOVE | | | | | | |

Short group label = long group label

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

Baseline= Pre-vaccination at <Day 1, Day 61>

Post-vaccination = Post vaccination at <Day 8, Day 68>

## Template Table 45 Summary of hematology and biochemistry results by grade at 7 days post dose <1, 2 > versus baseline (<Day 1, Day 61>) <analysis set name>

| | | | <ea< th=""><th>up &gt;</th></ea<> | up > | |
|---|---|---|---|---|---|
| Laboratory parameter | Baseline | Post-vaccination | N | n | % |
| <each parameter=""></each> | Unknown | Unknown | | | |
| | | <each grade=""></each> | | | |
| | <each grade=""></each> | Unknown | | | |
| | | <each grade=""></each> | | | |
| | Total | Unknown | | | |
| | | <each grade=""></each> | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Baseline= Pre-vaccination at <Day 1, Day 61>

Post-vaccination = Post vaccination at <Day 8, Day 68>

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

Note: Templates 45 and 46 will be generated post dose 1 with results at Visit 2 (Day 8) versus baseline at Day 1, and post dose 2 with results at Visit 5 (Day 68) versus baseline at Day 61.

#### Template Table 46 Summary of hemoglobin change from baseline at 7 days postdose <1, 2> (Exposed set)

| | | <e< th=""><th>ach gr</th><th>oup&gt;</th></e<> | ach gr | oup> |
|---|---|---|---|---|
| Laboratory parameter | | N | n | % |
| Hemoglobin - change from baseline | UNKNOWN | | | |
| | GRADE 0 | | | |
| | GRADE 1 | | | |
| | GRADE 2 | | | |
| GRADE 3 | | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period

n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Note: This table will be generated post dose 1 with results at Visit 2 (Day 8) and Day 1 as baseline, and post dose 2 with results at Visit 5 (Day 68) and Day 61 as baseline.

Template Figure 10 Boxplot of <each hematology/biochemistry parameter> (Exposed Set)



Note: This graph is given as an example. It will be adapted to display one boxplot per group and per timepoint, all timepoints available (5 TPs: Screening, Days 1, 8, 61, 68). For Part A, one graph will be generated displaying the 4 groups. For Part B, 3 graphs will be generated displaying 4 groups: 3 RSV groups (30/60/120 -Plain, - AS01E or - AS01B) and the Placebo group.

89

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# Template Table 47 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis set name>

| | | | ich gr<br>N=XX) | • | <each group=""> N=XXXX</each> | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

Template Table 48 Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis set name>

| SAE Related SAE Fatal SAE Related Fatal | | | <eacl< th=""><th>n group</th><th>&gt;</th><th><each< th=""><th>•</th></each<></th></eacl<> | n group | > | <each< th=""><th>•</th></each<> | • | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System<br>Organ Class (CODE) | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | , | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Fatal SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | , | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related Fatal | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| SAE | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |

90

Short group label = long group label

N = number of subjects with administered dose

n/% = number/percentage of subjects reporting the symptom at least once

n\* = Number of events reported

Related = assessed by the investigator as related

27-JAN-2020

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

#### 12.5. Analysis of RTI

Template Table 49 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis set name>

| | | | <b>&lt;</b> E | ach | gro | up> | | al | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI | | | | | 95% | | | |
| Samples | RSV status | N | r | າ % | LL | UL | N | n | % | LL | UL |
| Nasal/throat swab at assessment visit | RSV+ | | | | | | | | | | |
| | RSV- | | | | | | | | | | |
| | All | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by qRT-PCR at least once

RSV-= subjects tested as RSV negative by gRT-PCR

All= subjects with at least one qRT-PCR result available

N = number of subjects in each group or in Total

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template Table 50 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis set name>

| | | | <ea< th=""><th>ach</th><th>gro</th><th>up&gt;</th><th></th><th>1</th><th colspan="2">Total</th><th></th></ea<> | ach | gro | up> | | 1 | Total | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% CI<br>N n % LL UL N | | | | | 95% | | | |
| Samples | RSV status | N | n | % | LL | UL | N | n | % | LL | UL |
| Nasal swab at home | RSV+ | | | | | | | | | | |
| | RSV- | | | | | | | | | | |
| | All | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by gRT-PCR at least once

RSV-= subjects tested as RSV negative by qRT-PCR

All= subjects with at least one qRT-PCR result available

N = number of subjects in each group

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

## Template Table 51 Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <Exposed set>

| | RSV A + | | | | | RSV B + | | | |
|---|---|---|---|---|---|---|---|---|---|
| Days after<br>RTI onset | Swab | N | n | % | mean | N | n | % | mean |
| 0-2 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |
| 3-4 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |
| >4 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |

Days after RTI onset = number of days between start of RTI symptoms and collection date

N=Number of swabs with gRT-PCR results available

n/%= number/percentage of swabs tested as RSV A/B positive by gRT-PCR

mean= mean of the viral load computed on RSV A/B positive swabs

Template Table 52 Descriptive statistics of the viral load of the RSV- confirmed RTI episodes, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <at home> <Exposed Set>

| | | <each group=""><br/>N=</each> | Total<br>N= |
|-----------|------------|-------------------------------|-------------|
| Туре | Parameters | Value | Value |
| RSV A + | N | | |
| | Mean | | |
| | Min | | |
| | Q1 | | |
| | Median | | |
| | Q3 | | |
| | Max | | |
| RSV B + | ••• | | |
| All RSV + | | | |

92

Short group label = long group label

RSV A+= RSV A positive samples by gRT-PCR

RSV B+-= RSV B positive samples by qRT-PCR

All RSV += All RSV positive samples by qRT-PCR

N = Number of swabs with qRT-PCR results available

n= number/percentage of samples in each category

Q1 and Q3 = 25th and 75th percentiles

Min/Max = Minimum/Maximum

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

# Template Table 53 Number and percentage of subjects reporting co-infections with respiratory viruses, as measured by multiplex PCR on RSV A/B positive RTI samples collected <at assessment visit, at home> <Exposed Set>

| | | | RSV I<br>N = | |
|------------------------|---|---|--------------|-------|
| | | | 9 | 5% CI |
| Categories | n | % | LL | UL |
| Influenza A Virus | | | | |
| Influenza B Virus | | | | |
| <each virus=""></each> | | | | |
| Total | | | | |

N = number of swabs tested RSV positive by qRT-PCR

### Template Table 54 Clinical signs and symptoms associated with RTI episodes (Exposed set)

| | | | SV RTI<br>=XXXX | | on RSV RTI<br>N=XXXX | | Total<br>=XXXX |
|---|---|---|---|---|---|---|---|
| Characteristics | Categories | N | % | n | % | n | % |
| Heart Rate increase (beats/min) | 10-20 | | | | | | |
| | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Respiratory rate increase (breaths/min) | 5-10 | | | | | | |
| | 10-15 | | | | | | |
| | 15-20 | | | | | | |
| | 20-25 | | | | | | |
| Systolic blood pressure increase (mmHg) | 10-20 | | | | | | |
| | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Diastolic blood pressure increase (mmHg) | 10-20 | | | | | | |
| | 20-30 | | | | | | |
| | 30-40 | | | | | | |
| | 40-50 | | | | | | |
| Oxygen saturation decrease (%) | 1-2 | | | | | | |
| | 3-4 | | | | | | |
| | 5-6 | | | | | | - |
| | 7-8 | | | | | | |
| Upper respiratory symptoms | <each symptom=""></each> | | | | | | _ |
| Lower respiratory symptoms | <each symptom=""></each> | | | | | | + |
| . , , , , | , , | | | | | | |

93

27-JAN-2020

n/% = number/percentage of swabs tested positive by multiplex in a given category

Total= number of swabs tested positive for at least one virus

LL, UL= Exact 95% Lower and Upper confidence limits

208851 (RSV-OA=ADJ-002) Statistical Analysis Plan Amendment 1

| | Categories | RSV RTI<br>N=XXXX | | Non RSV RTI<br>N=XXXX | | | Total<br>=XXXX |
|---|---|---|---|---|---|---|---|
| Characteristics | | N | % | n | % | n | % |
| qPCR result | RSV A+ | | | | | | |
| | RSV B+ | | | | | | |
| | RSV - | | | | | | |
| Self-collected Nasal swab | RSV+ | | | | | | |
| | RSV- | | | | | | |
| | NA | | | | | | |
| Medically attended visit | Emergency room | | | | | | |
| • | Hospitalisation | | | | | | |
| | Medical personnel | | | | | | |
| | None | | | | | | |
| SAE associated to the episode | Yes | | | | | | |
| · | No | | | | | | |

RSV RTI= RTI episode tested as RSV positive by qRT-PCR on nasal/throat swab collected at assessment visit Non-RSV RTI= RTI episode tested as RSV negative by qRT-PCR on nasal/throat swab collected at assessment visit N = number of RTI episodes in each category or in total

For vital signs, change from baseline (increase/decrease) will be displayed by category: category of 10 units increase for heart rate, systolic and diastolic BP, 5 units increase for respiratory rate, and 1% decrease for oxygen saturation (to be adapted at the time of dry run if needed)

n = number of RTI episodes in the corresponding category

 $<sup>% =</sup> n / N \times 100$ 

208851 (RSV-OA=ADJ-002) SAP Amendment 1 Final

#### Template Table 55 Listing of RTI episodes reported during RTI surveillance in Part B (Exposed set)

| Group | Sub. | Age at | Sex | Episode nb | Start | End | Date of | Nb of signs | Date | RSV A | RSV B | Date | RSV-A | RSV-B | Medically | SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | No. | Dose 1 | | | date of | date of | assessment | and | nasal | positive | positive | nasal | positive | positive | attended | related to |
| | | | | | episode | episode | visit | symptoms | swab | (site) | (site) | swab at | (home) | (home) | visit | RTI |
| | | | | | | | | | on site | | | home | | | | episode |
| | | | | | | | | | | Yes/No | Yes/No | | Yes/No | Yes/No | | Yes/No |

Short group label = long group label

27-JAN-2020 95

208851 (RSV-OA=ADJ-002) SAP Amendment 1 Final

Template Figure 11 GMTs and 95% CIs of RSV A Neutralizing antibody titer at baseline for subjects reporting RTI episodes (RSV RTI vs or non RSV RTI vs No RTI), by groups pooled according to the adjuvant content <Exposed Set>



This graph is provided as an example, template will be finalized at the time of the dry-run. It will display the GMTs and 95% CIs for subjects reporting confirmed RSV RTI episodes vs subjects reporting Non-RSV RTI episodes vs subjects who did not report any RTI episode (NON RTI), in the RSV groups pooled according to the adjuvant content (Plain, AS01E, AS01B).

96

27-JAN-2020

208851 (RSV-OA=ADJ-002) SAP Amendment 1 Final

#### 12.6. Additional templates (Amendment 1)

### Template Table 56 Distribution of hematology and biochemistry parameters at baseline with respect to normal laboratory ranges <analysis set name>

| | | | ach grou | p> | <each group=""></each> | | |
|---|---|---|---|---|---|---|---|
| Laboratory parameter | Range indicator at baseline | N | n | % | N | n | % |
| <each parameter=""></each> | UNKNOWN | | | | | | |
| | BELOW | | | | | | |
| | WITHIN | | | | | | |
| | ABOVE | | | | | | |

Short group label = long group label

N = number of subjects with available results for the specified laboratory parameter in a given baseline category n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter

### Template Table 57 Summary of follow-up time (in days) up to <DLP or last contact> (Exposed Set)

| | <each group=""> N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|
| | Value | Value |
| Number of days in the study | | |
| N | XXX | Xxx |
| Mean | XXX.X | XXX.X |
| Median | XXX.X | XXX.X |
| Minimum | XXX | Xxx |
| Maximum | XXX | Xxx |

Short group label = long group label

N = total number of subjects

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

208851 (RSV-OA=ADJ-002) SAP Amendment 1 Final

#### Template Table 58 Summary of subjects by unsolicited adverse event category

| | | ch group><br>I=XXXX |
|---|---|---|
| At least one uncellaited adverse event within 20 day of any vessingtion | n* | Xxx |
| At least one unsolicited adverse event within 30-day of any vaccination | | XXX |
| | n<br>% | XX.X |
| | 95% CI | |
| At least one related uncelligited adverse event within 20 day of any vaccination | 95% CI<br>n* | (xx.x ; xx.x) |
| At least one related unsolicited adverse event within 30-day of any vaccination | | XXX |
| | n<br>% | XXX |
| | | XX.X |
| | 95% CI | (xx.x; xx.x) |
| At least one medically attended unsolicited adverse event within 30-day of any | n* | XXX |
| vaccination | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| At least one serious unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | n* | XXX |
| a load one concae anconcae autoros cront ap to 21. Crotaey one | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| At least one serious related uncellisited adverse event cur to DLD or attidu and | n* | NOW. |
| At least one serious related unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | | XXX |
| | n<br>o/ | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| At least one potential immune-mediated disorder (pIMD) <up dlp="" or="" study<="" td="" to=""><td>n*</td><td>XXX</td></up> | n* | XXX |
| end> | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |
| At least one related potential immune-mediated disorder (pIMD) <up dlp="" or<="" td="" to=""><td>n*</td><td>XXX</td></up> | n* | XXX |
| study end> | <b>-</b> | |
| Study Grids | //<br>% | XXX |
| | 95% CI | XX.X |
| | 90 % CI | (xx.x; xx.x) |
| At least one fatal unsolicited adverse event <up dlp="" end="" or="" study="" to=""></up> | n* | xxx |
| | n | XXX |
| | % | XX.X |
| | 95% CI | (xx.x; xx.x) |

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once 95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

| _ | Statisticai Analysis Plan Fina |
|---|---|
| <b>gsk</b> GlaxoSmithKline | Statistical Analysis Plan |
| Detailed Title: | A Phase I/II, randomized, placebo-controlled, observer-blind, multicenter study to evaluate the safety, reactogenicity and immunogenicity of GSK Biologicals' investigational respiratory syncytial virus (RSV) vaccine (adjuvanted with AS01 <sub>E</sub> or AS01 <sub>B</sub> or unadjuvanted) when administered intramuscularly according to a 0, 2 month schedule in adults aged 18-40 or 60-80 years. |
| eTrack study number and Abbreviated Title | 208851 (RSV OA=ADJ-002) |
| Scope: | All data pertaining to the above study (except IDMC analyses) |
| Date of Statistical Analysis<br>Plan | Final: 14 January 2019 |
| Co-ordinating author: | (Statistician) |
| Reviewed by: | PPD (Clinical and Epidemiology Project Lead) PPD (Clinical Research and Development Lead) PPD (Lead statistician) PPD (Lead statistical analyst) PPD (Scientific writer) PPD (Stat Peer Reviewer) PPD (Regulatory Affairs) PPD (SERM physician) PPD (Safety scientist) PPD (Public disclosure representative) PPD (CLS – Clinical Read-outs) PPD (CMI Expert representative) |
| Approved by: | PPD (Clinical and Epidemiology Project Lead) PPD (Lead statistician) PPD (Statistician) PPD (Lead Scientific writer) PPD (Lead stat Analyst) |

APP 9000058193 Statistical Analysis Plan Template (Effective date: 12 November 2018)

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

#### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| LIS | T OF A | BBREVIA | ATIONS | 12 |
| 1. | DOC | JMENT H | ISTORY | 14 |
| 2. | STUD | Y DESIG | N | 14 |
| _ | 0D 1E | | TNDDOINTO | 04 |
| 3. | 3.1. | | ENDPOINTSes | |
| | J. 1. | 3.1.1. | Primary objective | |
| | | 3.1.2. | Secondary objectives | |
| | | 3.1.3. | Tertiary objectives | |
| | 3.2. | Endpoir | nts | |
| | | 3.2.1. | Primary endpoints | 22 |
| | | 3.2.2. | Secondary endpoints | |
| | | 3.2.3. | Tertiary endpoints | 23 |
| 4. | ANAL | YSIS SET | TS | 24 |
| | 4.1. | Definition | on | 24 |
| | | 4.1.1. | Exposed Set | 24 |
| | | 4.1.2. | , , | |
| | 4.2. | | for eliminating data from Analysis Sets | |
| | | 4.2.1. | | |
| | | 4.2.2. | Elimination from Per-protocol analysis Set (PPS) | |
| | | | 4.2.2.1. Excluded subjects | 25 |
| 5. | STAT | ISTICAL A | ANALYSES | 2 <mark>7</mark> |
| | 5.1. | Demogr | aphy | 2 <mark>7</mark> |
| | | 5.1.1. | Analysis of demographics/baseline characteristics planned | |
| | | | in the protocol | |
| | | 5.1.2. | | |
| | 5.2. | | re | 28 |
| | | 5.2.1.<br>5.2.2. | <b>√</b> 1 1 1 | 28 |
| | 5.3. | | Additional considerations | |
| | 5.5. | 5.3.1. | ogenicityAnalysis of immunogenicity planned in the protocol | |
| | | 0.0.1. | 5.3.1.1. Within groups evaluation - humoral immune | 20 |
| | | | response | 28 |
| | | | 5.3.1.2. Within groups evaluation - Cell-mediated | |
| | | | immune response | 29 |
| | | | 5.3.1.3. Between groups evaluation (Part B only) | |
| | | 5.3.2. | Additional considerations | 31 |
| | | | 5.3.2.1. Within groups – humoral immune response | 31 |
| | | | 5.3.2.2. Within groups – Cell-mediated immune | |
| | | | response | |
| | <b>-</b> 4 | A 1 | 5.3.2.3. Between groups analysis | |
| | 5.4. | | s of safety and reactogenicity | 36 |
| | | 5.4.1. | Analysis of safety and reactogenicity planned in the protocol | 36 |
| | | 5.4.2. | Additional considerations | |
| | | O. 1.Z. | , taditional conductations | |

| | | | 5.4.2.1. | Solicited Adverse Events | |
|---|---|---|---|---|---|
| | | | 5.4.2.2. | Unsolicited Adverse Events | 39 |
| | | | 5.4.2.3. | Combined Solicited and Unsolicited Adverse Events | 39 |
| | | | 5.4.2.4. | Clinical Safety Laboratory Investigations | |
| | | | 5.4.2.5. | Concomitant Medication | |
| | 5.5. | Analysis | | Part B | |
| | | 5.5.1. | | of RTI planned in the protocol | |
| | | 5.5.2. | Additional | considerations | 41 |
| 6. | ANAL' | YSIS INTE | ERPRETAT | TON | 41 |
| 7. | CONE | UCT OF A | ANALYSES | S | 41 |
| | 7.1. | | | es | |
| | 7.2. | Statistical considerations for interim analyses | | | |
| 8. | CHAN | GES FRO | M PLANNI | ED ANALYSES | 43 |
| 9. | | | | ERIVATION RULES AND STATISTICAL | 4.4 |
| | | | | data | |
| | 9.1. | | | data | |
| | | 5.1.1. | Dates | | |
| 10. | | XES | | | |
| | 10.1. | | | tandard data derivations and statistical methods | |
| | | | | events to vaccine doses | |
| | | 10.1.2. | | of missing data<br>Dates | |
| | | | | Laboratory data | |
| | | | 10.1.2.2. | | |
| | | | 10.1.2.5. | 10.1.2.3.1. Studies with electronic diaries | |
| | | | 10.1.2.4. | | |
| | | 10.1.3. | - | ration | |
| | | | | Age at vaccination in years | |
| | | | | Temperature | |
| | | | 10.1.3.4. | Geometric mean titers (GMTs) and | |
| | | | | concentrations (GMCs) | 47 |
| | | | 10.1.3.5. | Onset day | |
| | | | | Duration of events | 47 |
| | | | 10.1.3.7. | Counting rules for combining solicited and | |
| | | | | unsolicited adverse events | 47 |
| | | | 10.1.3.8. | Counting rules for occurrences of solicited | 47 |
| | | 10.1.4. | Dienlay of | adverse eventsdecimals | |
| | | 10.1.4. | 10.1.4.1. | | |
| | | | 10.1.4.1. | | |
| | | | 10.1.4.2. | | |
| | | 10.1.5. | | methodology | |
| | | | | Exact confidence intervals around proportions | |
| | | | | Adjusted GMT or GMC ratios | |
| | 10.2. | TFL ToC | | | |

| | | | 208851 (RSV OA=ADJ-002)<br>Statistical Analysis Plan Final |
|---|---|---|---|
| 11. | REFE | RENCES | 49 |
| 12. | STUD | Y MOCK TFLS | 50 |
| | 12.1. | Demography | 50 |
| | | Exposure | |
| | | Immunogenicity | |
| | | 12.3.1. Within groups | |
| | | 12.3.2. Between groups | |
| | 12.4. | Safety | |
| | | Analysis of RTI | |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

#### **LIST OF TABLES**

| | | PAGE |
|---------|--------------------|------|
| Table 1 | Groups description | 18 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

#### **LIST OF FIGURES**

| | | PAGE |
|----------|--------------|--------|
| Figure 1 | Study design | <br>14 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

#### **LIST OF TEMPLATES**

| | F | PAGE |
|---|---|---|
| Template 1 | Summary of demography and baseline characteristics (Exposed Set) | 50 |
| Template 2 | Number of subjects by country and center (Exposed Set) | 51 |
| Template 3 | Number of subjects by study steps (Exposed Set) | 51 |
| Template 4 | Summary of vital signs (Exposed Set) | 52 |
| Template 5 | Summary of study completion with reason for withdrawal (Exposed Set) | 53 |
| Template 6 | Summary of visit attendance (Exposed Set) | 53 |
| Template 7 | Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set) | 53 |
| Template 8 | Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set) | 53 |
| Template 9 | Summary of subject disposition from Randomized Set to Exposed set (Randomized set) | 54 |
| Template 10 | Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set) | 54 |
| Template 11 | Summary of subject disposition from Exposed Set to End of study (Exposed set) | 54 |
| Template 12 | Deviations from protocol for age and intervals between study visits (Exposed set) | 55 |
| Template 13 | Number of enrolled subjects by country | 55 |
| Template 14 | Number of enrolled subjects by age category | 55 |
| Template 15 | Minimum and maximum visit dates <analysis name="" set=""></analysis> | 55 |
| Template 16 | Exposure to study vaccines by vaccine (Exposed Set) | 56 |
| Template 17 | Number and percentage of subjects with <antibody concentration="" titer=""> equal to or above <cut-off unit=""> and <gmt cs=""> <analysis name="" set=""></analysis></gmt></cut-off></antibody> | 56 |
| Template 18 | <gmt cs=""> and their 95% CIs for <antibody concentrations="" titers=""> <analysis name="" set=""></analysis></antibody></gmt> | 57 |

| Template 19 | Geometric mean of the individual ratio of <antibody (units)="" concentrations="" titers=""> post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | . 57 |
|---|---|---|
| Template 20 | Distribution of <antibody concentrations="" titers=""> <per protocol="" set=""></per></antibody> | . 58 |
| Template 21 | Distribution of <antibody concentrations="" titers=""> fold increase post-vaccination compared to pre-vaccination <per protocol="" set=""></per></antibody> | . 58 |
| Template 22 | Reverse cumulative distribution curve of <antibody concentrations="" titers=""> in the <group label=""> group <per protocol="" set=""></per></group></antibody> | .59 |
| Template 23 | Kinetics of < antibody GMT/Cs> on subjects with results available at all timepoints up to <day 14="" 91,="" month=""> <per protocol="" set=""></per></day> | .60 |
| Template 24 | Individual results of <rsv a="" antibody="" neutralizing="" titer=""> at <time point=""> versus pre-vaccination in <group label=""> and Placebo_B groups <per protocol="" set=""></per></group></time></rsv> | .61 |
| Template 25 | Individual results of <rsv a="" antibody="" b="" neutralizing="" rsv="" titer="" versus=""> at <time point=""> , on pooled RSV groups <per protocol="" set=""></per></time></rsv> | . 62 |
| Template 26 | Geometric mean ratios of the fold increase (Pre to Post - vaccination) between RSVPreF3 IgG antibody concentrations and <rsv-a, rsv-b=""> neutralising antibody titers <per protocol="" set=""></per></rsv-a,> | .63 |
| Template 27 | Individual results of the fold increase (post over pre-vaccination) of RSVPreF3 IgG antibody concentrations versus <rsv a,="" b="" rsv=""> neutralizing antibody titers at <time point=""> in <group label=""> <per protocol="" set=""></per></group></time></rsv> | . 63 |
| Template 28 | Descriptive statistics of the frequency of RSVPreF3 specific-<br>CD4+ T cells expressing at least <2 markers among IL-2,<br>CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per<br>Protocol Set&gt;</per<br> | . 64 |
| Template 29 | Descriptive statistics of the frequency of RSVPreF3 specific-<br>CD4+ T cells expressing at least <2 markers among IL-2,<br>CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by<br>pre-vaccination category <per protocol="" set=""></per> | .64 |
| Template 30 | Boxplots with individual data of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> | . 65 |
| Template 31 | Frequency of RSVPreF3 specific CD4+ T-cells expressing any combination of markers among IL-2, CD40L, TNFa, IFNg in | |

| | <pre><group label=""> group at Day 31 and Day 91 (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per></group></pre> |
|---|---|
| Template 32 | Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <per protocol="" set="">66</per> |
| Template 33 | Descriptive statistics of the frequency of RSVPreF3 specific-<br>memory B-cells (per million of memory B cells, by Elispot) – Part<br>B <per protocol="" set=""></per> |
| Template 34 | Descriptive statistics of the fold increase (post over prevaccination) of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <per protocol="" set=""></per> |
| Template 35 | Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <per protocol="" set=""></per> |
| Template 36 | Comparisons of the 9 RSV formulations versus Placebo in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at one month post <dose (day="" 1="" 2="" 31),="" 91)="" dose=""> (ANCOVA model, Dunnett's test) – Part B <per protocol="" set=""></per></dose></rsv> |
| Template 37 | Comparisons of the mean responses post dose 2 (Day 91) versus post dose 1 (Day 31) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> on pooled groups according to adjuvant content (ANCOVA model) – Part B <per protocol="" set=""></per></rsv> |
| Template 38 | Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) - Part B <per protocol="" set=""></per></rsv> |
| Template 39 | Comparisons of the RSV groups (by antigen dose level) in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,=""> at Day 91 (ANCOVA model) – Part B <per protocol="" set=""></per></rsv> |
| Template 40 | Parameters of the ANCOVA model for the comparison between RSV groups in terms of <rsv 2="" a="" among="" antibody="" at="" cd4="" cd40l,="" cells="" expressing="" ifng="" il-2,="" least="" markers="" neutralizing="" rsvpref3-specific="" t="" titers,="" tnfa,="">- Part B <analysis name="" set=""></analysis></rsv> |
| Template 41 | Compliance in completing solicited adverse events information (Exposed Set) |

| Template 42 | Incidence and nature of <grade 3=""> symptoms (solicited and unsolicited) <with causal="" relationship="" to="" vaccination=""> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis name="" set=""></analysis></with></grade> | 73 |
|---|---|---|
| Template 43 | Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <analysis name="" set=""></analysis> | 74 |
| Template 44 | Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <analysis name="" set=""></analysis> | 74 |
| Template 45 | Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <cohort name=""></cohort> | 75 |
| Template 46 | Number of days with < local/general > solicited symptoms during < the 7-day (Days 1-7), the whole > post-vaccination period < analysis set name > | 77 |
| Template 47 | Incidence of solicited <local, general=""> adverse events reported during the 7-day (Days 1-7) post-vaccination period following each dose <exposed set=""></exposed></local,> | 78 |
| Template 48 | Percentage of subjects reporting the occurrence of <grade 3=""> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal="" relationship="" to="" vaccination=""> within the 30-day (Days 1-30) post-vaccination period <analysis name="" set=""></analysis></with></grade> | 78 |
| Template 49 | List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <exposed set=""></exposed> | <mark>7</mark> 9 |
| Template 50 | Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment <analysis name="" set=""></analysis> | <b>7</b> 9 |
| Template 51 | Listing of SAEs <analysis name="" set=""></analysis> | 79 |
| Template 52 | Listing of pregnancies reported during the study period in Part A <analysis name="" set=""></analysis> | 80 |
| Template 53 | Number and percentage of subjects taking concomitant medication during the <xx>-day (Days 1-<xx>) post-vaccination period by dose and overall <analysis name="" set=""></analysis></xx></xx> | 80 |
| Template 54 | Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <analysis name="" set=""></analysis> | 81 |

| Template 55 | Summary of hematology and biochemistry results by maximum grade at <visit (day="" 2="" 5="" 68)="" 8),="" visit=""> versus baseline (<day 1,="" 61="" day="">) <analysis name="" set=""></analysis></day></visit> | 81 |
|---|---|---|
| Template 56 | Summary of maximum hemoglobin change from baseline at <visit (day="" 2="" 5="" 68)="" 8),="" visit=""> (Exposed set)</visit> | 82 |
| Template 57 | Boxplot of <each biochemistry="" hematology="" parameter=""> (Exposed Set)</each> | 82 |
| Template 58 | Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis name="" set=""></analysis> | 83 |
| Template 59 | Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis name="" set=""></analysis> | 83 |
| Template 60 | Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis name="" set=""></analysis> | 84 |
| Template 61 | Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis name="" set=""></analysis> | 84 |
| Template 62 | Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <exposed set=""></exposed> | 85 |
| Template 63 | Descriptive statistics of the viral load of the RSV- confirmed RTI episodes, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <at home=""> <exposed set=""></exposed></at> | 85 |
| Template 64 | Number and percentage of subjects reporting co-infections with respiratory viruses, as measured by multiplex PCR on RSV A/B positive RTI samples collected <at assessment="" at="" home="" visit,=""> <exposed set=""></exposed></at> | 86 |
| Template 65 | Clinical signs and symptoms associated with RTI episodes (Exposed set) | 87 |
| Template 66 | Listing of RTI episodes reported during RTI surveillance in Part B (Exposed set) | 88 |
| Template 67 | GMTs and 95% CIs of RSV A Neutralizing antibody titer at baseline for subjects reporting RTI episodes (RSV RTI vs or non RSV RTI vs No RTI), by groups pooled according to the adjuvant content <exposed set=""></exposed> | 88 |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

#### LIST OF ABBREVIATIONS

AE Adverse event

ALT Alanine Aminotransferase

ANCOVA Analysis of Covariance

ANOVA Analysis of Variance

AST Aspartate Aminotransferase

BUN Blood Urea Nitrogen

CD40L Cluster of Differentiation 40 Ligand

CI Confidence Interval

CMI Cell-Mediated Immunity

CMV Cytomegalovirus

CSR Clinical Study Report

CTRS Clinical Trial Registry Summary

eCRF electronic Case Report Form

eDiary electronic Diary

ELU/ml ELISA unit per milliliter

ELISA Enzyme-linked immunosorbent assay

EoS End of Study

ES Exposed Set

FDA Food and Drug Administration

GMC Geometric mean antibody concentration

GMT Geometric mean antibody titer

GSK GlaxoSmithKline

ICS Intracellular Cytokine Staining

IDMC Independent Data Monitoring Committee

IFN-γ Interferon Gamma
IgG Immunoglobulin G

IL Interleukin

LL Lower Limit of the confidence interval

LLOQ Lower Limit Of Quantification

Mcg or μg Microgram

MedDRA Medical Dictionary for Regulatory Activities

PBMC Peripheral Blood Mononuclear Cells

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

PCR Polymerase Chain Reaction

PD Protocol Deviation

pIMD Potential Immune-Mediated Disease

PPS Per Protocol Set
PT Preferred Term

qRT-PCR Quantitative Reverse Transcription Polymerase Chain Reaction

RSV Respiratory Syncitial Virus RTI Respiratory Tract Infection

SAE Serious adverse event
SAP Statistical Analysis Plan

SBIR GSK Biological's Internet Randomization System

SD Standard Deviation

SR Study Report

TFL Tables Figures and ListingsTNF-α Tumor Necrosis Factor alpha

TOC Table of Content

UL Upper Limit of the confidence interval

WBC White Blood cells

#### 1. DOCUMENT HISTORY

| Date | Description | Protocol Version |
|-------------|---------------|--------------------|
| 14-JAN-2019 | Final version | Final: 11 SEP 2018 |

#### 2. STUDY DESIGN

Figure 1 Study design



BS S: Blood sample for safety (hematology/biochemistry)

BS H: Blood sample for humoral immune responses

BS C: Blood sample for cell-mediated immune responses (for CD4+/CD8+ and/or memory B-cell testing)

FU: Follow-up; PCR: Polymerase Chain Reaction

\* Visit 1 should take place no longer than 30 days after the Screening Visit. In case Visit 1 occurs more than 30 days after the Screening Visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection for safety laboratory assessment must be repeated (maximum one re-screening per subject is allowed). Only laboratory results from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF. Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. The subject can only be randomized once the investigator receives the results and confirms the eligibility criteria.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

- \*\* In Part A, a first IDMC evaluation of safety data up to Day 31 based on all subjects (~12 per group or at least 8 per group in case of slow recruitment) will be performed before proceeding with administration of Dose 2 in Part A and Dose 1 in Part B. A second IDMC evaluation will be performed based on safety data up to Day 68 for all subjects. Part B of the study can only be initiated upon favorable outcome of the first IDMC safety evaluation in Part A.
- \*\*\* In Part B, a third and fourth IDMC evaluation of safety data up to Day 8 and Day 68, respectively, for the first enrolled and vaccinated subjects (~10 per group or at least 8 per group in case of slow recruitment) will be performed. Additional IDMC evaluations will happen during the conduct of the study.
- <sup>†</sup> In case of RTI symptoms during the RSV seasons (approximately from October to March), the subject will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab at the site. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- <sup>£</sup> Analysis 1 will be performed on all data collected up to Day 91 for at least primary and secondary endpoints based on both study parts (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). Analysis 2 will be performed when all safety data up to Month 8 (Visit 7) are available. The analyses will be based on data as clean as possible.
- Experimental design: Phase I/II, observer-blind, randomized, controlled, multi-country study with 2 parts (i.e., Part A in young adults aged 18-40 years with 4 parallel groups and Part B in older adults aged 60-80 years with 10 parallel groups).
- **Primary Completion Date (PCD):** last visit of the vaccination phase in Part B (Visit 6 [Day 91]).
- End of Study (EoS): Last testing results released of samples collected up to Visit 8 in Part B (Month 14) (for assays related to primary and secondary endpoints only).
- **Treatment allocation:** Subjects will be randomized using a centralised randomization system on internet (SBIR) on Day 1.

In Part A, the aim is to enrol approximately 48 subjects (~12 per group) aged 18-40 years. The randomization algorithm will use a minimisation procedure accounting for center and gender.

In Part B, the aim is to enrol approximately 700 subjects (~70 per group) aged 60-69 years and approximately 300 subjects (~30 per group) aged 70-80 years. The randomization algorithm will use a minimisation procedure accounting for age, center and gender in each step.

#### Study groups:

For the investigational RSV vaccines in Part A and Step 1 in Part B, the RSVPreF3 high-dose formulation containing 120 µg RSVPreF3 will be used to prepare the vaccines for all dose groups (i.e., 30 µg, 60 µg and 120 µg dose groups). For Step 2 in Part B, the RSVPreF3 low-dose and mid-dose formulations (containing 30 µg and 60 µg RSVPreF3, respectively) will be used for the groups receiving 30 µg and 60 µg of RSVPreF3, respectively, and the RSVPreF3 high-dose formulation will be used for the 120 µg dose groups. As the reconstitution methods for the vaccines administered to subjects enrolled in Step 1 and 2 of Part B will be different, separate study groups have been identified (referred to as B1 and B2). Throughout this document, the combined groups for Steps 1 and 2 are mentioned when referring to the number of groups in Part B (10 groups).

- Control: placebo.
- Vaccination schedule: Two vaccine doses administered intramuscularly at Day 1 and Day 61.
- Blinding: observer-blind.

The vaccination phases of each study part (Epoch 002) will be observer-blind. A first statistical analysis will be performed on data available up to one month post-Dose 2 (Visit 6, Day 91). Given that summary safety results may unblind some specific subjects, the persistence phase of Part B (Epoch 003) will be considered as single-blind with subjects remaining blinded up to study end (Visit 8 [Month 14]). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

- RTI surveillance in Part B: Active and passive surveillance will only be carried out during RSV seasons (approximately from October to March) throughout the entire Part B of the study:
  - Active surveillance: study participants will be contacted by the investigator/study staff every 2 weeks to identify if they experience an RTI.
  - Passive surveillance: study participants are instructed to contact the investigator/study staff as soon as they experience an RTI.

At the beginning of RSV seasons, study participants will be reminded of the start of the RTI surveillance.

#### • Sampling schedule:

#### In Part A:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the electronic Case Report Form (eCRF). The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for cytomegalovirus (CMV) status determination will be drawn from all subjects.
- Blood samples for safety assessment (hematology/biochemistry) will be drawn from all subjects on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).
- Blood samples for humoral immunogenicity and cell-mediated immunity
   (CMI) testing will be drawn from all subjects at Days 1, 31, 61 and 91 (Visits 1, 3, 4 and 6).

#### In Part B:

- At Screening (Pre-Day 1), a blood sample for eligibility assessment will be drawn from all subjects. In case Visit 1 occurs more than 30 days after the Screening visit, a re-screening visit should be scheduled before Visit 1 during which blood sample collection must be repeated (maximum one re-screening per subject is allowed). Medical history, physical examination and review of inclusion/exclusion criteria must be repeated if a re-screening visit occurs. Only data from the re-screening visit, if it occurs, will be taken into consideration and recorded in the eCRF. The subject can however only be randomized once the investigator receives the safety assessment results and confirms the eligibility criteria.
- At Day 1 (Visit 1), a blood sample for CMV status determination will be drawn from all subjects.
- **Blood samples for safety assessment** (hematology/biochemistry) will be drawn from all subjects and on Days 1, 8, 61 and 68 (Visits 1, 2, 4 and 5).
- Blood samples for humoral immunogenicity and CMI testing will be drawn from all subjects at Days 1, 31, 61, 91, Month 8 and Month 14 (Visits 1, 3, 4, 6, 7 and 8).
- Nasal/throat swabs: In case of RTI symptoms during the RSV season (approximately from October to March), the study participants will be asked to collect a nasal swab at home and contact the investigator/study staff to schedule an assessment visit for collection of an additional nasal/throat swab by qualified staff from the study team. The assessment visit should take place as soon as possible after the start of symptoms (ideally within 48 hours, but no later than 7 days).
- **Type of study:** self-contained.
- **Data collection:** eCRF. Solicited symptoms will be collected using an electronic subject Diary (eDiary). Unsolicited symptoms will be collected using a paper subject Diary.
- **Safety monitoring:** The study will be conducted in 2 parts with oversight by an IDMC. The investigator is not permitted to start vaccinating the subjects in the next step in each part until receipt of the favorable outcome of the respective safety evaluations by the IDMC.
  - Part A: Approximately 48 young adults aged 18-40 years will be enrolled and vaccinated with the first dose. If the IDMC evaluation on data up to 30 days post Dose 1 is favorable, the Part A study participants will be vaccinated with the second dose and Part B of the study will be initiated.
  - Part B: This part will be conducted in a 2-step staggered design to ensure maximum safety of the participating subjects. In Step 1, approximately 100 subjects will be enrolled and vaccinated. Safety evaluations based on unblinded data from those first 100 subjects will be performed by the IDMC to allow the start of Step 2. In Step 2, the remaining study participants (N≅900) will be recruited and vaccinated.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

In total, 6 IDMC meetings for safety evaluation are foreseen in the vaccination phase of the study (Epoch 002), i.e., 2 meetings in Part A and 4 meetings in Part B.

During the persistence phase of Part B (Epoch 003), 2 IDMC meetings will be planned with an interval of approximately 6 months.

If any safety concern is identified by the investigator or the sponsor, *ad-hoc* safety evaluations by the IDMC may be performed.

Analysis planned for IDMC evaluations are described in a separate document (SAP for IDMC).

#### • Group description for analysis:

For analysis based on subjects in Part A and Part B Step 1 (B1), the group labels listed in table below will be used in the TFLs.

For final analysis based on subjects from Part B Steps 1 and 2, the groups will be pooled (B1 and B2) and the Pooled group labels will be used in the TFLs.

Table 1 Groups description

| Group label in tables | Group definition for footnote | Pooled Group label in tables | Pooled Group definition for footnote |
|---|---|---|---|
| 30-PLAIN_A | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part A | NA | |
| 60-PLAIN_A | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part A | NA | |
| 120-<br>PLAIN_A | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part A | NA | |
| Placebo_A | subjects receiving Placebo in Part A | NA | |
| 30-<br>PLAIN_B1 | subjects receiving unadjuvanted<br>30 mcg RSVPreF3 in Part B Step<br>1 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |
| 30-<br>PLAIN_B2 | subjects receiving unadjuvanted<br>30 mcg RSVPreF3 in Part B Step<br>2 | 30-PLAIN_B | subjects receiving unadjuvanted 30 mcg RSVPreF3 in Part B |
| 60-<br>PLAIN_B1 | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B Step<br>1 | 60-PLAIN_B | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part B |
| 60-<br>PLAIN_B2 | subjects receiving unadjuvanted<br>60 mcg RSVPreF3 in Part B Step<br>2 | 60-PLAIN_B | subjects receiving unadjuvanted 60 mcg RSVPreF3 in Part B |
| 120-<br>PLAIN_B1 | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B Step<br>1 | 120-PLAIN_B | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part B |
| 120-<br>PLAIN_B2 | subjects receiving unadjuvanted<br>120 mcg RSVPreF3 in Part B Step<br>2 | 120-PLAIN_B | subjects receiving unadjuvanted 120 mcg RSVPreF3 in Part B |
| 30-<br>AS01E_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 30-AS01E_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |

| Group label in tables | Group definition for footnote | Pooled Group label in tables | Pooled Group definition for footnote |
|---|---|---|---|
| 30-<br>AS01E_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 30-AS01E_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |
| 60-<br>AS01E_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 60-AS01E_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |
| 60-<br>AS01E_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 60-AS01E_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |
| 120-<br>AS01E_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 1 | 120-AS01E_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |
| 120-<br>AS01E_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E<br>in Part B Step 2 | 120-AS01E_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01E in<br>Part B |
| 30-<br>AS01B_B1 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 30-AS01B_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| 30-<br>AS01B_B2 | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 30-AS01B_B | subjects receiving 30 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| 60-<br>AS01B_B1 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 60-AS01B_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| 60-<br>AS01B_B2 | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 60-AS01B_B | subjects receiving 60 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| 120-<br>AS01B_B1 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 1 | 120-AS01B_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| 120-<br>AS01B_B2 | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B<br>in Part B Step 2 | 120-AS01B_B | subjects receiving 120 mcg<br>RSVPreF3 adjuvanted with AS01B in<br>Part B |
| Placebo_B1 | subjects receiving Placebo in Part<br>B Step 1 | Placebo_B | subjects receiving Placebo in Part B |
| Placebo_B2 | subjects receiving Placebo in Part<br>B Step 2 | Placebo_B | subjects receiving Placebo in Part B |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

For some of the comparison analyses in Part B, the RSV vaccine groups will be pooled according to their adjuvant content and the following group names will be used in the TFLs:

| Pooled Group label in tables | Pooled Group definition for footnote | Groups to be pooled |
|---|---|---|
| PLAIN_B | subjects receiving unadjuvanted RSVPreF3 in Part B (30, 60 or 120 μg) | 30_PLAIN_B1, 30_PLAIN_B2,<br>60_PLAIN_B1, 60_PLAIN_B2,<br>120_PLAIN_B1, 120_PLAIN_B2 |
| AS01E_B | subjects receiving RSVPreF3 adjuvanted with AS01E in Part B (30, 60 or 120 μg) | 30_AS01E_B1, 30_ AS01E_B2,<br>60_ AS01E_B1, 60_ AS01E_B2,<br>120_ AS01E_B1, 120_ AS01E<br>_B2 |
| AS01B_B | subjects receiving RSVPreF3 adjuvanted with AS01B in Part B (30, 60 or 120 μg) | 30_AS01B_B1, 30_ AS01B_B2,<br>60_ AS01B_B1, 60_ AS01B_B2,<br>120_ AS01B_B1, 120_ AS01B<br>_B2 |

For the analysis by age category, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | 60-69Y | 60-69 years old subjects |
| 2 | 70-80Y | 70-80 years old subjects |

For the analysis by CMV status before vaccination, the following sub-group names will be used in the TFLs:

| Sub-group order in tables | Sub-group label in tables | Sub-group definition for footnote |
|---|---|---|
| 1 | CMV+ | Subjects CMV positive before vaccination |
| 2 | CMV- | Subjects CMV negative before vaccination |

#### 3. OBJECTIVES/ENDPOINTS

#### 3.1. Objectives

#### 3.1.1. Primary objective

#### For Part A and Part B:

• To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccine administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

#### 3.1.2. Secondary objectives

#### For Part A and Part B:

- To characterize the humoral immune responses (including dose-response) in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).
- To characterize the cell-mediated immune responses in relation to the investigational RSV vaccine formulations administered IM according to a 0, 2 month schedule, up to one month after the last dose (Day 91, Visit 6).

#### For Part B:

- To evaluate the safety and reactogenicity of 2 doses of the investigational RSV vaccines administered IM according to a 0, 2 month schedule, up to the end of follow-up (Month 14, Visit 8).
- To evaluate the occurrence of RSV-associated respiratory tract infections (RTI) during the RSV season in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.

#### 3.1.3. Tertiary objectives

#### For Part A and Part B:

To further characterize the cell-mediated immune responses to investigational RSV vaccine formulations.

#### For Part B:

- To further characterize immune responses to investigational RSV vaccine formulations.
- To characterize persistence of immune responses to the investigational RSV vaccine formulations at Month 8 (Visit 7) and Month 14 (Visit 8).
- To further evaluate the occurrence of RSV-associated RTI (including co-infections with other respiratory viruses) during the RSV seasons in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI.

• To evaluate the occurrence of RSV-associated RTI during the RSV season using self-collected nasal swabs.

#### 3.2. Endpoints

#### 3.2.1. Primary endpoints

#### For Part A and Part B:

- Occurrence of AEs from first vaccination up to 30 days after the second vaccination (Day 91):
  - Occurrence of each solicited local and general AE during a 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) after each vaccination.
  - Occurrence of any unsolicited AE during a 30-day follow up period (i.e., on the day of vaccination and 29 subsequent days) after each vaccination.
  - Occurrence of any hematological (erythrocytes, WBC and differential count, platelets count and hemoglobin level) and biochemical (ALT, AST, creatinine, BUN and uric acid) laboratory abnormalities at Days 1, 8, 61 and 68.
  - Occurrence of all Grade 3 non-serious AEs (solicited and unsolicited) during the 30-day follow-up period after each vaccination.
  - Occurrence of SAEs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

#### For Part B only:

 Occurrence of pIMDs from Dose 1 up to 30 days after the second vaccine dose (Day 91).

#### 3.2.2. Secondary endpoints

#### For Part A and Part B:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), on the day of second vaccination (Day 61) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.
- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro.

#### For Part B only:

- Occurrence of RSV-associated RTI (as measured by qRT-PCR in nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons, up to the end of follow-up.
- Occurrence of SAEs from Dose 1 up to the end of follow-up.
- Occurrence of pIMDs from Dose 1 up to the end of follow-up.

#### 3.2.3. Tertiary endpoints

#### For Part A and Part B:

- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31), pre-Dose 2 (Day 61) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro.

#### For Part B only:

- Humoral immune response with respect to components of the investigational vaccine at pre-vaccination (Day 1) and 30 days post-Dose 2 (Day 91):
  - Neutralizing antibody titers against RSV serotype B in all subjects.
  - RSVPreF3 site 0 specific antibody concentrations in a subset of subjects who received the selected vaccine formulation or placebo.
- Cell-mediated immune response profile with respect to components of the investigational vaccine at pre-vaccination (Day 1), 30 days post-Dose 1 (Day 31) and 30 days post-Dose 2 (Day 91):
  - Frequency of RSVPreF3-specific memory B-cells in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Persistence of the humoral immune response with respect to components of the investigational vaccine at Months 8 and 14:
  - Neutralizing antibody titers against RSV serotype A.
  - RSVPreF3-specific IgG antibody concentrations.
- Persistence of the cell-mediated immune response profile with respect to components of the investigational vaccine:
  - Frequency of RSVPreF3-specific CD4+ and/or CD8+ T-cells identified as expressing one or any combination of immune marker(s) in vitro, in all subjects (Month 8) and in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo (Month 14).
- Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ in vitro, in all subjects (Month 8) and in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo (Month 14).
- Frequency of RSVPreF3-specific memory B-cells at Month 14 in a subset of subjects who received the selected level of antigen dose (3 RSV vaccine formulations) or placebo.
- Any further exploratory immunology to detect RSV-related immune responses, such as but not limited to:
  - Antibodies against specific protein F epitopes.
  - Potential new immunological markers for protection.
  - Cross-reactive neutralizing antibody titters against hMPV
- Occurrence of RSV-associated RTI, including co-infections with other respiratory viruses (as measured by multiplex PCR in self-collected nasal swab samples and nasal/throat swab samples collected during the assessment visit for potential RSV-RTI) during the RSV seasons.
- Occurrence of RSV-associated RTI as measured by qRT-PCR in self-collected nasal swab samples during the RSV seasons, up to the end of follow-up.

## 4. ANALYSIS SETS

#### 4.1. Definition

# 4.1.1. Exposed Set

The Exposed Set (ES) will include all subjects with study vaccine administration documented.

A safety analysis based on the ES will include all vaccinated subjects.

An immunogenicity analysis based on ES will include all vaccinated subjects for whom immunogenicity data are available.

The ES analysis will be performed per treatment actually administered at Dose 1.

# 4.1.2. Per-Protocol Set for analysis of immunogenicity

The Per-Protocol set (PPS) for analysis of immunogenicity will be defined by time point (and this to include all eligible subjects' data up to the time of important protocol deviations). The PPS will include all evaluable subjects in the ES:

- Meeting all eligibility criteria.
- For whom the administration route of the vaccine was as according to protocol.

- For whom the study vaccine was administered as per protocol.
- Who did not receive a concomitant medication/ product leading to exclusion from a PP analysis, as described in Section 6.6.2 of the protocol, up to the considered time point.
- Who did not present with a medical condition leading to exclusion from a PP analysis, as described in Section 6.7 of the protocol, up to the considered time point.
- Who complied with the vaccination schedule, as specified in the protocol.
- Who complied with the timings of the post-vaccination blood sampling for immune response evaluation, as specified in the protocol.
- For whom post-vaccination immunogenicity results are available for at least one assay component at the corresponding time points.

# 4.2. Criteria for eliminating data from Analysis Sets

Elimination codes are used to identify subjects to be eliminated from analysis. Detail is provided below for each set.

# 4.2.1. Elimination from Exposed Set (ES)

Code 1030 (Study vaccine not administered at all) and code 900 (invalid informed consent or fraudulent data) will be used for identifying subjects eliminated from ES.

# 4.2.2. Elimination from Per-protocol analysis Set (PPS)

# 4.2.2.1. Excluded subjects

A subject will be excluded from the PPS analysis under the following conditions.

For codes 1040, 1070, 1080, 1090, 2040, 2060, 2080: subjects will be eliminated from a specific visit (at which the condition is met) onwards.

For codes 2090, 2100, 2120: subjects will be eliminated at the specific visit at which the condition is met.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 900 | Invalid informed consent or fraudulent data | All | All |
| 1030 | Study vaccine not administered at all | All | All |
| 1040 | Administration of concomitant vaccine(s) forbidden in the protocol: Any investigational or non-registered vaccine other than the study vaccine used during the study period A vaccine not foreseen by the study protocol administered during the period starting 30 days before the first dose and ending 30 days after the last vaccine dose, except for inactivated and subunit influenza vaccines which can be administered up to 14 days before or from 30 days after each vaccination. | All | Immunology |
| 1050 | Randomisation failure | All | Immunology |
| 1060 | Randomisation code was broken | All | Immunology |
| 1070 | Vaccination not according to protocol: Incomplete vaccination course Subject was vaccinated with the correct vaccine but containing a lower volume Wrong replacement or study vaccine administered (not compatible with the vaccine regimen associated to the treatment number) Route of the study vaccine is not intramuscular Wrong reconstitution of administered vaccine | All | Immunology |
| 1080 | Vaccine temperature deviation vaccine administered despite a Good Manufacturing Practices (GMP) no-go temperature deviation | Vaccination visits 1 and 4 | Immunology |
| 1090 | Expired vaccine administered | Vaccination visits 1 and 4 | Immunology |
| 2010 | Protocol violation (inclusion/exclusion criteria) | All | Immunology |
| 2040 | Administration of any medication forbidden by the protocol Any investigational or non-registered medication used during the study period Immunosuppressants or other immune-modifying drugs administered chronically (i.e., more than 14 consecutive days in total) during the study period Long-acting immune-modifying drugs administered at any time during the study period Immunoglobulins and/or any blood products administered during the study period | All | Immunology |
| 2060 | Intercurrent medical condition Subjects may be eliminated from the PPS if, during the study, they incur a condition that has the capability of altering their immune response or are confirmed to have an alteration of their initial immune status (other than RSV infection). | All | Immunology |
| 2080 | Subjects did not comply with vaccination schedule: Part A: number of days between dose 1 and dose 2 is outside [55-80 days] Part B: number of days between dose 1 and dose 2 is outside [55-75 days] | Visit 4 | Immunology |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

| Code | Condition under which the code is used | Visit<br>(timepoints)<br>where the<br>code is<br>applicable | Applicable for analysis set |
|---|---|---|---|
| 2090 | Subjects did not comply with blood sample schedule at a specific visit: Number of days between dose 1 and visit 3 blood sample is outside [30-37 days] Number of days between dose 2 and visit 6 blood sample is outside [30-37 days] Part B only: Number of days between dose 2 and visit 7 blood sample is outside [170-190 days] Number of days between dose 2 and visit 8 blood sample is outside [350-395 days] | Visits 3, 6, 7 and 8 | Immunology |
| 2100 | Immunological results not available post-vaccination No immunological result at visit x for all 3 following tests: RSV A Neutralising antibody titer, RSVPreF3- specific IgG antibody concentration and RSVPreF3- specific CD4+ T cells frequency | Visits 3, 4, 6, 7, 8 | Immunology |
| 2120 | Obvious incoherence or abnormality or error in data Unreliable released data as a result of confirmed sample mismatch or confirmed inappropriate sample handling at lab | Visits 1, 3, 4, 6, 7, 8 | Immunology |

# 5. STATISTICAL ANALYSES

Note that standard data derivation rules and stat methods are described in "business rules document" and will not be repeated below. The study specific data derivation rules and stat methods will be described in section 9.

# 5.1. Demography

# 5.1.1. Analysis of demographics/baseline characteristics planned in the protocol

Demographic characteristics (age at first vaccination in years, gender, race and ethnicity) will be summarized by group using descriptive statistics:

- Frequency tables will be generated for categorical variable such as race.
- Mean, median, standard error and range will be provided for continuous data such as age.

The distribution of subjects will be tabulated as a whole and per group and for each age category (60-69 years and 70-80 years in Part B only).

Withdrawal status will be summarized by group using descriptive statistics:

- The number of subjects enrolled into the study as well as the number of subjects excluded from PP analyses will be tabulated.
- The numbers of withdrawn subjects will be tabulated according to the reason for withdrawal

## 5.1.2. Additional considerations

The analysis of demographic characteristics by group will be performed on the ES and on the PPS.

Demography and baseline characteristics will also be summarized by country.

Vital signs (heart rate, respiratory rate, systolic/diastolic blood pressure, pulse oximetry) reported at visit 1 (Part A and Part B) will be summarized by group using descriptive statistics.

# 5.2. Exposure

# 5.2.1. Analysis of exposure planned in the protocol

NA

#### 5.2.2. Additional considerations

The number of doses of study vaccines administered will be tabulated by group and by vaccine.

# 5.3. Immunogenicity

# 5.3.1. Analysis of immunogenicity planned in the protocol

The primary analysis will be performed on the PPS for immunogenicity and, if in any study group the percentage of vaccinated subjects with serological results excluded from the PPS for analysis of immunogenicity is at least 10%, a second analysis will be performed on the ES.

## 5.3.1.1. Within groups evaluation - humoral immune response

For each group, at each time point that blood samples are collected for humoral immune response and for each assay (unless otherwise specified):

## In Part A and Part B:

- Percentage of subjects above pre-defined threshold and their exact 95% CI will be tabulated.
- GMCs/GMTs and their 95% CI will be tabulated and represented graphically.
- Geometric mean of ratios of antibody titer/concentrations at each post-vaccination time point over pre-vaccination (Day 1) will be tabulated with 95% CI.
- Antibody titer/concentration will be displayed using reverse cumulative curves.
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will be computed and tabulated using descriptive statistics.

## In Part B only:

- The distributions of antibody titers/concentrations will be tabulated.
- Individual post-vaccination results (at Days 31 and 91) versus pre-vaccination results (Day 1) will be plotted using scatter plots. Results of the placebo group will be used as a reference
- Distribution of the fold increase of the antibody titers/concentrations (post- over prevaccination titers) will be tabulated.
- The kinetics of GMT/GMCs will be plotted as a function of time for subjects with results available at all time points.

The immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

The humoral immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

## 5.3.1.2. Within groups evaluation - Cell-mediated immune response

The following parameters will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI:

## In Part A and Part B:

- Frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, upon in vitro stimulation and background substracted, measured by ICS using PBMCs.
- Frequency of CD4+ and/or CD8+ T-cells expressing **any combination of immune marker(s)** among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs (see details in section 5.3.2.2).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

• Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.

## In Part B only:

- Frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.
- Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

This will be displayed overall and by pre-vaccination category: <Q1, Q1-Q3, >Q3, where Q1/Q3 are respectively the 25<sup>th</sup> and the 75<sup>th</sup> percentiles of the results at pre-vaccination computed on pooled groups.

In addition, vaccine response in terms of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , will be explored and summarised by group.

The descriptive immunogenicity analysis will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years) in Part B only.

The cell-mediated immune response by CMV status before vaccination might be explored in Parts A and B. This will be done if at least 10% of the subjects are included in each CMV status category (CMV positive and CMV negative).

## 5.3.1.3. Between groups evaluation (Part B only)

Statistical analyses will be performed to compare the 9 RSV investigational vaccine formulations in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

The between-groups analysis will be performed using an ANCOVA model, in several steps as follows:

- 1. The 9 RSV formulations will be first compared to the Placebo in order to identify groups whose means are significantly higher from the mean of the Placebo group, in terms of RSV-A neutralizing antibody titers and RSVPreF3-specific CD4+ T-cells at Day 31 and Day 91 (One-sided alpha=2.5%, Dunnett's adjustment test for multiplicity).
- 2. The effect of the second vaccination will be evaluated by comparing the means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31), of the groups pooled according to their adjuvant content (AS01<sub>B</sub>, AS01<sub>E</sub> and Plain), in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibody titers (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose).

Based on the results of this test, the next comparisons will be performed either at Day 91 or at Day 31.

- 3. Appropriate contrasts will be implemented to compare the RSV formulations as follows:
  - To demonstrate the adjuvant effect (on pooled groups according to their adjuvant content: AS01B, AS01E, Plain), by testing sequentially AS01B and AS01E versus Plain (One-sided alpha=2.5% for each superiority test: Adjuvant >Plain) in terms of RSVPreF3-specific CD4+ T-cells and RSV-A neutralizing antibodies and, if applicable, by comparing AS01B vs AS01E.
  - To demonstrate linearity of increase in immune response when increasing the antigen dose in each adjuvanted group in terms of RSV-A neutralizing antibody and/or RSVPreF3-specific CD4+ T-cells.
  - Further ANCOVA t-tests would demonstrate superiority of 120 μg or 60 μg, should a quadratic effect be demonstrated.
  - Similar exploratory comparisons might also be performed on the RSVPreF3
     ELISA antibody concentrations if deemed necessary.

## 5.3.2. Additional considerations

## 5.3.2.1. Within groups – humoral immune response

- Correlations between assays of the humoral response will be investigated using scatter plots generated on pooled RSV groups:
  - RSVPreF3-specific IgG versus RSV A neutralizing antibody titer at each timepoint,
  - RSV A versus RSV B neutralizing antibody titer at Pre-vaccination and Day 91
  - RSVPreF3-specific IgG versus RSV-B neutralizing antibody titer at Prevaccination and Day 91

The same analysis will be performed on the fold increase post over pre-vaccination.

• The fold increase (post over pre-vaccination) of the RSVPreF3 IgG antibody concentrations versus the fold increase (post over pre-vaccination) of RSV-A and RSV B neutralizing antibody titers will also be displayed graphically by group using scatter plots.

## 5.3.2.2. Within groups – Cell-mediated immune response

**Descriptive statistics** of the cell-mediated immune response will be tabulated and displayed graphically using boxplots (min, Q1, median, Q3, max), by group and timepoint.

The RSVPreF3-specific CD4+/CD8+ T cell frequencies will be obtained by subtracting the background value to the antigen-induced value, and by setting to 1 all values less than or equal to zero for geomean calculation and graphical representation. Frequencies will be expressed as the number of cells per million of CD4+/CD8+ T cells.

More specifically, the frequencies of RSVPreF3-specific CD4+ T cells expressing at least 2 cytokines [ $Freq^{2+}$ ] will be computed as follows:

$$Freq_{Background}^{2^{+}} = \frac{n_{background}^{2^{+}}}{N_{Background}^{CD4}}$$
 and  $Freq_{Induction}^{2^{+}} = \frac{n_{Induction}^{2^{+}}}{N_{Induction}^{CD4}}$ ,

And

$$Freq_{Specific}^{2+} = Freq_{Induction}^{2+} - Freq_{Background}^{2+}$$

where

 $n_{Background}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with medium only (background)

 $n_{Induction}^{2+}$  = number of CD4+ T cells expressing at least 2 cytokines after stimulation with a pool of peptides covering RSVPreF3 (induction)

 $N_{Back/Ind}^{CD4}$  = Total number of CD4 T cells involved in the assay (background or induction)

Same computations will be done for all CMI responses that will be analysed, i.e.:

- Frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ, as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least 2 markers including at least 1 cytokine\* among CD40L, 41BB, IL-2, TNF-α, IFN-γ, IL-13, and IL-17, as measured by ICS using PBMCs.
  - \* cytokines are IL-2, TNF-\alpha, IFN-\gamma, IL-13, and IL-17
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IFN-γ (Th1-like response), as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/CD8+ T-cells expressing at least IL-13 (Th2-like response), as measured by ICS using PBMCs.
- Frequency of RSVPreF3-specific CD4+/ CD8+ T-cells expressing at least IL-17 (Th17-like response), as measured by ICS using PBMCs.
- Co-expression profile: Frequency of RSVPreF3-specific CD4+ T-cells expressing any combination of marker(s) among CD40L, IL-2, TNF-α, IFN-γ, as measured by ICS using PBMCs, at Day 31 and Day 91 (15 combinations).

**Vaccine response** in terms of RSVPreF3-specific CD4+ T cells frequencies expressing at least 2 markers among CD40L, IL-2, TNF-α, IFN-γ will be explored as follows:

• Distribution of the fold increase: the percentage of subjects with at least a 2-fold, 4-fold, 6-fold, 8-fold, 10-fold increase post-vaccination as compared to pre-vaccination (Post over Pre) will be tabulated by timepoint and by group.

For the computation of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing **at least 2 marker(s)** among IL-2, CD40L, TNF- $\alpha$ , IFN- $\gamma$ , the results **below the LLOQ** of the assay will be replaced by the value of the LLOQ.

# 5.3.2.3. Between groups analysis

Statistical comparisons will be performed on the logarithm base 10 transformed results, in terms of RSV-A neutralizing antibody titers and frequency of RSVPreF3-specific CD4+ T-cells expressing at least 2 markers among IL-2, CD40L, TNF-α, IFN-γ.

# a. Comparisons versus Placebo:

The 9 RSV formulations will be compared to the Placebo (control group) at Day 31 and Day 91 using an ANCOVA model with the Dunnett's adjustment method for multiplicity. The model will include the treatment group and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. Geometric mean ratios between groups and associated Dunnett's adjusted 95% CIs of the ratios will be tabulated.

The Dunnett's test is specifically designed for situations where all groups are to be compared against one "Reference" group. It is commonly used after ANCOVA has rejected the hypothesis of equality of the means of the distributions.

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test (where=(visit=D91));
CLASS treatmnt Adj agecat;
MODEL log(titer)=treatmnt baseline agecat / ddfm=KR DDFM=KR
outpm=pred_model cl;
REPEATED / group=Adj ; /* test homogeneity of variances and consider
different variance by adjuvant content if appropriate */
LSMEANS treatmnt / ALPHA=0.05 Adjust=Dunnett pdiff=control ("Placebo")
CL;
RUN;
```

# b. Comparisons between RSV groups:

The difference between RSV groups will be evaluated using an ANCOVA model including the adjuvant content (AS01B, AS01E, Plain), the antigen dose (30, 60, 120  $\mu$ g), the visit (Day 31, Day 91) and the age category (age at Dose 1: 60-69 or 70-80 years) as fixed effects, and the pre-vaccination log10-transformed titer as covariate. The adjuvant by antigen interaction will also be tested, and included in the model if significant at 10% (p-value <10%).

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Based on this global model, appropriate contrasts will be used to perform the following comparisons:

1. Effect of the second vaccination:

The means one month post-Dose 2 (Day 91) and one month post-Dose 1 (Day 31) will be compared within each pooled group according to adjuvant content (AS01B, AS01E and Plain) (One-sided alpha=2.5% for each superiority test: 2 doses> 1 dose). Geometric mean ratios and associated 95% CIs will be tabulated.

1. Adjuvant effect:

The adjuvant effect will be tested sequentially as follow (One-sided alpha=2.5% for each superiority test):

- 1. AS01B versus Plain
- 2. AS01E versus Plain
- 3. AS01B versus AS01E.

Geometric mean ratios and their 95% CIs will be computed for each comparison.

The same comparisons will also be performed by age category.

1. Antigen dose-response: test linear and quadratic effect of the antigen dose. Depending on significance of those 2 effects, ANCOVA t-tests might be done to demonstrate superiority of 120 μg or 60 μg.

Geometric mean ratios and their 95% CIs will be computed for each pairwise comparison within each adjuvant content family (120  $\mu$ g vs 60  $\mu$ g, 120  $\mu$ g vs 30  $\mu$ g, 60  $\mu$ g vs 30  $\mu$ g for Plain, AS01E and AS01B groups).

Here is an example of SAS code that will be used:

```
PROC MIXED DATA=test;
  class Adj(1B, 1E, PL) Ag(30, 60, 120) visit(PD1, PD2) subject agecat;
  model log(titer) = Adj Ag visit Adj*Ag Adj*visit Ag*visit Adj*Ag*visit
baseline baseline*visit agecat / DDFM=KR S outpm=pred_model cl;
  REPEATED visit / SUBJECT=subject type=unr group=Adj;
  /* test homogeneity of variances and consider different variance by
  adjuvant content if appropriate */
  LSMEANS Adj*visit /E slice=visit CL PDIFF ALPHA=0.05; /*option E to see
  coefficients assigned to each effect */
  LSMEANS Adj*visit /E slice=Adj CL PDIFF ALPHA=0.05;
  LSMEANS Adj*Ag*visit / slice=visit CL PDIFF ALPHA=0.05;
  /* contrasts to be added for each comparison of interest */
  QUIT;
```

The inferential analysis on the RSVPreF3-specific CD4+ T cells will be performed on the log-transformation frequency of the CD4+ T cells expressing at least 2 markers (background or induction) computed by adding an offset of 0.5 cells to the number of activated CD4+ T cells (Delta method, see below). These transformations are deemed appropriate for further inferential analyses provided the incidence of activated CD4+ T-cells is below 4%.

Considering:

$$\begin{split} X_{ijk} &= \log\!\!\left(\frac{n_{background}^{2+} + 0.5}{N_{Background}^{CD4}}\right) \text{, the log background frequency, and} \\ Y_{ijk} &= \log\!\!\left(\frac{n_{Induction}^{2+} + 0.5}{N_{Induction}^{CD4}}\right) \text{, the log induction frequency} \end{split}$$

The following model can be used to analyse the log-transformed ratio between induction and background frequencies, and provide estimates of the RSVPreF3-specific frequency (Delta Method- Inference on Induction/background data):

$$Y_{ijk} = \mu_{jk} + \alpha_j . y_{i0k} + \beta x_{ijk} + \varepsilon_{ijk}$$
, with 
$$(\overline{Y_{jk} - x_{jk}})\Big|_{\overline{y}_0, \overline{x}} = \mu_{jk} + \alpha_j . \overline{y}_0 + \beta . \overline{x}$$
, LS means conditional to  $\overline{y}_0$  and  $\overline{x}$ 

where:

i, j, k=subject i, visit j, group k;  $\overline{y}_0$ = mean log induction frequency at pre-vaccination,

 $\bar{x}$ = mean log background after vaccination.

Note: This analysis is assuming that the background is the same for all groups and all timepoints. This assumption will be checked during the analysis.

Geometric means (GMs) of post-vaccination RSVPreF3-specific CD4+ T cell frequency and 95% CIs, will be calculated conditionally to the means of the pre-vaccination log-transformed CD4+ T cell frequency following induction with RSVPreF3 and the post-vaccination log-transformed CD4+ T cell frequency under background conditions.

The test and the 95% CIs for treatment comparisons will be calculated according to the delta method on the log-transformed ratio of RSVPref3-specific frequency relative to the background frequency estimates:

$$\hat{Z}_{jk} = 10^{\wedge} (\hat{Y}_{jk} - \overline{x}) - 1 = \frac{10^{\wedge} (\hat{Y}_{jk}) - 10^{\wedge} (\overline{x})}{10^{\wedge} (\overline{x})}$$
, and

$$Log(\hat{W}_{jk}) = Log\left(\frac{\hat{Z}_{jk_2}}{\hat{Z}_{jk_1}}\right) = Log\left(\frac{10^{\wedge}(\hat{Y}_{jk_2}) - 10^{\wedge}(\overline{x})}{10^{\wedge}(\hat{Y}_{jk_1}) - 10^{\wedge}(\overline{x})}\right), \text{ where}$$

 $\hat{Z}_{jk}$ = mean increase from background to induction frequency relative to background frequency at visit j for treatment k, and

 $\hat{W}_{jk}$  = vaccine effect on the antigen specific frequency following adjustment for background frequency.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

# Algorithm for calculations of Confidence Intervals of antigen-specific CMI response using the Delta-Method

Analysis results transformations:

- 1. The LSM and CI are back-transformed on the original scale to provide Geometric Mean Ratios of the induction frequency over background frequency.(Induction\_freq GM / Background freq GM)
- 2. Unity is removed from the Geometric Mean Ratios & CI ((Induction\_freq GM Background\_freq GM) / Background\_freq GM)
- 3. The result in 2 is multiplied by the geometric mean of background frequency used to calculate the LSM to provide the geometric means for the antigen-specific frequency.(Induction freq GM Background freq GM)
- 4. The log-transformed of the result in 2 is calculated and the difference between test group and control group is calculated.Log(Induction\_freq GM\_test Background\_freq GM) Log(Induction\_freq GM\_control Background\_freq GM)
- 5. The confidence interval of the result in 4 is calculated through the delta-method, using student-t distribution and the number of degree of freedom provided by MIXED for the difference in LSM.
- 6. The result in 4 is back-transformed to original scale to provide the fold-increase in the frequency of antigen-specific frequency.(Induction\_freq GM\_t Background freq GM) / (Induction freq GM c Background freq GM)

# 5.4. Analysis of safety and reactogenicity

# 5.4.1. Analysis of safety and reactogenicity planned in the protocol

The percentage of subjects with at least one local AE (solicited and unsolicited), with at least one general AE (solicited and unsolicited) and with any AE during the 7-day or 30-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, for Grade 3 AEs considered related to vaccination and for Grade 3 non-serious AEs.

The percentage of subjects with any AE (solicited and unsolicited) resulting in a medically attended visit during the 30-day follow-up period will also be tabulated after each dose and overall.

The percentage of subjects reporting each individual solicited local AE (any grade and Grade 3) and solicited general AE (any grade, Grade 3, any related and Grade 3 related) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.

For fever, the number and percentage of subjects reporting fever by half degree (°C) cumulative increments during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) will be tabulated for each group after each dose and overall.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Similar tabulations will be performed for any fever with a causal relationship to vaccination and for Grade 3 (> 39.0°C/102.2°F) causally related fever.

For each group and for each hematology and biochemistry parameter:

- The percentage of subjects having hematology and biochemistry results below or above the laboratory normal ranges will be tabulated by time point.
- The summary of grading post-vaccination will be tabulated versus baseline. (Grades will be based on the FDA Guidance for Industry "Toxicity Grading Scale for Healthy Adults and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials", see APPENDIX C in the protocol. Those laboratory parameters not included on FDA Toxicity Grading Scale will not be graded).

The percentage of subjects with any unsolicited AEs during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) with its exact 95% CI will be tabulated by group and by Medical Dictionary for Regulatory Activities (MedDRA) preferred term. Similar tabulation will be done for Grade 3 unsolicited AEs, for any causally related unsolicited AEs, for Grade 3 causally related unsolicited AEs and for unsolicited AEs resulting in a medically attended visit. The verbatim reports of unsolicited AEs will be reviewed by a physician and the signs and symptoms will be coded according to the MedDRA Dictionary for Adverse Reaction Terminology. Every verbatim term will be matched with the appropriate Preferred Term.

The percentage of subjects with at least one report of SAE classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. SAEs will also be described in detail.

For Part A only, pregnancy and pregnancy outcomes will be listed (if applicable).

For Part B only, the percentage of subjects with at least one pIMD classified by the MedDRA Preferred Terms and reported during the entire study period will be tabulated with exact 95% CI. PIMDs will also be described in detail.

The percentage of subjects using concomitant medication (any medication, any antipyretic and any antipyretic taken prophylactically, respectively) during the 7-day follow-up period (i.e., on the day of vaccination and 6 subsequent days) and during the 30-day follow-up period (i.e., on the day of vaccination and 29 subsequent days) will be summarized by group after each vaccine dose and overall.

The analysis of safety will also be performed by age category (age at Dose 1: 60-69 years and 70-80 years in Part B only).

## 5.4.2. Additional considerations

All analyses will be descriptive and will be based on the Exposed Set (ES).

Compliance in completing solicited adverse events information will be tabulated after each dose and overall.

The percentage of subjects with at least **one local solicited** AE, with at least **one general solicited** AE and with **any solicited** AE during the 7-day follow-up period will be tabulated with exact 95% confidence interval (CI) after each dose and overall. The same computations will be done for Grade 3 AEs, for any AEs considered related to vaccination, and for Grade 3 AEs considered related to vaccination.

The number of days with solicited symptoms reported during the **7-day follow-up period** will be tabulated for each solicited adverse event, after each dose using descriptive statistics (mean, min, Q1, median, Q3, maximum).

The same tabulation will be done for Grade 3 symptoms, and also during **the whole post-vaccination period** (to include the total number of days for symptoms ongoing beyond the follow-up period).

The incidence of each solicited symptom (any grade and grade 3) will also be represented graphically per group and per dose.

Analysis of solicited symptoms will also be done on the **pooled groups according to adjuvant content** (AS01B, AS01E, Plain), overall and by age category.

#### 5.4.2.1. Solicited Adverse Events

Solicited adverse events will be reported daily during the 7-day (from Day 1 to Day 7) follow up period after each vaccination, using structured diaries. Missing or non-evaluable measurements will not be replaced.

In order to summarize the data, the maximum intensity of local injection site redness/swelling (in mm) and fever (in °C) will be categorized as follows:

| Grading | Redness/swelling | Fever |
|---------|------------------|-----------------------------------------|
| 0: | ≤ 20 mm | < 38.0°C (100.4°F) |
| 1: | > 20 - ≤ 50 mm | ≥ 38.0°C (100.4°F) - ≤ 38.5°C (101.3°F) |
| 2: | > 50 - ≤ 100 mm | > 38.5°C (101.3°F) - ≤ 39.0°C (102.2°F) |
| 3: | > 100 mm | > 39.0°C (102.2°F) |

Fever is defined as temperature  $\geq 38.0^{\circ}\text{C} / 100.4^{\circ}\text{F}$  (regardless of the location of measurement). The preferred location for measuring temperature in this study will be the oral cavity. Body temperature will also be summarized by  $0.5^{\circ}\text{C}$  increments as follows:  $\geq 38.0, >38.5, >39.0, >39.5, >40.0^{\circ}\text{C}$ .

Each subject's data will be summarized according to the maximal severity observed during the follow-up period for each adverse event and each dose, followed by a summary across subjects and across doses.

#### 5.4.2.2. Unsolicited Adverse Events

When an unsolicited adverse event occurs more than once for a subject, the maximal severity and strongest relationship to the vaccine group will be counted. The selection of unsolicited AEs reported during the follow-up period will be done using the day of onset.

The analysis of unsolicited adverse events includes the following categories:

- Any unsolicited adverse event.
- Possibly related unsolicited adverse events.
- Grade 3 unsolicited adverse events
- Grade 3 possibly related unsolicited adverse events.
- Serious adverse events (SAEs)
- Possibly related SAEs.
- Potential Immune-Mediated disease (pIMDs, in Part B only)
- Medically attended adverse events

SAEs and pIMDs reported during the entire study period will be tabulated.

In addition, the following time periods will be considered to report SAEs/pIMDs at the first and second analyses (E1\_02 and E1\_03, see section 7.1):

- from Dose 1 up to 30 days post dose 2 (or up to 90 days post dose 1 for subjects who did not received the second dose)
- from Dose 1 up to 6 months\* post dose 2 (or up to 8 months\* post dose 1 for subjects who did not received the second dose).
  - \* months will be converted in days in order to select the events for the output tables.
- Listing of AEs/SAEs leading premature withdrawal from study or to interruption of vaccination will be described in detail.

## 5.4.2.3. Combined Solicited and Unsolicited Adverse Events

A summary of subjects with all combined solicited (regardless of their duration) and unsolicited adverse events will be provided. Solicited adverse events will be coded by MedDRA as per the following codes

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

| Solicited symptom | Lower level term code | Corresponding Lower level term decode |
|---|---|---|
| Pain | 10022086 | Injection site pain |
| Erythema | 10015150 | Erythema |
| Swelling | 10053425 | Swelling at injection site |
| Fatigue | 10016256 | Fatigue |
| Fever | 10016558 | Fever |
| Gastrointestinal symptoms | 10017944 | Gastrointestinal disorder |
| Headache | 10019211 | Headache |
| Myalgia | 10028411 | Myalgia |
| Shivering | 10040558 | Shivering |
| Arthralgia | 10003239 | Arthralgia |

For clintrial.gov and EudraCT posting purposes, a summary of combined solicited and unsolicited non-serious adverse events will be produced by System Organ Class and preferred terms and according to occurrence of each event.

## 5.4.2.4. Clinical Safety Laboratory Investigations

In case of invalid or missing results or clinically significant grade 3 and above abnormal laboratory findings, a repeat testing may be done to confirm the first result (see Protocol section 7.1.4). For the analysis, the following rules will be applied:

- In general, the first result will be considered, except if this result is missing.
- In case of retesting for a grade 3 at pre-vaccination, the retesting will be considered if the result is < grade 3.

#### 5.4.2.5. Concomitant Medication

Medications will be coded using the GSKDRUG dictionary.

# 5.5. Analysis of RTI for Part B

# 5.5.1. Analysis of RTI planned in the protocol

The analysis will be performed on the ES.

Any RTI episode for which a visit for the assessment of potential RSV-RTI has been performed (with nasal/throat swab sampling) will be considered for the analysis. The assessment of RSV infection will be performed using qRT-PCR on nasal/throat swabs separately for samples collected by the subject and those collected by an appropriately qualified person (i.e., medical or nursing) at the assessment visit.

The proportion of subjects with at least one RSV-associated RTI (with 95 % CI) will be calculated by group.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Descriptive analyses (mean, median, min, max) of viral load assessed by quantitative PCR (RSV-A/B) of RSV-RTI will be performed by study group.

The incidence rate of all-cause RTI (with 95% CI) will be calculated by group. These will also be presented by co-infection identified by multiplex PCR.

#### 5.5.2. Additional considerations

The mean viral load of the RSV positive-RTI samples will also be reported by collection method (at assessment visit or at home) and by collection time (0-2, 3-4, >4 days between RTI onset date of symptoms and collection date).

Information collected at assessment visit will be described for RSV RTI episodes versus Non-RSV RTI episodes, as tested by qRT-PCR on nasal/throat swabs collected at assessment visit. It will include: vital signs, clinical symptoms, self-collected nasal swab result, medically attended visit and SAE related to the episode.

RTI episodes will be described in detail in a listing. In addition, baseline RSV A Neutralizing antibody titer (GMT and 95% CIs) will be presented graphically by RTI episode status (RSV-RTI vs Non RSV-RTI vs No RTI).

## 6. ANALYSIS INTERPRETATION

All analyses will be descriptive with the aim to characterize the difference in safety/reactogenicity or immunogenicity between groups.

All comparisons will be exploratory. They should be interpreted with caution considering that there is no adjustment for multiplicity for these comparisons, except for the comparisons of all RSV formulations vs Placebo (Dunnett's adjustment).

## 7. CONDUCT OF ANALYSES

# 7.1. Sequence of analyses

The analyses will be performed stepwise:

• A first analysis will be performed on all data available and as clean as possible, when data for at least primary and secondary endpoints up to Day 91 are available (except for cell-mediated immune response at pre-Dose 2 [Day 61] in Part A and Part B and the occurrence of RSV RTI in Part B). This will include results from all subjects in Part A and Part B. This analysis will be considered as final for those endpoints. A clinical study report will be written.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

At this point, the statistician will be unblinded (i.e., individual subject treatment assignments will be available), but no individual listings will be provided to the study team. Given that summary safety results may unblind some specific subjects, the study will be considered as single-blind from this point onwards, with subjects remaining blinded up to study end (Visit 8, Month 14). The investigators will not be provided with the individual data listings or with the randomization listings until the end of study analysis.

- A second analysis will be performed when all safety data up to Month 8 (Visit 7) are available (data as clean as possible). At this time, the following analyses will be performed:
  - The safety analysis of data up to 6 months post-Dose 2.
  - The analysis of all qPCR data available at that time.
  - The analysis of any additional laboratory results up to one month post-Dose 2 that may become available for all planned subjects in Part B.
- A third immunogenicity analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 8 are available, to evaluate the persistence up to 6 months post-Dose 2 in Part B.
- A fourth analysis will be performed when data for at least tertiary immunogenicity endpoints related to persistence (humoral and cell-mediated immunogenicity) up to Month 14 (Visit 8) are available for the subjects enrolled in Step 1 of Part B. This analysis will include any additional laboratory results that may become available at that time.
  - No individual listings will be provided before the final end of study analysis.
- The final end of study analysis will be performed when all data for at least primary and secondary endpoints up to study conclusion are available (Month 14). All available tertiary endpoints will also be analysed in this step. Individual listings will only be provided at this stage. An integrated clinical study report containing all available data will be written and made available to the investigators.

If the data for tertiary endpoints become available at a later stage, (an) additional analysis/ analyses will be performed. These data will be documented in annex(es) to the study report and will be made available to the investigators at that time.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

| Description | Analysis<br>ID | Disclosure Purpose<br>(CTRS=public posting, SR=study report,<br>internal) | Reference for TFL TOC |
|---|---|---|---|
| Final analysis | E1_01 | SR, CTRS | See column A in TFL TOC |
| Analysis up to Day 91 | E1_02 | SR, CTRS | See column B in TFL TOC |
| Analysis up to<br>Month 8 (safety<br>and PCR) | E1_03 | Internal | See column C in TFL TOC |
| Analysis up to<br>Month 8 (immuno) | E1_04 | Internal | See column D in TFL TOC |
| Analysis up to<br>Month 14 (Part B<br>Step 1) | E1_05 | Internal | See column E in TFL TOC |

# 7.2. Statistical considerations for interim analyses

All analyses will be conducted on final data (as clean as possible) and therefore no statistical adjustment for interim analyses is required.

# 8. CHANGES FROM PLANNED ANALYSES

The fold-increase parameter for CMI (post over pre-vaccination) that will be summarised by group using descriptive statistics (N, geometric mean [GM], min, Q1, median, Q3, max) at each time point during which blood samples are collected for CMI has been adapted as follows:

• *Fold increase (Post over pre-vaccination)* of the frequency of RSVPreF3-specific CD4+ T-cells identified as expressing at least 2 marker(s) among IL-2, CD40L, TNF-α, IFN-γ, *as measured by ICS using PBMCs*.

This analysis was also added for the Memory B cells:

• Fold increase (post over pre-vaccination) of the frequency of RSVPreF3-specific memory B-cells, as measured by ELISpot using PBMCs.

All additional analysis planned compared to protocol are described in the "Additional considerations sections". The mains ones to be included in the CSR are also described below (changes indicated in bold):

- Demography and baseline characteristics will be summarized by country.
- Vital signs at baseline will be described by group using descriptive statistics.
- Exposure to study vaccine will be tabulated by group and by vaccine
- The ratio of fold increase (post over pre-vaccination) of RSVPreF3 ELISA antibody concentrations over the fold increase (post over pre-vaccination) of RSV neutralizing antibody titers will be reported for RSV-A *and RSV B*.
- Comparisons with Placebo will be done *at Day 31* and Day 91, for both RSV A Neutralizing antibody *and CD4+ T cells expressing at least 2 markers*.

- Analyses of solicited symptoms were added: incidence of any/local/general solicited AEs, number of days with solicited AEs, analysis on pooled groups according to adjuvant content.
- RTI episodes: analysis of viral load by collection method and collection time was added, as well as the description of signs and symptoms for RSV-RTI vs Non-RSV RTI cases.

# 9. NON-STANDARD DATA DERIVATION RULES AND STATISTICAL METHODS

The following sections describe additional derivation rules and statistical methods which are not presented in section 10.1).

# 9.1. Handling of missing data

## 9.1.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following rules will be applied:

- Adverse event start dates with missing day:
  - If the month is not the same as the vaccine dose, then the imputed start date will be the 1st of the month
  - If the event starts in the same month as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the vaccine dose given during that month. If 'before vaccination' is selected, the imputed date will be one day before the vaccine dose given during that month.
- Adverse event start dates with missing day and month:
  - If the year is not the same as the vaccine dose, then the imputed start date will be the 1st of January.
  - If the event starts in the same year as the vaccine dose, the flag indicating if the event occurred before or after vaccination (AE.AESTRTPT) will be used to complete the date. If 'after vaccination' is selected, the imputed start date will match the first vaccine dose given during that year. If 'before vaccination' is selected, the imputed date will be one day before the first vaccine dose given during that year.
- Adverse event end dates with missing day: the imputed end date will be the last day of the month (30 or 31) or the study conclusion date whichever comes first.
- Adverse event end dates with missing day and month: the imputed end date will be the last day of the year (31st of December) or the study conclusion date whichever comes first.

All other cases of incomplete AE or concomitant medication/vaccination start date will follow the standard rules above.

## 10. ANNEXES

# 10.1. Business rules for standard data derivations and statistical methods

This section contains GSK Vaccines' standard rules for data display and derivation for clinical and epidemiological studies. These rules will be applied along with those detailed in section 9 (additional study-specific rules).

# 10.1.1. Attributing events to vaccine doses

The dose relative to an event is the most recent study dose given to a subject prior to the start of a given event. For example, if the start date of an adverse event is between Dose 1 and Dose 2, the relative dose will be Dose 1.

If an event starts on the same day as a study dose, the relative dose will be derived from the additional information provided in the CRF using the contents of the flag indicating if the event occurred before or after vaccination. If 'after vaccination' is selected, the relative dose for the event will be the one administered on the start day of the event. If 'before vaccination' is selected, the relative dose for the event will be the dose prior to this one

# 10.1.2. Handling of missing data

#### 10.1.2.1. Dates

When partially completed dates (i.e. with missing day or month) are used in calculations, the following standard rules will be applied:

- A missing day will be replaced by 15
- A missing day and month will be replaced by June 30<sup>th</sup>.

See also exceptions in section 9.1.

## 10.1.2.2. Laboratory data

Missing laboratory results (including immunological data) will not be replaced.

# 10.1.2.3. Daily recording of solicited symptoms

## 10.1.2.3.1. Studies with electronic diaries

For studies using electronic diaries for the collection of solicited symptoms, symptoms will be considered present only when a daily recording of grade 1 or more is present.

## 10.1.2.4. Unsolicited adverse events

Missing severity, relationship with study vaccine, and outcome of unsolicited adverse events will not be replaced and will appear as 'UNKNOWN' in all statistical output.

## 10.1.3. Data derivation

## 10.1.3.1. Age at vaccination in years

When age at vaccination is to be displayed in years, it will be calculated as the number of complete calendar years between the date of birth and the date of vaccination. For example:

DOB = 10SEP1983, Date of vaccination = 09SEP2018 -> Age = 34 years

DOB = 10SEP1983, Date of vaccination = 10SEP2018 -> Age = 35 years

## 10.1.3.2. Temperature

Temperatures will be presented in degrees Celsius (°C). Temperatures reported in degrees Fahrenheit (°F) will be converted as follows:

Temperature (Celsius) =  $((Temperature (Fahrenheit) - 32) \times 5)/9$ 

Conversion of temperature from °Fahrenheit to °C will be performed according to SDTM specifications.

## 10.1.3.3. Numerical serology results

Numerical serology results will be derived from the content of IS.ISORRES in the SDTM dataset. For assays with a specific cut-off, the following derivation rules apply:

| IS.ISORRES | Derived value |
|-----------------------------------------|---------------|
| "NEG", "-", or "(-)" | cut-off/2 |
| "POS", "+", or "(+)" | cut-off |
| "< value" and value is <= assay cut-off | cut-off/2 |
| "< value" and value is > assay cut-off | value |
| "> value" and value is < assay cut-off | cut-off/2 |
| "> value" and value is >= assay cut-off | value |
| "value" and value is < cut-off | cut-off/2 |
| "value" and value is >= cut-off | value |
| All other cases | missing |

# 10.1.3.4. Geometric mean titers (GMTs) and concentrations (GMCs)

Geometric Mean Titer (GMT) or Concentration (GMC) calculations are performed by taking the inverse logarithm of the mean of the log titer or concentration transformations. Antibody titers or concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMT/GMC calculation. The cut-off value is defined by the laboratory before the analysis and is described in the protocol.

# 10.1.3.5. Onset day

The onset day for an event (e.g. AE, medication, vaccination) is the number of days between the last study vaccination and the start date of the event. This is 1 for an event occurring on the same day as a vaccination (and reported as starting after vaccination).

#### 10.1.3.6. Duration of events

The duration of an event with a start and end date will be the number of days between the start and end dates plus one day, i.e. an event that starts on 03MAR2018 and ends on 12MAR2018 has a duration of 10 days.

The duration of solicited events will be calculated as the sum of the individual days with the symptom reported at grade 1 or higher.

# 10.1.3.7. Counting rules for combining solicited and unsolicited adverse events

For output combining solicited and unsolicited adverse events, all serious adverse events will be considered general events since the administration site flag is not included in the expedited adverse event CRF pages.

Multiple events with the same preferred term which start on the same day are counted as only one occurrence.

# 10.1.3.8. Counting rules for occurrences of solicited adverse events

When the occurrences of solicited adverse events are summarized, each event recorded as having occurred during a specific period will be counted as only one occurrence regardless of the number of days on which it occurs.

## 10.1.4. Display of decimals

## 10.1.4.1. Percentages

Percentages and their corresponding confidence limits will be displayed with:

- no decimals when there are fewer than 50 subjects in each tabulated group
- one decimal when there are at least 50 subjects in at least one tabulated group

Exceptions will be made for percentages that are not 0% or 100% but appear as 0% or 100% due to rounding. For these specific cases the number of decimals will be increased until the displayed value is no longer 0% or 100%. Examples are given in the following table.

| n/N | Displayed percentage |
|-------------|----------------------|
| 10/45 | 22% |
| 1/45 | 2% |
| 10/55 | 18.2% |
| 1/55 | 1.8% |
| 1/300 | 0.3% |
| 1/3000 | 0.03% |
| 1/30000 | 0.003% |
| 299/300 | 99.7% |
| 2999/3000 | 99.97% |
| 29999/30000 | 99.997% |

- The display of additional decimals for values close to 0% or 100% will be applied only to point estimates and not confidence limits, which can be rounded and displayed as 0% or 100%.
- Values of exactly 0% or 100% will be presented with no decimals regardless of the number of subjects per tabulated group.

## 10.1.4.2. Demographic/baseline characteristics statistics

The mean, median, and standard deviation for continuous baseline characteristics will be presented with one decimal.

The minimum and maximum values and quartile values (if required) will be presented with the same number of decimals as the observed values.

The maximum and minima of transformed body temperatures will be displayed with one decimal.

# 10.1.4.3. Serological summary statistics

The number of decimals used when displaying geometric mean titers (GMT) or concentrations (GMC) and their confidence limits is shown in the following table:

| GMT or GMC value | Number of decimals to display |
|------------------|-------------------------------|
| <0.1 | 3 |
| >=0.1 and <10 | 2 |
| >=10 and <1000 | 1 |
| >=1000 | 0 |

When multiple categories of GMT or GMC values are present in the same table, the number of decimals displayed should match that of the smallest category (i.e. the one with the higher number of decimals). For example, if GMT or GMC values of <0.1 appear in the same table as values of >=0.1 and <10, 3 decimals should be displayed for both.

GMT or GMC ratios and their confidence limits will be displayed with 2 decimals regardless of the actual values.

# 10.1.5. Statistical methodology

# 10.1.5.1. Exact confidence intervals around proportions

The exact confidence intervals around within-group proportions are derived using the method of Clopper and Pearson [Clopper, 1934].

## 10.1.5.2. Adjusted GMT or GMC ratios

When between-group GMT or GMC ratios are computed and adjusted for two-level categorical co-variables, these co-variables should be included as dummy continuous variables in the SAS procedure.

## 10.2. TFL ToC

The TFL TOC provides the list of tables/figures/listings that will be generated at each analysis. It can be found in eTMF folder section 11.01.01.

The mock tables/figures referred under column named 'layout' can be found in section 12.

# 11. REFERENCES

Clopper CJ, Pearson E. The Use of Confidence or Fiducial Limits Illustrated in the case of the Binomial. *Biometrika*. 1934;26:404-13.

# 12. STUDY MOCK TFLS

The following drafted standard and study specific mocks will be used. Note that standard templates might be updated based on the last version of the standard catalogue used at the time of analysis. Titles and footnotes will be adapted accordingly.

The data display, title and footnotes are for illustration purpose and will be adapted to the study specificity as indicated in the TFL TOC. Note that there may be few changes between the study specific SAP mock TFL and the final TFLs as editorial/minor changes do not require a SAP amendment.

# 12.1. Demography

Template 1 Summary of demography and baseline characteristics (Exposed Set)

| | <each group=""><br/>N=XXXX</each> | | Total<br>N=XXXX | |
|---|---|---|---|---|
| | Value or n | % | Value or n | % |
| Age (years) at first vaccination | | | | |
| N | XXX | | XXX | |
| Mean | XXX.X | | XXX.X | |
| Standard Deviation | XXX.X | | XXX.X | |
| Median | XXX.X | | XXX.X | |
| Minimum | XXX | | XXX | |
| Maximum | XXX | | XXX | |
| Sex | | | | |
| Male | XXX | XX.X | XXX | XX.X |
| Female | XXX | XX.X | XXX | XX.X |
| Ethnicity | | | | |
| <each ethnicity=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Race | | | | |
| <each race=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |
| Age category | | | | |
| <each age="" category=""></each> | XXX | XX.X | XXX | XX.X |
| | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n/% = number / percentage of subjects in a given category

Value = value of the considered parameter

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

# Template 2 Number of subjects by country and center (Exposed Set)

| | | <each<br>N=X</each<br> | • . | Tot<br>N=XX | |
|---|---|---|---|---|---|
| Country | Center-Investigator Name | n | % | n | % |
| <each< td=""><td><each center-investigator="" name=""></each></td><td>XXX</td><td>XX.X</td><td>XXX</td><td>XX.X</td></each<> | <each center-investigator="" name=""></each> | XXX | XX.X | XXX | XX.X |
| country> | All | XXX | XX.X | XXX | XX.X |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given center or country

 $% = (n/N) \times 100$ 

# Template 3 Number of subjects by study steps (Exposed Set)

| | | group><br>XXX | | otal<br>XXXX |
|---------------|---|---------------|---|--------------|
| Steps | n | % | n | % |
| Part A | | | | |
| Part B Step 1 | | | | |
| Part B Step 2 | | | | |

Short group label = long group label

N = total number of subjects

n = number of subjects in a given category

 $% = (n/N) \times 100$ 

# Template 4 Summary of vital signs (Exposed Set)

| | | | <each group=""><br/>N=XXXX</each> | Total<br>N=XXXX |
|---|---|---|---|---|
| Visit | Characteristics | Parameters | Value | Value |
| <each visit=""></each> | | n | XXX | XXX |
| | , | Mean | xxx.x | xxx.x |
| | | SD | xxx.x | xxx.x |
| | | Median | XXX.X | xxx.x |
| | | Minimum | XXX | xxx |
| | | Maximum | XXX | xxx |
| | Respiratory rate ( <unit>)</unit> | n | XXX | XXX |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | xxx |
| | | Maximum | XXX | XXX |
| | Systolic Blood pressure ( <unit>)</unit> | n | XXX | xxx |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | xxx |
| | Diastolic blood pressure ( <unit>)</unit> | n | XXX | xxx |
| | | Mean | XXX.X | xxx.x |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX<br>XXX.X<br>XXX.X<br>XXX<br>XXX<br>XXX<br>XXX |
| | Pulse oximetry ( <unit>)</unit> | n | XXX | xxx |
| | | Mean | XXX.X | XXX.X |
| | | SD | XXX.X | XXX.X |
| | | Median | XXX.X | XXX.X |
| | | Minimum | XXX | XXX |
| | | Maximum | XXX | XXX |
| | Pre-vaccination Temperature (C) | n | | |
| | | Mean | | |
| | | SD | | |
| | | Median | | |
| | | Minimum | | |
| | | Maximum | | |

Short group label = long group label

N = total number of subjects

Value = value of the considered parameter

n = number of subjects in a given category

N with data = number of subjects with documentation of the corresponding data

SD = standard deviation

# Template 5 Summary of study completion with reason for withdrawal (Exposed Set)

| | <each (<br="">N=X)</each> | | Total<br>N=XXXX | |
|---|---|---|---|---|
| | n | % | n | % |
| Completed the study | XXX | XX.X | XXX | XX.X |
| Withdrawn from the study | XXX | XX.X | XXX | XX.X |
| Primary reason for withdrawal : | | | | |
| <each reason=""></each> | XXX | XX.X | XXX | XX.X |

Short group label = long group label

## Template 6 Summary of visit attendance (Exposed Set)

| | | | <each group=""><br/>N=XXXX</each> | | otal<br>XXXX |
|---|---|---|---|---|---|
| Visit | Status | n | % | n | % |
| <each visit=""></each> | Attended | XX | XX.X | XX | XX.X |
| | Did not attend yet | XX | XX.X | XX | XX.X |
| | Withdrawal at visit or earlier | XX | XX.X | XX | XX.X |
| | Did not attend | XX | XX.X | XX | XX.X |

Short group label = long group label

N = Number of subjects in each group or in total

n/% = number / percentage of subjects in a given category

Template 7 Summary of important protocol deviations leading to elimination from any analyses (Enrolled Set)

| Category<br>Sub-category | | <each group=""> N=XXX</each> | | | Total<br>N=XXX | |
|---|---|---|---|---|---|---|
| | Осс | n | % | Осс | n | % |
| At least one Important Protocol Deviation | | | | | | |
| < Each category > | | | | | | |
| <each sub-category=""></each> | | | | | | |

Short group label = long group label

N = Total number of subjects

Occ = number of occurrences = number of important protocol deviations

n/% = number / percentage of subjects with important protocol deviations

Template 8 Summary of subject disposition from Enrolled set to Randomized set (Enrolled Set)

| | | otal<br>N= |
|-----------------------------------------------|---|------------|
| | n | % |
| Withdrawals prior to randomization | | |
| <withdrawal 1="" reason=""></withdrawal> | | |
| <withdrawal 2="" reason=""></withdrawal> | | |
| Number of subjects included in randomized set | | |

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Template 9 Summary of subject disposition from Randomized Set to Exposed set (Randomized set)

| | | ch group> | | tal<br>XXXX |
|---|---|---|---|---|
| | n % | | n | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Exposed set | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Template 10 Summary of subject disposition from Exposed Set to Per Protocol Set at visit x (Exposed set)

| | | h group><br>=XXXX | Total N=XXXX | |
|---|---|---|---|---|
| | n | n % | | % |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Number of subjects included in the Per Protocol set at visit x | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Template 11 Summary of subject disposition from Exposed Set to End of study (Exposed set)

| | <each group=""> N=XXXX</each> | | | otal<br>XXXX |
|---|---|---|---|---|
| | n | % | n | % |
| Eliminations | | | | |
| <elimination (code)="" 1="" reason=""></elimination> | | | | |
| <elimination (code)="" 2="" reason=""></elimination> | | | | |
| Withdrawals | | | | |
| <withdrawal 1="" reason=""></withdrawal> | | | | |
| <withdrawal 2="" reason=""></withdrawal> | | | | |
| Number of subjects who completed the study | | | | |
| Completed with 1 dose | | | | |
| Completed with 2 doses | | | | |

Short group label = long group label

N = Number of subjects

n = number of subjects enrolled by center

% = n / Number of subjects with available results x 100

Template 12 Deviations from protocol for age and intervals between study visits (Exposed set)

| | | | <each grou<="" th=""><th colspan="2"><each group=""></each></th><th>&gt;</th></each> | <each group=""></each> | | > |
|---|---|---|---|---|---|---|
| Type of interval | Interval range | | Value or n | % | Value or n | % |
| Age | <age range=""></age> | N | XXX | | xxx | |
| | | n | XXX | XX.X | XXX | xx.x |
| | | Minimum | xxx | | XXX | |
| | | Maximum | XXX | | xxx | |
| each interval cetween study visit> | <interval range=""></interval> | N | XXX | | XXX | |
| · | | n | XXX | XX.X | XXX | xx.x |
| | | Minimum | XXX | | xxx | |
| | | Maximum | XXX | | XXX | |

Template 13 Number of enrolled subjects by country

| | | <each group=""> N = XXX</each> | Total<br>N = XXX |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Country | <each country=""></each> | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given country or for all countries

Template 14 Number of enrolled subjects by age category

| | | <each group=""><br/>N =</each> | Total<br>N = |
|---|---|---|---|
| Characteristics | Categories | n | n |
| Age category | Adults [18-64 years] | | |
| | Adults [65-84 years] | | |
| | Missing | | |

Short group label = long group label

N = Number of enrolled subjects

n= number of enrolled subjects included in each group or in total for a given age category or for all age categories Missing = age at study vaccination unknown

Template 15 Minimum and maximum visit dates <analysis set name>

| | | <each group=""></each> | <each group=""></each> | Overall |
|---|---|---|---|---|
| Visit Description | Parameter | Date | Date | Date |
| < each informed consent> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| [Randomization] | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| _ | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| <each visit=""></each> | Minimum | DDMMYYYY | DDMMYYYY | DDMMYYYY |
| | Maximum | DDMMYYYY | DDMMYYYY | DDMMYYYY |

Short group label = long group label

# 12.2. Exposure

Template 16 Exposure to study vaccines by vaccine (Exposed Set)

| | | <each<br>group</each<br> | n<br>>N=XXXX | <each< th=""><th>group&gt;<br/>X</th></each<> | group><br>X |
|---|---|---|---|---|---|
| Vaccine administered | Number of subjects receiving | n | % | n | % |
| < Vaccine A> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | XXX | XX.X | XXX | XX.X |
| < Each vaccine> | Exactly 1 vaccination | XXX | XX.X | XXX | XX.X |
| | Exactly 2 vaccinations | XXX | XX.X | XXX | XX.X |
| | At least 1 vaccination | xxx | XX.X | xxx | xx.x |

Short group label = long group label

N = number of subjects in each group or in total included in the considered analysis set

# 12.3. Immunogenicity

# 12.3.1. Within groups

Template 17 Number and percentage of subjects with <antibody titer /concentration> equal to or above <cut-off unit> and <GMT/Cs> <analysis set name>

| | | | | >=cut-off unit | | | | | GMT/C | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | 959 | % CI | | 95% | % CI | |
| Antibody | Group | Timing | N | n | % | LL | UL | value | LL | UL | Min | Max |
| <each antibody=""></each> | <each<br>group&gt;</each<br> | <each timing=""></each> | | | | | | | | | | |

Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

N = Number of subjects with available results

n% = number/percentage of subjects with titer/concentration equal to or above specified value

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

MIN/MAX = Minimum/Maximum

Short timing label = long timing label

n = number of subjects/doses in the given category

<sup>% =</sup> percentage of subjects in the given category

Template 18 <GMT/Cs> and their 95% Cls for <antibody titers/ concentrations> <analysis set name>



Short group label = long group label

GMT/C = geometric mean antibody titer/concentration

95% CI = 95% confidence interval

Short timing label = long timing label

Note: This graph is provided as an example.

For RSV A Nab and RSVPreF3- specific IgG Ab, it will be adapted to display all the groups (4 groups for Part A, 10 groups for Part B) and all available timepoints (4 TPs up to Day 91, 6 TPs up to study end for Part B).

If needed for Part B, this graph might be split in several graphs: either by adjuvant content vs Placebo or by antigen content vs Placebo.

Same graph will be generated for RSV B NAb with 2 timepoints (10 groups, at Days 1 and 91), and for RSVPreF3 site 0 Ab with 2 groups and 2 timepoints (selected formulation and Placebo groups, at Days 1 and 91).

Template 19 Geometric mean of the individual ratio of <antibody titers/concentrations (units)> post-vaccination compared to pre-vaccination <Per Protocol Set>

| | | | <gmt,c> ratio</gmt,c> | | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% C | | | | |
| Group | N | Time point | <gmt,c></gmt,c> | Time point | <gmt,c></gmt,c> | Ratio order | Value | LL | UL |
| - | | description | | description | | | | | |
| <each< td=""><td>XXX</td><td>PI(D31)</td><td></td><td>PRE</td><td></td><td>PI(D31) / PRE</td><td></td><td></td><td></td></each<> | XXX | PI(D31) | | PRE | | PI(D31) / PRE | | | |
| group> | | | | | | | | | |
| | | <each point="" time=""></each> | | PRE | | <time point=""> / PRE</time> | | | |

Short group label = long group label

<GMT,C> = geometric mean antibody <titer,concentration>

N = Number of subjects with available results at the two considered time points

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

# Template 20 Distribution of <antibody titers/concentrations> <Per Protocol Set>

| | | <eac< th=""><th>h gro</th><th></th><th></th><th colspan="3"><each group=""></each></th><th></th><th></th></eac<> | h gro | | | <each group=""></each> | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | <95> | % CI | | | | <95>% CI | |
| Antibody | Timing | <titer concentration=""></titer> | N | n | % | LL | UL | N | n | % | LL | UL |
| <each antibody=""></each> | <each timing=""></each> | < cut-off1 | XX | ХХ | XX.X | XX.X | XX.X | xx | XX | XX.X | XX.X | XX.X |
| | | >= cut-off1 | xx | xx | XX.X | xx.x | XX.X | xx | xx | XX.X | xx.x | XX.X |
| | | >= cut-off2 | хх | XX | XX.X | XX.X | XX.X | xx | xx | XX.X | XX.X | XX.X |
| | | >= cut-off3 | xx | xx | XX.X | XX.X | XX.X | ХХ | xx | XX.X | XX.X | xx.x |

Short group label = long group label

N = number of subjects with available results

n/% = number/percentage of subjects with <titer, concentration> within the specified criterion

<95>% CI = <95>% confidence interval; LL = Lower Limit, UL = Upper Limit

Short timing label = long timing label

Template 21 Distribution of <antibody titers/concentrations> fold increase post-vaccination compared to pre-vaccination <Per Protocol Set>

| Fiming<br>each timing> | FI | N | ch gro | • | 95% | CI. | | ch gro | • | | <b>^</b> 1 |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | N | | | 3J /0 | CI | | | | 95% | CI . |
| each timing> | | ., | n | % | LL | UL | N | n | % | LL | UL |
| | < 1 | xx | xx | XX.X | XX.X | XX.X | XX | XX | XX.X | XX.X | XX.X |
| | >= 1 | xx | xx | xx.x | XX.X | XX.X | xx | xx | xx.x | xx.x | xx.x |
| | >= 2 | xx | xx | XX.X | xx.x | XX.X | XX | xx | XX.X | xx.x | xx.x |
| | >= 4 | xx | xx | xx.x | xx.x | xx.x | xx | xx | xx.x | xx.x | xx.x |
| | >= 6 | xx | xx | XX.X | XX.X | XX.X | XX | xx | XX.X | xx.x | XX.X |
| | >= 8 | xx | xx | xx.x | xx.x | xx.x | xx | xx | XX.X | xx.x | xx.x |
| | >= 10 | xx | xx | xx.x | xx.x | xx.x | XX | xx | XX.X | xx.x | xx.x |
| | | >= 2<br>>= 4<br>>= 6<br>>= 8 | >= 2 | >= 2 | >= 2 | >= 2 | >= 2 | >= 2 | >= 2 | >= 2 | >= 2 |

Short group label = long group label

FI= Fold Increase post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available

n/% = number/percentage of subjects with <titer, concentration > fold change meeting the specified criterion

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

Short timing label = long timing label

Template 22 Reverse cumulative distribution curve of <antibody titers/concentrations> in the <group label> group <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: this graph is provided as an example. It will be generated by group, and will be adapted to display the 4 timepoints (PRE, D31, D61, D91) for the considered group. For Part B, same graphs will also be generated at Day 91 with groups according to adjuvant content or antigen content vs Placebo.

For RSV B Nab and RSVPreF3 site 0 specific Ab, the figure will display only 2 timepoints (Days 1 and 91).
Template 23 Kinetics of < antibody GMT/Cs> on subjects with results available at all timepoints up to <Day 91, Month 14> <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. Template will be adapted to display all the groups (10 groups for Part B) and all the timepoints (4 TPs up to Day 91, 6 TPs up to study end).

Template 24 Individual results of <RSV A Neutralizing antibody titer> at <time point> versus pre-vaccination in <group label> and Placebo\_B groups <Per protocol set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated as follows:

RSV A Nab at Day 31 and Day 91, for each RSV groups (18 graphs)

RSVPref3 IgG at Day 31 and Day 91, for each RSV groups (18 graphs)

RSV B Nab at Day 91, for the selected formulation (1 graph)

Template 25 Individual results of <RSV A versus RSV B Neutralizing antibody titer> at <time point> , on pooled RSV groups <Per protocol set>



Note: this graph is provided as an example. It will be generated on pooled RSV groups as follows:

RSV A Nab vs RSVPreF3 IgG at each timepoint

RSV A Nab vs RSV B Nab at Pre and Day 91

RSV B Nab vs RSVPreF3 IgG at Pre and Day 91

The same graphs will be generated on fold increase Post over Pre.

Template 26 Geometric mean ratios of the fold increase (Pre to Post -vaccination) between RSVPreF3 IgG antibody concentrations and <RSV-A, RSV-B> neutralising antibody titers <Per protocol set>

| | GM ra | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | | | | 95% | CI |
| Timepoint | Group | N RSVPref3 95% CI <rsv-a, b=""> 95% Value LL</rsv-a,> | | | | | LL | UL | | |
| • | - | | IgG GMF | LL | UL | Nab GMF | LL | UL | | |
| PI(D31)/PR<br>E | <each group=""></each> | | | | | | | | | |
| <each<br>timepoint&gt;</each<br> | | | | | | | | | | |
| • | | | | | | | | | | |

Short group label = long group label

N = Number of subjects with available results at the two considered time points (post and pre) for both RSVPreF3 lgG and <RSV-A, B> Nab

GMF = Geometric mean fold increase Pre to Post-vaccination

GM ratio of FI=Geometric mean ratio of fold increase (Pre to Post)

95% CI = 95% confidence interval; LL = lower limit, UL = upper limit

Short timing label = long timing label

Template 27 Individual results of the fold increase (post over pre-vaccination) of RSVPreF3 IgG antibody concentrations versus <RSV A, RSV B> neutralizing antibody titers at <time point> in <group label> <Per protocol set>



Short group label = long group label

Note: This graph is provided as an example. It will be generated as follows:

Y axis=RSVPreF3 IgG vs X axis=RSV A Nab, at Days 31 and 91, for each RSV group (18 graphs)

Y axis= RSVPreF3 lgG vs X axis=RSV B Nab at Day 91, for the selected formulation (1 graph)

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 28 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| lmmune<br>Marker | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>xxxx</td></at> | <each timing=""></each> | N | XXXX | xxxx |
| markers> | | GM | XX.X | xx.x |
| | | SD | | |
| | | Minimum | XX.X | xx.x |
| | | Q1 | XX.X | xx.x |
| | | Median | XX.X | xx.x |
| | | Q3 | XX.X | xx.x |
| | | Maximum | XX.X | xx.x |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Note: this table will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC).

Template 29 Descriptive statistics of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS), by pre-vaccination category <Per Protocol Set>

| | | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|---|
| Immune | Pre-vaccination status | | | | |
| Marker | | Timing | Statistic | value | value |
| <at 2<="" least="" td=""><td><q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<></td></at> | <q1< td=""><td><each timing=""></each></td><td>N</td><td>XXXX</td><td>XXXX</td></q1<> | <each timing=""></each> | N | XXXX | XXXX |
| markers> | | | GM | XX.X | XX.X |
| | | | SD | | |
| | | | Minimum | XX.X | XX.X |
| | | | Q1 | XX.X | XX.X |
| | | | Median | XX.X | XX.X |
| | | | Q3 | XX.X | XX.X |
| | | | Maximum | XX.X | XX.X |
| | [Q1-Q3] | <each timing=""></each> | <each< td=""><td></td><td></td></each<> | | |
| | - | | parameter> | | |
| | >Q3 | | | | |
| | Total | | | | |

Short group label = long group label

<Q1= subjects with pre-vaccination frequency < Q1 of the frequencies at pre-vaccination computed on pooled groups Q1-Q3= subjects with pre-vaccination frequency within [Q1-Q3] of the frequencies at pre-vaccination computed on pooled groups

>Q3=subjects with pre-vaccination frequency < Q3 of the frequencies at pre-vaccination computed on pooled groups N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Template 30 Boxplots with individual data of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol set>



Short group label = long group label

Short timing label = long timing label

Note: This graph is provided as an example. Depending on the analysis, it will display groups and timepoints as follows:

Part A: 1 graph with 4 groups and 3 (D1, D31, D91) or 4 timepoints (D1, D31, D61, D91)

Part B: 3 graphs with 4 groups (either by adjuvant content or by antigen content vs Placebo), and 3 timepoints (D1, D31, D91) or 5 timepoints (up to Month 8) or 6 timepoints (up to Month 14, only for selected Ag dose and Placebo)

This graph will be generated for each CMI response defined in section 5.3.2.2 (see TFL TOC).

For Part B, the same graph will be generated for memory B-cells, with 4 groups (selected Ag dose with Plain/AS01E/AS01B, and Placebo) and 4 timepoints (PRE, D31, D91, M14).

Template 31 Frequency of RSVPreF3 specific CD4+ T-cells expressing any combination of markers among IL-2, CD40L, TNFa, IFNg in <group label> group at Day 31 and Day 91 (per million of CD4+ T cells, by ICS) <Per Protocol Set>



Short group label = long group label Short timing label = long timing label

Note: This graph is provided as an example. It will be generated by group and will be adapted to display Q1-Median-Q3 for each combination of the markers (15) at Day 31 and Day 91.

Template 32 Descriptive statistics of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least <2 markers among IL-2, CD40L, TNFa, IFNg> (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immune Marker | Timing | Statistic | value | Value |
| <at 2<="" least="" td=""><td><each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each></td></at> | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>Xxxx</td></each> | N | XXXX | Xxxx |
| markers> | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results at both timepoints (pre and post)

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 33 Descriptive statistics of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| Immuno assay | Timing | Statistic | <each group=""> value</each> | <each group=""> value</each> |
|---|---|---|---|---|
| | • | Stations<br>N | | |
| Memory B cells | <each timing=""></each> | N | XXXX | XXXX |
| | | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

Short timing label = long timing label

Template 34 Descriptive statistics of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-memory B-cells (per million of memory B cells, by Elispot) – Part B <Per Protocol Set>

| | | | <each group=""></each> | <each group=""></each> |
|---|---|---|---|---|
| Immuno assay | Timing | Statistic | value | value |
| Memory B cells | <each post-<="" td="" timing=""><td>N</td><td>XXXX</td><td>XXXX</td></each> | N | XXXX | XXXX |
| | vaccination> | GM | XX.X | XX.X |
| | | SD | | |
| | | Minimum | XX.X | XX.X |
| | | Q1 | XX.X | XX.X |
| | | Median | XX.X | XX.X |
| | | Q3 | XX.X | XX.X |
| | | Maximum | XX.X | XX.X |

Short group label = long group label

N= Number of subjects with available results

GM= Geometric mean

SD= Standard Deviation

Q1 and Q3= 25th and 75th percentiles

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 35 Distribution of the fold increase (post over pre-vaccination) of the frequency of RSVPreF3 specific-CD4+ T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg (per million of CD4+ T cells, by ICS) <Per Protocol Set>

| | | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th></th><th></th><th><ea< th=""><th>ch gro</th><th>up&gt;</th><th></th><th></th></ea<></th></ea<> | ch gro | up> | | | <ea< th=""><th>ch gro</th><th>up&gt;</th><th></th><th></th></ea<> | ch gro | up> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | , | | | 95% | CI | | | | 95% ( | )I |
| Assay | Timing | FI | N | n | % | LL | UL | N | n | % | LL | UL |
| <assay name=""></assay> | <each timing=""></each> | < 2 | xx | XX | XX.X | XX.X | XX.X | XX | xx | XX.X | XX.X | XX.X |
| | | >= 2 | xx | xx | xx.x | xx.x | xx.x | xx | xx | xx.x | xx.x | xx.x |
| | | >= 4 | xx | xx | xx.x | xx.x | xx.x | xx | xx | XX.X | xx.x | xx.x |
| | | >= 6 | xx | xx | xx.x | xx.x | xx.x | xx | xx | XX.X | xx.x | xx.x |
| | | >= 8 | xx | xx | xx.x | xx.x | xx.x | xx | xx | xx.x | xx.x | xx.x |
| | | >= 10 | xx | xx | xx.x | XX.X | xx.x | xx | xx | xx.x | XX.X | xx.x |

Short group label = long group label

FI= Fold increase Post over pre-vaccination result

N = number of subjects with pre and corresponding post-vaccination results available n/% = number/percentage of subjects with fold increase meeting the specified criterion

95% CI = 95% confidence interval; LL = Lower Limit, UL = Upper Limit

### 12.3.2. Between groups

Template 36 Comparisons of the 9 RSV formulations versus Placebo in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at one month post <dose 1 (Day 31), dose 2 (Day 91)> (ANCOVA model, Dunnett's test) – Part B <Per Protocol set>

| Assay | Timepoint | RSV group | N | GM <t,f> ratio</t,f> | Dunne | tt's 95% CI | Dunnett's |
|---|---|---|---|---|---|---|---|
| | | | | (RSV over Placebo) | LL | UL | p-value |
| <assay name=""></assay> | <day 31,="" 91="" day=""></day> | 30-PLAIN_B | | | | | |
| - | | 60-PLAIN_B | | | | | |
| | | 120-PLAIN_B | | | | | |
| | | 30-AS01E_B | | | | | |
| | | 60-AS01E_B | | | | | |
| | | 120-AS01E_B | | | | | |
| | | 30-AS01B_B | | | | | |
| | | 60-AS01B_B | | | | | |
| | | 120-AS01B_B | | | | | |

Short group label = long group label

N= Number of subjects with both pre- and post-vaccination results available

GM<T,F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

RSV Vaccine is considered superior to Placebo if one-sided p-value <0.025

Dunnett's 95% CI = 95% confidence interval based on Dunnett's adjustment, LL = lower limit, UL = upper limit ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the treatment and age category as fixed effects

Template 37 Comparisons of the mean responses post dose 2 (Day 91) versus post dose 1 (Day 31) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> on pooled groups according to adjuvant content (ANCOVA model) – Part B <Per Protocol set >

| Assay | RSV group | N | GM <t,f> ratio</t,f> | 95% | CI | p-value |
|---|---|---|---|---|---|---|
| _ | | | (D91/D31) | LL | UL | |
| <assay name=""></assay> | PLAIN_B | | | | | |
| | AS01E_B | | | | | |
| | AS01B_B | | | | | |

Short pooled group label = long pooled group label

N= Number of subjects with results available at both timepoints

GM<T,F>= = Geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

PII D91 is considered as significantly higher to PI D31 if one-sided p-value <0.025

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance);

LL = lower limit. UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the adjuvant content, antigen dose and age category as fixed effects

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 38 Comparisons of the RSV groups pooled according to their adjuvant content (Plain, AS01E, AS01B) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) - Part B <Per Protocol set>

| | | | G | Group 1 | | | | Group 2 | | | | | GM <t,f> ratio<br/>(Group 1 /<br/>Group 2)</t,f> | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | | 5%<br>CI | | | | | 5%<br>CI | | 95% | CI | |
| | | Group 1 | N | GM <t,f></t,f> | LL | UL | Group 2 | N | GM <t,f></t,f> | | | Value | LL | UL | p- |
| Assay | Timepoint | | | | | | | | | LL | UL | | | | value |
| <assay< td=""><td><each< td=""><td>AS01B_B</td><td></td><td></td><td></td><td></td><td>PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<></td></assay<> | <each< td=""><td>AS01B_B</td><td></td><td></td><td></td><td></td><td>PLAIN_B</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | AS01B_B | | | | | PLAIN_B | | | | | | | | |
| name> | timing> | AS01E_B | | | | | PLAIN_B | | | | | | | | |
| | | AS01B_B | | | | | AS01E_B | | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance);

LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and adjuvant content, antigen dose and age category as fixed effects Group 1 is considered superior to Group 2 if one-sided p-value <0.025

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 39 Comparisons of the RSV groups (by antigen dose level) in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg> at Day 91 (ANCOVA model) – Part B <Per Protocol set >

| | | | Gr | oup 1 | | | Gı | oup 2 | | GM <t,f<br>(Grou</t,f<br> | ıp 1 / | ) | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 5%<br>CI | | | | 5%<br>CI | | 95% | CI | |
| Assay | Timepoint | Group 1 | N | GM <t,f></t,f> | | Group 2 | N | GM <t,f></t,f> | | Value | LL | | p-value |
| <assay< td=""><td><each< td=""><td>120-</td><td></td><td></td><td></td><td>60-</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<></td></assay<> | <each< td=""><td>120-</td><td></td><td></td><td></td><td>60-</td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | 120- | | | | 60- | | | | | | | |
| name> | timing> | PLAIN_B | | | | PLAIN_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | PLAIN_B | | | | PLAIN_B | | | | | | | |
| | | 60-PLAIN_B | | | | 30- | | | | | | | |
| | | | | | | PLAIN_B | | | | | | | |
| | | 120- | | | | 60- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 60- | | | | 30- | | | | | | | |
| | | AS01E_B | | | | AS01E_B | | | | | | | |
| | | 120- | | | | 60- | | | | | | | |
| | | AS01B_B | | | | AS01B_B | | | | | | | |
| | | 120- | | | | 30- | | | | | | | |
| | | AS01B_B | | | | AS01B_B | _ | | | | | <u> </u> | |
| | | 60- | | | | 30- | | | | | | | |
| 01 | | AS01B_B | | | | AS01B_B | | | | | | | |

Short group label = long group label

GM<T,F> = geometric mean antibody <titer, frequency> adjusted for covariates (ANCOVA model)

N = Number of subjects with both pre- and post-vaccination results available

95% CI = 95% confidence interval for the adjusted GMT (Ancova model: adjustment for covariates - pooled variance); LL = lower limit, UL = upper limit

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and the treatment, age category and gender as fixed effects Group 1 is considered superior to Group 2 if one-sided p-value <0.025Template

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

# Template 40 Parameters of the ANCOVA model for the comparison between RSV groups in terms of <RSV A Neutralizing antibody titers, RSVPreF3-specific CD4 T cells expressing at least 2 markers among IL-2, CD40L, TNFa, IFNg>– Part B <analysis set name>

| Timepoint | Variable | DF | <b>Fvalue</b> | p-value |
|---|---|---|---|---|
| <each timepoint=""></each> | Pre-vaccination log <titer, frequency=""></titer,> | | | |
| | Age category | | | |
| | Adjuvant | | | |
| | Antigen | | | |
| | Visit | | | |
| | Linear effect of antigen | | | |
| | Quadratic effect of antigen | | | |
| | Antigen*Adjuvant | | | |

Antigen = Antigen dose (3 levels: 30, 60, 120 mcg)

Adjuvant = Adjuvant content (3 levels: no adjuvant, AS01E, AS01B)

Antigen\*Adjuvant = interaction between antigen dose and adjuvant

ANCOVA model on the log-transformed <titers, frequencies> with the pre-vaccination log-transformed <titer, frequency> as covariate, and adjuvant content, antigen dose and age category as fixed effects DF = degrees of freedom

Interaction (Antigen \* Adjuvant) considered as statistically significant if p-value <0.100

Main factors (Pre-vaccination, antigen, adjuvant) considered as statistically significant if p-value <0.050 (model including interaction)

### **12.4.** Safety

Template 41 Compliance in completing solicited adverse events information (Exposed Set)

| | <each group=""></each> | | |
|---|---|---|---|
| DOSE | N | n | Compliance (%) |
| Vaccination at Visit 1 | xxx | xxx | xx.x |
| Vaccination at Visit 4 | xxx | xxx | xx.x |
| TOTAL | xxx | xxx | xx.x |

Short group label = long group label

N=Number of administered vaccinations

n = number of vaccinations with solicited symptom information completed

Compliance (%) =  $(n / N) \times 100$ 

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 42 Incidence and nature of <grade 3> symptoms (solicited and unsolicited) <with causal relationship to vaccination> reported during the XX-day (Days 1-XX) post-vaccination period following each dose and overall <analysis set name>

| | | <each group=""></each> | | | | | | < | Each g | roup> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | 95% | 95% CI | | | | 95 | % CI | | |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General<br>symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General<br>symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General<br>symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | General symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| | Local symptoms | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose

For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 43 Incidence of any symptoms (solicited and unsolicited) resulting in medically attended visit, reported during the 30-day (Days 1-30) post-vaccination period following each dose and overall <analysis set name>

| | | | <ea< th=""><th>ach gro</th><th>up&gt;</th><th></th><th colspan="6"><each group=""></each></th></ea<> | ach gro | up> | | <each group=""></each> | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% | 95% CI | | | | | 5% CI |
| Dose | Symptoms | N | n | % | LL | UL | N | n | % | LL | UL |
| DOSE 1 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| DOSE 2 | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | XXX | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding administered dose

n/% = number/percentage of subjects presenting at least one type of symptom following the corresponding dose For overall/dose:

N = number of administered dose

n/% = number/percentage of doses followed by at least one type of symptom

For overall/subject:

N = number of subjects with at least one administered dose

n/% = number/percentage of subjects presenting at least one type of symptom

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template 44 Incidence of solicited local symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <analysis set name>

| | | | <e< th=""><th>ach</th><th>grou</th><th>p&gt;</th><th></th></e<> | ach | grou | p> | |
|---|---|---|---|---|---|---|---|
| | | | | | _ | 95 % | CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| DOSE 1 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| DOSE 2 | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/DOSE | <each symptom=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| OVERALL/SUBJECT | <each symptom=""></each> | All | | | | | |
| · | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

## Template 45 Incidence of solicited general symptoms reported during the 7-day (Days 1-7) post-vaccination period following each dose and overall <cohort name>

| | | | <each group=""></each> | | | |
|---|---|---|---|---|---|---|
| | | | 95 % CI | | | |
| Dose | Symptom | Туре | N | n % | LL | UL |
| DOSE 1 | <each except="" fever="" symptom="" –=""></each> | All | | | | |
| | | Grade ≥2 | | | | |
| | | Grade 3 | | | | |
| | | Related | | | | |
| | | Grade ≥2 Related | | | | |
| | | Grade 3 Related | | | | |
| | Fever (°C) | All | | | | |
| | 1 3751 ( 3) | ≥38.0 | | | | |
| | | >38.5 | | | | |
| | | >39.0 | | | | |
| | | >39.5 | | | | |
| | | >40.0 | | | | |
| | | Related | | 1 | + | + |
| | | ≥38.0 Related | | | + | |
| | | >38.5 Related | | | | |
| | | >39.0 Related | | | | |
| | | >39.5 Related | | | | |
| | | >40.0 Related | | | | |
| DOSE 2 | <each except="" fever="" symptom="" –=""></each> | All | | | | |
| | | Grade ≥2 | | | | |
| | | Grade 3 | | | | |
| | | Related | | | | |
| | | Grade ≥2 Related | | | | |
| | | Grade 3 Related | | | | |
| | Fever (°C) | All | | | | |
| | | ≥38.0 | | | | |
| | | >38.5 | | | | |
| | | >39.0 | | | | |
| | | >39.5 | | | | |
| | | >40.0 | | | | |
| | | Related | | | | |
| | | ≥38.0 Related | | | | |
| | | >38.5 Related | | | | |
| | | | | 1 | | |
| | | >39.0 Related | | | | |
| | | >39.5 Related | | | | |
| 0\/EDALL/D00E | Zoob symmetry | >40.0 Related | | 1 | | |
| OVERALL/DOSE | <each except="" fever="" symptom="" –=""></each> | All | | | | |
| | | Grade ≥2 | | | | |
| | | Grade 3 | | | | |
| | | Related | | | | |
| | | Grade ≥2 Related | | | | |
| | | Grade 3 Related | | | | |
| | Fever (°C) | All | | | | |
| | ( - / | ≥38.0 | | | | |
| | | >38.5 | | | | |
| | | >39.0 | | | | |

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

| | | | <e< th=""><th>ach</th><th>grou</th><th>ıp&gt;</th><th></th></e<> | ach | grou | ıp> | |
|---|---|---|---|---|---|---|---|
| | | | | | | 95 % | CI |
| Dose | Symptom | Туре | N | n | % | LL | UL |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |
| OVERALL/SUBJECT | <each except="" fever="" symptom="" –=""></each> | All | | | | | |
| | | Grade ≥2 | | | | | |
| | | Grade 3 | | | | | |
| | | Related | | | | | |
| | | Grade ≥2 Related | | | | | |
| | | Grade 3 Related | | | | | |
| | Fever (°C) | All | | | | | |
| | , , | ≥38.0 | | | | | |
| | | >38.5 | | | | | |
| | | >39.0 | | | | | |
| | | >39.5 | | | | | |
| | | >40.0 | | | | | |
| | | Related | | | | | |
| | | ≥38.0 Related | | | | | |
| | | >38.5 Related | | | | | |
| | | >39.0 Related | | | | | |
| | | >39.5 Related | | | | | |
| | | >40.0 Related | | | | | |

Short group label = long group label

For each dose:

N = number of subjects with the corresponding documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once following the corresponding dose For Overall/dose:

N = number of documented doses

n/% = number/percentage of doses followed by at least one type of symptom

For Overall/subject:

N = number of subjects with at least one documented dose

n/% = number/percentage of subjects reporting the type of symptom at least once

95%CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

## Template 46 Number of days with <local/general> solicited symptoms during <the 7-day (Days 1-7), the whole> post-vaccination period <analysis set name>

| | | | <each group=""></each> |
|---|---|---|---|
| Dose | Symptom | Statistic | Value |
| DOSE 1 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| DOSE 2 | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |
| OVERALL/DOSE | <each symptom=""></each> | n | |
| | | Mean | |
| | | Minimum | |
| | | Q1 | |
| | | Median | |
| | | Q3 | |
| | | Maximum | |

Short group label = long group label

n = number of doses with the symptom

Q1 = 25th percentile

Q3= 75th percentile

Template 47 Incidence of solicited <local, general> adverse events reported during the 7-day (Days 1-7) post-vaccination period following each dose <Exposed set>



Short group label = long group label

Note: this graph is provided as an example. It will be adapted to display the percentage of subjects reporting each local or general symptom, any grade and grade 3, by group and by dose. Template will be discussed at the time of the dry-run.

Template 48 Percentage of subjects reporting the occurrence of <grade 3> unsolicited AEs classified by MedDRA Primary System Organ Class and Preferred Term <with causal relationship to vaccination> within the 30-day (Days 1-30) post-vaccination period <analysis set name>

| | | <eac< th=""><th>h grou<br/>(XX</th><th>p&gt;</th><th></th><th></th><th colspan="5">Total<br/>N=XXXX</th></eac<> | h grou<br>(XX | p> | | | Total<br>N=XXXX | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95% CI | | | | 95% | CI | |
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | LL | UL | n* | N | % | LL | UL |
| | At least one symptom | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | xx.x | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XX.X | XX.X | XXX | Xxx | XX.X | XX.X | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

n\* = number of events reported

n/% = number/percentage of subjects reporting the symptom at least once

95% CI = exact 95% confidence interval; LL = Lower Limit, UL = Upper Limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

### Template 49 List of (S)AEs and solicited adverse events leading to study/treatment discontinuation <Exposed set>

| Sub<br>. No | Countr<br>y | Gende<br>r | AE<br>Descriptio<br>n | SA<br>E | Causalit<br>y | Vaccinatio<br>n and visit | Type of discontinuation * |
|---|---|---|---|---|---|---|---|

Short group label = long group label

## Template 50 Listing of potential immune-mediated disorders (pIMDs) reported as identified by predefined list of preferred terms and/or by investigator assessment <analysis set name>

| Group | Sub.<br>No. | Gender | Country | Age<br>at<br>onset<br>(Year) | Primary System<br>Organ Class |
|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | |
| group> | | | | | |

| | Sub. | | | Day of | | | | | SAE | pIMD source |
|---|---|---|---|---|---|---|---|---|---|---|
| Group | No. | Medical visit type | Dose | onset | Duration | Intensity | Causality | Outcome | (Y/N) | |
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | | | | |
| group> | | | | | | | | | | |

Short group label = long group label

### Template 51 Listing of SAEs <analysis set name>

| Group | Sub.<br>No. | Gender | Country | Race | Age at onset (Year) | Verbatim | Preferred Term |
|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | |
| group> | | | | | | | |

| Group | Primary System<br>Organ Class | Medical visit type | Day<br>of<br>onset | Duration | Intensity | Causality | Outcome |
|---|---|---|---|---|---|---|---|
| <each< td=""><td></td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | | | | | | | |
| group> | | | | | | | |

Short group label = long group label

<sup>\*</sup> type of discontinuation refers to whether the discontinuation is a treatment discontinuation or study follow-up discontinuation

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

### Template 52 Listing of pregnancies reported during the study period in Part A <analysis set name>

| Gr | ou | Sub | Countr | Rac | Age at | Previou | LM | Days | Age at | Date of | Pregnanc | Date of | Gestational |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| p | | | у | е | vaccinatio | s Dose | Р | betwee | deliver | deliver | у | outcom | weeks at |
| | | No. | | | n | | dat | n LMP- | у | у | Outcome | е | birth/miscarriag |
| | | | | | | | е | vacc | (Year) | | | | е |
| | | | | | | | | | | | | | /termination |

Short group label = long group label

LMP=Last Mentrual Period

Template 53 Number and percentage of subjects taking concomitant medication during the <XX>-day (Days 1-<XX>) post-vaccination period by dose and overall <analysis set name>

| | | | <each group=""></each> | | | > | | • | <each< th=""><th colspan="2">group&gt;</th></each<> | group> | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | <95 | >% CI | | | | <95 | >% CI |
| Dose | | N | n | % | LL | UL | N | N | % | LL | UL |
| DOSE x | Any | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| OVERALL/DOSE | Any | xx | XX | XX.X | XX.X | XX.X | XX | Хх | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| OVERALL/SUBJECT | Any | XX | XX | XX.X | XX.X | XX.X | XX | Хx | XX.X | XX.X | XX.X |
| | Antipyretics | | | | | | | | | | |
| | Prophylactic antipyretics | XX | XX | XX.X | XX.X | XX.X | XX | Хх | XX.X | XX.X | XX.X |

Short group label = long group label

For each dose:

N = total number of subjects with the corresponding administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

For overall/dose:

N = number of administered doses

n/% = number/percentage of doses after which the specified type of concomitant medication was taken at least once during the considered period

For overall/subject:

N = total number of subjects with at least one administered dose

n/% = number/percentage of subjects who took the specified type of concomitant medication at least once during the considered period

95% CI = Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 54 Distribution of change from baseline in hematology and biochemistry with respect to normal laboratory ranges <analysis set name>

| | | | | <ea< th=""><th>ach gro</th><th>up&gt;</th><th><e:< th=""><th>ach gro</th><th>up&gt;</th></e:<></th></ea<> | ach gro | up> | <e:< th=""><th>ach gro</th><th>up&gt;</th></e:<> | ach gro | up> |
|---|---|---|---|---|---|---|---|---|---|
| Laboratory parameter | Timing | Range<br>indicator at<br>Baseline (PRE) | Range<br>indicator at<br>timing | N | n | % | N | n | % |
| <each parameter=""></each> | <each< td=""><td>UNKNOWN</td><td>UNKNOWN</td><td></td><td></td><td></td><td></td><td></td><td></td></each<> | UNKNOWN | UNKNOWN | | | | | | |
| | timing> | | BELOW | | | | | | |
| | | | WITHIN | | | | | | |
| | | | ABOVE | | | | | | |
| | | BELOW | UNKNOWN | | | | | | |
| | | | BELOW | | | | | | |
| | | | WITHIN | | | | | | |
| | | | ABOVE | | | | | | |
| | | WITHIN | UNKNOWN | | | | | | |
| | | | BELOW | | | | | | |
| | | | WITHIN | | | | | | |
| | | | ABOVE | | | | | | |
| | | ABOVE | UNKNOWN | | | | | | |
| | | | BELOW | | | | | | |
| | | | WITHIN | | | | | | |
| | | | ABOVE | | | | | | |

Short group label = long group label

N = number of subjects with available results for the specified laboratory parameter and timing in a given baseline category

n/% = number/percentage of subjects in the specified category

Below = below the normal laboratory range defined for the specified laboratory parameter

Within = within the normal laboratory range defined for the specified laboratory parameter

Above = above the normal laboratory range defined for the specified laboratory parameter Short timing label = long timing label

Template 55 Summary of hematology and biochemistry results by maximum grade at <Visit 2 (Day 8), Visit 5 (Day 68)> versus baseline (<Day 1, Day 61>) <analysis set name>

| | | | <eac< th=""><th>ch gro</th><th>oup &gt;</th></eac<> | ch gro | oup > |
|---|---|---|---|---|---|
| Laboratory parameter | Baseline<br>( <day 1,="" day<br="">61&gt;)</day> | Visit <2,5> ( <day 8,<br="">Day 68&gt;)</day> | N | n | % |
| <each parameter=""></each> | Unknown | Unknown | | | |
| | | <each grade=""></each> | | | |
| | <each grade=""></each> | Unknown | | | |
| | | <each grade=""></each> | | | |
| | Total | Unknown | | | |
| | | <each grade=""></each> | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Note: This table will be generated post dose 1 at Visit 2 (Day 8) versus baseline at Day 1, and also post dose 2 at Visit 5 (Day 68) versus baseline at Day 61.

Template 56 Summary of maximum hemoglobin change from baseline at <Visit 2 (Day 8), Visit 5 (Day 68)> (Exposed set)

| | | <ea< th=""><th colspan="6"><each group=""></each></th></ea<> | <each group=""></each> | |
|---|---|---|---|---|
| Laboratory parameter | | N | n | % |
| Hemoglobin - change from baseline | UNKNOWN | | | |
| | GRADE 0 | | | |
| | GRADE 1 | | | |
| | GRADE 2 | | | |
| | GRADE 3 | | | |

Short group label = long group label

N = number of subjects with at least one available result for the specified laboratory parameter and follow-up period

n/% = number/percentage of subjects reporting at least once the laboratory event when the maximum grading over the follow-up period is considered

Note: This table will be generated post dose 1 at Visit 2 (Day 8) with Day 1 as baseline, and also post dose 2 at Visit 5 (Day 68) with Day 61 as baseline.

Template 57 Boxplot of <each hematology/biochemistry parameter> (Exposed Set)



Note: This graph is given as an example. It will be adapted to display one boxplot per group and per timepoint, all timepoints available (5 TPs: Screening, Days 1, 8, 61, 68). For Part A, one graph will be generated displaying the 4 groups. For Part B, 3 graphs will be generated displaying 4 groups: 3 RSV groups (30/60/120 -Plain, - AS01E or -AS01B) and the Placebo group.

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 58 Solicited and unsolicited symptoms classified by MedDRA Primary System Organ Class and Preferred Term within the 30-day (Days 1-30) post-vaccination period including number of events - SAE excluded <analysis set name>

| | | <ea< th=""><th>ch gro</th><th>oup&gt;</th><th colspan="3"><each group=""> N=XXXX</each></th></ea<> | ch gro | oup> | <each group=""> N=XXXX</each> | | |
|---|---|---|---|---|---|---|---|
| Primary System Organ Class (CODE) | Preferred Term (CODE) | n* | n | % | n* | n | % |
| | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| <each (soc="" code)="" soc=""></each> | At least one PT related to the corresponding SOC | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

At least one symptom = at least one symptom experienced (regardless of the MedDRA Preferred Term)

N = number of subjects included in the considered analysis set in each group

n/% = number/percentage of subjects reporting the symptom at least once

Template 59 Number (%) of subjects with serious adverse events during the study period including number of events reported <analysis set name>

| | | | <eacl< th=""><th>h group&gt;</th><th>&gt;</th><th colspan="3"><each group=""> N=XXXX</each></th></eacl<> | h group> | > | <each group=""> N=XXXX</each> | | |
|---|---|---|---|---|---|---|---|---|
| Type of Event | Primary System Organ Class (CODE) | Preferred Term<br>(CODE) | n* | n | % | n* | n | % |
| SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |
| Related SAE | | At least one symptom | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | XXX | XXX | XX.X | XXX | XXX | XX.X |
| | | | xxx | XXX | XX.X | XXX | XXX | XX.X |
| Fatal SAE | | At least one symptom | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | <pre><each (soc="" code)="" soc=""></each></pre> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | | | xxx | XXX | XX.X | XXX | XXX | XX.X |
| Related Fatal | | At least one symptom | XXX | xxx | XX.X | xxx | xxx | XX.X |
| SAE | <each (soc="" code)="" soc=""></each> | <each (pt="" code)="" pt=""></each> | xxx | XXX | XX.X | XXX | XXX | XX.X |
| | | | XXX | XXX | XX.X | XXX | XXX | XX.X |

Short group label = long group label

N = number of subjects with administered dose

n/% = number/percentage of subjects reporting the symptom at least once

n\* = Number of events reported

Related = assessed by the investigator as related

n\* = number of events reported

### 12.5. Analysis of RTI

Template 60 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <analysis set name>

| | | | <ea< th=""><th>ach</th><th>gro</th><th>up&gt;</th><th></th><th>1</th><th>ota</th><th>l</th><th></th></ea<> | ach | gro | up> | | 1 | ota | l | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95% C | |
| Samples | RSV status | N | n | % | LL | UL | N | n | % | LL | UL |
| Nasal/throat swab at assessment visit | RSV+ | | | | | | | | | | |
| | RSV- | | | | | | | | | | |
| | All | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by qRT-PCR at least once

RSV-= subjects tested as RSV negative by qRT-PCR

All= subjects with at least one gRT-PCR result available

N = number of subjects in each group or in Total

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

Template 61 Number and percentages of subjects with at least one RSV-confirmed RTI episode post-vaccination, as measured by qRT-PCR in nasal swab samples collected at home <analysis set name>

| | | | <ea< th=""><th>ich</th><th>gro</th><th>up&gt;</th><th colspan="5">Total</th></ea<> | ich | gro | up> | Total | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | | | | | 95 | % CI | | | | 95% | % CI |
| Samples | RSV status | N | n | % | LL | UL | N | n | % | LL | UL |
| Nasal swab at home | RSV+ | | | | | | | | | | |
| | RSV- | | | | | | | | | | |
| | All | | | | | | | | | | |

Short group label = long group label

RSV+= subjects tested RSV positive by gRT-PCR at least once

RSV-= subjects tested as RSV negative by qRT-PCR

All= subjects with at least one qRT-PCR result available

N = number of subjects in each group

n/%= number/percentage of subjects in each category

95%CI= Exact 95% confidence interval; LL = lower limit, UL = upper limit

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 62 Mean of the viral load of the RSV-confirmed RTI episodes, as measured by qRT-PCR on nasal/throat swabs, by collection time and collection method <Exposed set>

| | | | F | RSV A | <b>\</b> + | | RS | V B + | |
|---|---|---|---|---|---|---|---|---|---|
| Days after<br>RTI onset | Swab | N | n | % | mean | N | n | % | mean |
| 0-2 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |
| 3-4 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |
| >4 | Nasal swab at home | | | | | | | | |
| | Nasal/throat swab at assessment visit | | | | | | | | |

Days after RTI onset = number of days between start of RTI symptoms and collection date

N=Number of swabs with gRT-PCR results available

n/%= number/percentage of swabs tested as RSV A/B positive by qRT-PCR

mean= mean of the viral load computed on RSV A/B positive swabs

Template 63 Descriptive statistics of the viral load of the RSV- confirmed RTI episodes, as measured by qRT-PCR in nasal/throat swab samples collected at assessment visit <at home> <Exposed Set>

| | | <each group=""><br/>N=</each> | Total<br>N= |
|---------|------------|-------------------------------|-------------|
| Туре | Parameters | Value | Value |
| RSV A + | n | | |
| | Mean | | |
| | Min | | |
| | Q1 | | |
| | Median | | |
| | Q3 | | |
| | Max | | |
| RSV B + | | | |
| All RSV | | | |
| + | | | |

Short group label = long group label

RSV A+= RSV A positive samples by gRT-PCR

RSV B+-= RSV B positive samples by qRT-PCR

All RSV += All RSV positive samples by qRT-PCR

N = Number of swabs with qRT-PCR results available

n= number/percentage of samples in each category

Q1 and Q3 = 25th and 75th percentiles

Min/Max = Minimum/Maximum

208851 (RSV OA=ADJ-002) Statistical Analysis Plan Final

Template 64 Number and percentage of subjects reporting co-infections with respiratory viruses, as measured by multiplex PCR on RSV A/B positive RTI samples collected <at assessment visit, at home > <Exposed Set>

| | | R | N= | SV RTI<br>N = |
|------------------------|---|---|--------|---------------|
| | | | 95% CI | |
| Categories | n | % | LL | UL |
| Influenza A Virus | | | | |
| Influenza B Virus | | | | |
| <each virus=""></each> | | | | |
| Total | | | | |

N = number of swabs tested RSV positive by qRT-PCR

n/% = number/percentage of swabs tested positive by multiplex in a given category

Total= number of swabs tested positive for at least one virus

LL, UL= Exact 95% Lower and Upper confidence limits

### Template 65 Clinical signs and symptoms associated with RTI episodes (Exposed set)

| | | RSV RTI<br>N=XXXX<br>n % | | RSV RTI<br>=XXXX | Total<br>N=XXXX | |
|---|---|---|---|---|---|---|
| Characteristics | Categories | | n | % | n | % |
| Heart Rate increase<br>(beats/min) | 10-20 | | | | | |
| , | 20-30 | | | | | |
| | 30-40 | | | | | |
| | 40-50 | | | | | |
| Respiratory rate increase (breaths/min) | 5-10 | | | | | |
| , | 10-15 | | | | | |
| | 15-20 | | | | | |
| | 20-25 | | | | | |
| Systolic blood pressure increase (mmHg) | 10-20 | | | | | |
| ( 0, | 20-30 | | | | | |
| | 30-40 | | | | | |
| | 40-50 | | | | | |
| Diastolic blood pressure increase (mmHg) | 10-20 | | | | | |
| ( 0/ | 20-30 | | | | | |
| | 30-40 | | | | | |
| | 40-50 | | | | | |
| Oxygen saturation decrease (%) | 1-2 | | | | | |
| . , | 3-4 | | | | | |
| | 5-6 | | | | | |
| | 7-8 | | | | | |
| Upper respiratory symptoms | <each symptom=""></each> | | | | | |
| | • | | | | | |
| Lower respiratory symptoms | <each symptom=""></each> | | | | | |
| qPCR result | RSV A+ | | | | | |
| | RSV B+ | | | | | |
| | RSV - | | | | | |
| Self-collected Nasal swab | RSV+ | | | | | |
| | RSV- | | | | | |
| | NA | | | | | |
| Medically attended visit | Emergency room | | | | | |
| | Hospitalisation | | | | | |
| | Medical personnel | | | | | |
| | None | | | | | |
| SAE associated to the episode | Yes | | | | | |
| | No | | | | | |

RSV RTI= RTI episode tested as RSV positive by qRT-PCR on nasal/throat swab collected at assessment visit Non-RSV RTI= RTI episode tested as RSV negative by qRT-PCR on nasal/throat swab collected at assessment visit N = number of RTI episodes in each category or in total

n = number of RTI episodes in the corresponding category

 $% = n / N \times 100$ 

For vital signs, change from baseline (increase/decrease) will be displayed by category: category of 10 units increase for heart rate, systolic and diastolic BP, 5 units increase for respiratory rate, and 1% decrease for oxygen saturation (to be adapted at the time of dry run if needed)

Template 66 Listing of RTI episodes reported during RTI surveillance in Part B (Exposed set)

| Grou | Su | Age | Se | Episo | Start | End | Date of | Nb of | Dat | RSV | RSV | Dat | RSV- | RSV- | Medica | SAE |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| р | b. | at | X | de nb | date | date | assessm | signs | е | Α | В | е | Α | В | lly | relate |
| | No. | Dos | | | of | of | ent visit | and | nas | positi | positi | nas | positi | positi | attende | d to |
| | | e 1 | | | episo | episo | | sympto | al | ve | ve | al | ve | ve | d visit | RTI |
| | | | | | de | de | | ms | swa | (site) | (site) | swa | (home | (home | | episo |
| | | | | | | | | | b | | | b at | ) | ) | | de |
| | | | | | | | | | on | | | hom | | | | |
| | | | | | | | | | site | | | е | | | | |
| | | | | | | | | | | Yes/N | Yes/N | | Yes/N | Yes/N | | Yes/N |
| | | | | | | | | | | 0 | 0 | | 0 | 0 | | 0 |

Short group label = long group label

Template 67 GMTs and 95% CIs of RSV A Neutralizing antibody titer at baseline for subjects reporting RTI episodes (RSV RTI vs or non RSV RTI vs No RTI), by groups pooled according to the adjuvant content <Exposed Set>



This graph is provided as an example, template will be finalized at the time of the dry-run. It will display the GMTs and 95% CIs for subjects reporting confirmed RSV RTI episodes vs subjects reporting Non-RSV RTI episodes vs subjects who did not report any RTI episode (NON RTI), in the RSV groups pooled according to the adjuvant content (Plain, AS01E, AS01B).